#### Stat Analysis Plan V3

A Phase 3, Multicenter Study with a 36-Week Open-Label Period Followed by a Randomized Double-Blind Withdrawal Period from Week 36 to Week 104 to Evaluate the Long-Term Efficacy and Safety of Ixekizumab (LY2439821) 80 mg Every 2 Weeks in Biologic Disease-Modifying Antirheumatic Drug-Naive Patients with Active Psoriatic Arthritis

NCT02584855

Approval Date: 25-Oct-2018

# 1. Statistical Analysis Plan:

I1F-MC-RHBF: Phase 3, Multicenter Study with a 36-Week Open-Label Period Followed by a Randomized Double-Blind Withdrawal Period from Week 36 to Week 104 to Evaluate the Long-Term Efficacy and Safety of Ixekizumab (LY2439821) 80 mg Every 2 Weeks in Biologic Disease-Modifying Antirheumatic Drug-Naive Patients with Active Psoriatic Arthritis

#### **Confidential Information**

The information contained in this Statistical Analysis Plan (SAP) is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiaries. This document and its associated attachments or appendices are subject to United States Freedom of Information Act Exemption 4.

#### Ixekizumab (LY2439821) Psoriatic Arthritis

Study I1F-MC-RHBF is a Phase 3, multicenter study with a 36-week initial open-label treatment period examining the effect of ixekizumab 80 mg every 2 weeks (Q2W) in patients with active psoriatic arthritis (PsA) who are conventional disease-modifying antirheumatic drug (cDMARD) inadequate responders (IRs) and biologic disease-modifying antirheumatic drug (bDMARD)-naive followed by a randomized, double-blind withdrawal period from Week 36 to Week 104 examining the effect of ixekizumab 80 mg Q2W compared to that of placebo.

Eli Lilly and Company Indianapolis, Indiana USA 46285 Protocol I1F-MC-RHBF Phase 3

Statistical Analysis Plan Version 1 electronically signed and approved by Lilly: 30 October 2015

Statistical Analysis Plan Version 2 electronically signed and approved by Lilly: 20 April 2017

Statistical Analysis Plan Version 3 electronically signed and approved by Lilly on date provided below

Approval Date: 25-Oct-2018 GMT

# 2. Table of Contents

| Section | Page |
|---|---|
| 1. Statistical Analysis Plan: I1F-MC-RHBF: Phase 3, Multicenter Study with a 36-Week Open-Label Period Followed by a Randomized Double-Blind Withdrawal Period from Week 36 to Week 104 to Evaluate the Long-Term Efficacy and Safety of Ixekizumab (LY2439821) 80 mg Every 2 Weeks in Biologic Disease-Modifying Antirheumatic Drug-Naive Patients with Active Psoriatic Arthritis | 1 |
| 2. Table of Contents | 2 |
| 3. Revision History | 8 |
| 4. Study Objectives | 11 |
| 4.1. Primary Objective | 11 |
| 4.2. Secondary Objectives | |
| 4.3. Exploratory Objectives | |
| 5. Study Design | |
| 5.1. Summary of Study Design | |
| <ul><li>5.2. Determination of Sample Size</li><li>5.3. Method of Assignment to Treatment</li></ul> | |
| 6. A Priori Statistical Methods 6.1. General Considerations | |
| 6.1.1. General Considerations for Analyses during Period 2 (Initial Open-Label Treatment Period) | |
| 6.1.1.1. Initial Open-Label Treatment Period Population | |
| 6.1.2. General Considerations for Analyses during Period 3 (Randomized Double-Blind Withdrawal Period) | |
| 6.1.2.1. Randomized Withdrawal ITT and Randomized Withdrawal Safety Populations | 19 |
| 6.1.2.2. Relapse Population | 21 |
| 6.1.3. General Considerations for Analyses during Period 2 and Period 3 Combined (Initial Open-Label Treatment and Randomized Double-Blind Withdrawal Periods) | 22 |
| 6.1.3.1. Ixekizumab 80 mg Q2W-Treated Patients from the Randomized Withdrawal ITT Population | 22 |
| 6.1.3.2. Nonrandomized Population | 23 |
| 6.1.4. General Considerations for Analyses during Period 4 (Post- | |
| Treatment Follow-up Period) | |
| 6.2. Adjustments for Covariates | |
| 6.3. Handling of Dropouts or Missing Data | 24 |

| 6.3 | 3.1. | Nonresponder Imputation (NRI) for Clinical Response | 24 |
|---|---|---|---|
| 6.3 | 3.2. | Modified Baseline Observation Carried Forward (mBOCF) | 24 |
| 6.4. | Mu | ticenter Studies | 25 |
| 6.5. | Mu | tiple Comparisons/Multiplicity | 25 |
| 6.6. | Use | of an "Efficacy Subset" of Patients | 25 |
| 6.6 | 5.1. | Analysis Populations | 25 |
| 6.7. | Pati | ent Disposition | 26 |
| 6.8. | Pati | ent Characteristics | 27 |
| 6.8 | 3.1. | Previous Therapy for Psoriatic Arthritis | 32 |
| 6.8 | 3.2. | Historical Illness and Preexisting Conditions | 33 |
| 6.9. | Trea | atment Compliance | 33 |
| 6.10. | | comitant Therapy | |
| 6.11. | . Effi | cacy Analyses | 36 |
| 6.1 | 1.1. | Primary Outcome and Methodology | 48 |
| 6.1 | 1.2. | Secondary Efficacy Analyses | 48 |
| 6.1 | 1.3. | Sensitivity Analyses | 48 |
| 6.12. | Bio | analytical and Pharmacokinetic/Pharmacodynamic Methods | 48 |
| 6.13. | Safe | ety Analyses | 48 |
| 6.1 | 3.1. | Extent of Exposure | 49 |
| 6.1 | 3.2. | Adverse Events | 50 |
| 6.1 | 3.3. | Deaths, Other Serious Adverse Events, and Other Notable | |
| | | Adverse Events | |
| 6 | 5.13.3. | 1. Deaths | 53 |
| 6 | 5.13.3. | 2. Serious Adverse Event Analyses | 53 |
| 6 | 5.13.3 | 3. Other Significant Adverse Events | 54 |
| 6.1 | 3.4. | Depression and Suicide-Related Patient Reported Outcomes | 54 |
| 6.1 | 3.5. | Clinical Laboratory Evaluation. | 55 |
| 6 | 5.13.5 | 1. Leukocytes (WBC) and Platelets | 58 |
| 6 | 5.13.5 | 2. Neutrophil Follow-Up | 58 |
| 6.1 | 3.6. | Vital Signs and Other Physical Findings. | 59 |
| 6.1 | 3.7. | Special Safety Topics including Adverse Events of Special | |
| | | Interest | |
| 6.1 | 3.8. | Immunogenicity | |
| 6 | 5.13.8. | | |
| | | 8.1.1. Sample Category Definitions | |
| | | 8.1.2. Patient Category Definitions | 75 |
| | 6.13 | 8.1.3. Definitions for Clinical Interpretation of Assay | 70 |
| , | 12.0 | Results | /6<br>79 |
| | | / Immun(Manicity/Anglycac | / V |

| 6.13.8.2.1. | Analyses of Characteristics of ADA Immune Response | 80 |
|---|---|---|
| 6.13.8.2.2. | Analyses of Treatment-Emergent ADA Effects on | |
| 6.13.8.2.3. | Analyses of Treatment-Emergent ADA on Specific | |
| . Subgroup | Analyses | 82 |
| 14.1. Effica | acy Subgroup Analysis | 82 |
| 14.2. Safet | y Subgroup Analysis | 84 |
| . Analysis fo | or Australian Submission | 85 |
| | | 85 |
| . Protocol D | eviations | 85 |
| . Interim An | nalyses and Data Monitoring | 100 |
| . Planned Ex | xploratory Analyses | 100 |
| 19.1. Plann | ed Exploratory Efficacy Analysis | 100 |
| | | 115 |
| _ | | |
| Jnblinding Pl | an | 131 |
| References | | 132 |
| Appendices | | 136 |
| | 6.13.8.2.2. 6.13.8.2.3. Subgroup J. 14.1. Effica 14.2. Safet J. Analysis for Care Excels. Protocol D. Interim Art. Planned Extension Plann | Response 6.13.8.2.2. Analyses of Treatment-Emergent ADA Effects on Efficacy 6.13.8.2.3. Analyses of Treatment-Emergent ADA on Specific Adverse Events. Subgroup Analyses 14.1. Efficacy Subgroup Analysis 14.2. Safety Subgroup Analysis Analysis for Australian Submission Analysis for United Kingdom National Institute for Health and Care Excellence Submission Protocol Deviations Interim Analyses and Data Monitoring Planned Exploratory Analyses 19.1. Planned Exploratory Efficacy Analysis 19.2. Planned Exploratory Health Outcomes/Quality-of-Life Analyses Annual Report Analyses Clinical Trial Registry Analyses Unblinding Plan References |

# **Table of Contents**

| Table | Page |
|---|---|
| Table RHBF.6.1. Geographic Regions | 25 |
| Table RHBF.6.2. Date of First Injection by Period and Analysis Population | 27 |
| Table RHBF.6.3. Description and Derivation of Primary and Secondary Efficacy Outcomes | 37 |
| Table RHBF.6.4. Description of Primary and Secondary Efficacy Analyses | 42 |
| Table RHBF.6.5. Categorical Criteria for Abnormal Treatment-Emergent Blood Pressures and Pulse Measurement, and Categorical Criteria for Weight Changes for Adults | 61 |
| Table RHBF.6.6. Definitions and Analyses of Special Safety Topics Including Adverse Events of Special Interest | 63 |
| Table RHBF.6.7. TE-ADA Status Dichotomous Variables for AE analysis | 79 |
| Table RHBF.6.8. Identification and Action of Important Protocol Deviations | 87 |
| Table RHBF.6.9. Description and Derivation of Additional Exploratory Outcomes | 101 |
| Table RHBF.6.10. Description of Planned Exploratory Efficacy Analyses | 106 |
| Table RHBF.6.11. Description and Derivation of Health Outcomes and Quality-of-Life Measures | 116 |
| Table RHBF.6.12. Description of Planned Exploratory Health Outcomes and Quality-of-Life Analyses | 124 |

# **Table of Contents**

| Figure | | Page |
|---|---|---|
| Figure RHBF.5.1. | Illustration of study design for Clinical Protocol I1F-MC-RHBF | 15 |
| Figure RHBF.6.1. | Sample definitions. | 75 |
| • | Patient categories (evaluable/unevaluable) based on sample status at aseline and post-baseline. | 76 |
| _ | Relationship of terms for clinical interpretation of assay results for valuable patients. | 77 |
| • | Flow chart of ADA assessment with clinical interpretation of the arious result possibilities. | 78 |

# **Table of Contents**

| Appendix | | Page |
|---|---|---|
| Appendix 1. | Algorithm for Calculating Classification for Psoriatic Arthritis (CASPAR) Total Score | 137 |
| Appendix 2. | Algorithm for Calculating Coates Criteria for Minimal Disease Activity (MDA) | 138 |
| Appendix 3. | Algorithm for Calculating Joint Counts | 139 |
| Appendix 4. | Algorithm for Calculating the Health Assessment Questionnaire—<br>Disability Index (HAQ-DI) | 140 |
| Appendix 5. | Algorithm for Determining American College of Rheumatology (ACR) Response | 142 |
| Appendix 6. | Derivation of SF-36v2® Health Survey, Acute Version Scores | 144 |
| Appendix 7. | Anti-infective Medications and Anatomical Therapeutic Chemical (ATC) Code List and Programming Guide | 150 |
| Appendix 8. | MedDRA Preferred Terms for Each Category Associated with Criterion 2 for Anaphylactic Allergic Reactions/Hypersensitivity Events | 156 |
| Appendix 9. | Allergic Reactions/Hypersensitivity MedDRA Preferred Terms | 158 |
| Appendix 10. | Algorithm for Calculating Composite Psoriatic Disease Activity Index (CPDAI) | 161 |
| Appendix 11. | Lilly-defined MedDRA V21.0 Preferred Terms for Inflammatory<br>Bowel Disease (IBD) | 163 |
| Appendix 12. | Lilly-defined MedDRA V21.0 Preferred Terms for Opportunistic Infections (OI) | 165 |

# 3. Revision History

Statistical Analysis Plan (SAP) Version 1 was approved on 30 October 2015 prior to first patient visit.

Two protocol amendments were completed after the SAP Version 1 was approved. Protocol amendment (a) was approved on 10 February 10 2016 and protocol amendment (b) was approved on 21 March 2017.

Statistical Analysis Plan (SAP) Version 2 was approved on 20 April 2017 prior to unblinding of patients randomized in the double-blind randomized withdrawal period. The changes incorporated in SAP Version 2 are as follows:

- Conventional disease-modifying antirheumatic drug (cDMARD) use was added
  as a stratification parameter to the primary analysis log-rank model. Protocol I1FMC-RHBF (RHBF) Section 12.2.6.1 indicates that only geographic region is used
  as a stratification parameter in the model. However, cDMARD use (past, current)
  is also a stratification parameter in the randomization scheme and should be added
  to the primary analysis model.
- Similarly, cDMARD use will be added as stratification parameter to the logistic regression model for the categorical efficacy and health outcomes analyses (see Protocol Section 12.2.1.2).
- Psoriatic arthritis (PsA) subtypes will not be included in the baseline patient characteristic analysis. Although this was stated in the protocol, the information is not collected.
- The missing data imputation method, modified baseline observation carried forward (mBOCF) was added to the SAP. This method will be used in addition to last observation carried forward (LOCF). If a case arises in which using these 2 methods is not consistent, the mBOCF method will be the primary method.
- Clarified the population for the Health Assessment Questionnaire—Disability Index (HAQ-DI) total score improvement ≥0.35 analysis. Patients need to have baseline HAQ-DI total score ≥0.35 to be considered for improvement.
- Clarified the definition for the analysis on tender entheseal points will be based on the assessment of the 18 entheseal points.
- Corrected the derivation for duration of exposure for Period 2 and Period 3 combined.
- Updates to the safety analysis per program safety analysis plan (PSAP) Version 7.
- Updates to the immunogenicity analysis per PSAP Version 7.
- Clarified that the longitudinal analyses will be summarized by treatment week instead of by visit and through 40 weeks of treatment.
- Added secondary analyses for C-reactive protein (CRP).

Statistical Analysis Plan (SAP) Version 3 was approved prior to unblinding of patients randomized in the double-blind randomized withdrawal period. The changes incorporated in SAP Version 3 are as follows:

- Added analyses for disease activity in PsA (DAPSA).
- Removed analyses for DLQI (0).
- Clarified that longitudinal analyses will be done by treatment week through the last observation for the Randomized Double-Blind Withdrawal Period and the Relapse Period.
- Clarified that only analyses within the Randomized Double-Blind Withdrawal Period will include missing data imputations (NRI for categorical endpoints and mBOCF for continuous endpoints).
- Clarified that pre-existing conditions are defined as having a start date prior to the date of informed consent and not prior to the date of first study drug injection.
- Clarified that the treatment compliance calculation for Period 3 does not include the loading dose.
- Removed analyses for treatment compliance and protocol deviation analyses for the relapse period and the combined Periods 2 and 3.
- Clarified that the time-to endpoints in Period 3 are calculated with respect to the start of Period 3 and not Period 2.
- Removed a majority of the safety analyses for the post-treatment follow-up period.
- Clarified that categorical analyses assessed during Period 3 will be assessed through 40 weeks of randomized treatment with the exception of the proportion of patients who relapse. The analyses for the proportion of patients who relapse will be assessed over the entire randomized withdrawal study period with cumulative rate. Additionally, the proportion of patients who relapse will be described by treatment week for the entire randomized withdrawal study period.
- Removed laboratory and vital sign analyses for change from baseline to each scheduled post-baseline visit.
- Removed laboratory and vital sign box plots.
- Added laboratory shift tables for neutrophils, leukocytes, platelets, and lymphocytes.
- Removed common adverse event section and moved the exposure-adjusted analysis details to the general consideration section.
- Removed the region pooling statement.
- For AESIs:
  - o removed analyses for elevated hepatic criteria;

- o removed the TEAE table for opportunistic infections by preferred term;
- o removed TEAE table for ISRs by preferred term within high-level terms; and
- o removed analyses for IBD and ILD with the except of TEAE by preferred tem by max severity by preferred term within category.
- Added a protocol deviation for patients who start on IXE in the Randomized Double-Blind Withdrawal Period prior to experiencing a relapse (no longer meeting Coates criteria for MDA in Period 3). These patients will also be removed from the PPS.
- Updated the derivation of the protocol deviations for entry criteria [1] and [4].
- Updated the statistical model for testing efficiacy subgroup interactions to the Coxproprotional hazards model.
- Added Appendix 2 for calculating Coates criteria for minimal disease activity (MDA).
- Clarified the algorithm for calculating Joint Counts (see Appendix 3).
- AESIs were updated per the updated with changes from the PSAP Verions 7 and 8.
- Made other minor typographical corrections and clarifications not affecting content.

# 4. Study Objectives

# 4.1. Primary Objective

The primary objective of the study is to compare ixekizumab 80 mg every 2 weeks (Q2W) with placebo in maintenance of treatment response, as measured by the time-to relapse during the randomized double-blind withdrawal period in cDMARD inadequate responders (cDMARD-IR) and biologic DMARD-naive (bDMARD-naive) patients with active PsA who meet randomization criteria (Coates criteria for minimal disease activity [MDA] for 3 consecutive months over 4 consecutive visits).

# 4.2. Secondary Objectives

The secondary objectives of the study are:

- to compare ixekizumab 80 mg Q2W with placebo in maintenance of treatment response, as measured by the proportion of patients who meet relapse criteria during the randomized double-blind withdrawal period in cDMARD-IR and bDMARD-naive patients with active PsA who meet randomization criteria (Coates criteria for MDA for 3 consecutive months over 4 consecutive visits)
- to evaluate the time-to loss of response for each individual component of MDA in the randomized double-blind withdrawal period
- to evaluate time-to first meeting Coates criteria for MDA during the initial openlabel treatment period (Period 2)
- to evaluate time-to achieving Coates criteria for MDA during the initial openlabel treatment period (Period 2) (Coates criteria for MDA for 3 consecutive months over 4 consecutive visits)
- to assess the efficacy of ixekizumab 80 mg Q2W after disease relapse after randomization in the randomized double-blind treatment period
- to assess the effect of treatment response as measured by the HAQ-DI of ixekizumab 80 mg Q2W throughout the study.

# 4.3. Exploratory Objectives

The exploratory objectives of the study are:

- to assess the clinical factors that predict Coates criteria for MDA
- to assess the time-to achieve other composite measurements of low disease activity, such as Disease Activity Score modified to include the 28 diarthrodial joint count, based on C-reactive protein (DAS28-CRP), Psoriatic Arthritis Disease Activity Score (PASDAS), Composite Psoriatic Disease Activity Index (CPDAI), and others during the initial open-label treatment period (Period 2)
- to assess the changes in health utility (European Quality of Life–5 Dimensions 5 Level [EQ-5D 5L]), Work Productivity and Activity Impairment–Specific Health Problem, and Dermatology Life Quality Index (DLQI) throughout the study

- to assess the changes in the health outcome endpoints Fatigue Severity Numeric Rating Scale (NRS) score, Itch NRS score (in the subgroup of patients with psoriatic skin lesions involving ≥3% body surface area [BSA] at baseline), Quick Inventory of Depressive Symptomatology-self report 16 items (QIDS-SR16) score, and Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS), and Mental Component Summary (MCS) scores and the 8 associated domains of SF-36 (Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health) throughout the study
- to explore biomarkers of disease or drug activity that may be contained in serum, plasma, and whole-blood messenger ribonucleic acid (RNA) and deoxyribonucleic acid (DNA) samples
- to assess the pharmacokinetic (PK)/pharmacodynamic (PD) relationship and immunogenicity of ixekizumab throughout the study by:
  - o characterizing the PK of ixekizumab, determining the magnitude of withinand between-patient variability, and identifying the potential intrinsic and extrinsic factors that may have an effect on the PK of ixekizumab
  - characterizing the exposure-response relationships for efficacy endpoints (for example, proportion of patients achieving Coates criteria for MDA from Week 36 through Week 64 and the maintenance of treatment effects), and identifying potential factors that may impact the efficacy endpoints
  - evaluating the potential development of anti-ixekizumab antibodies and its impact on patient safety, efficacy, and PK of ixekizumab.

# 5. Study Design

# 5.1. Summary of Study Design

Study RHBF is a Phase 3, multicenter study with a 36-week initial open-label treatment period examining the effect of ixekizumab 80 mg Q2W in patients with active PsA who are cDMARD-IRs and are bDMARD naive followed by a randomized double-blind withdrawal period from Week 36 to Week 104 examining the effect of ixekizumab 80 mg Q2W compared with that of placebo. Patients who do not meet the randomized withdrawal criteria will continue on ixekizumab 80 mg Q2W uninterrupted during the randomized double-blind withdrawal period. All randomized patients who no longer meet Coates criteria for MDA at any visit after entering the randomized double-blind withdrawal period will receive ixekizumab 80 mg Q2W for the remainder of the study period. In addition, efficacy and safety will be assessed for up to a total of 2 years for patients who participate throughout the entire 2-year study.

The study consists of 4 periods:

- **Period 1:** screening period (Visits 1 and 1A) lasting from 4 to 30 days before Week 0 (Visit 2)
- **Period 2:** initial open-label treatment period from Week 0 (baseline, Visit 2) up to Week 36 (Visit 12)
- **Period 3:** randomized double-blind withdrawal period from Week 36 to Week 104 (Visit 29). Patients who have been treated with ixekizumab 80 mg Q2W for at least 36 weeks and have achieved 4 consecutive visits of meeting Coates criteria for MDA from Week 36 up to Week 64 will be eligible for randomization at the visit at which these criteria are met.
- **Period 4:** post-treatment follow-up period occurring from the early termination visit (ETV) or the last scheduled visit for a minimum of 12 weeks after that visit, up to 24 weeks if the patient's neutrophil count is low. All patients withdrawing from the study after receiving even 1 dose of study treatment will proceed directly to Period 4.

Figure RHBF.5.1 illustrates the study design.

All procedures to be conducted during the study, including timing of all procedures, are indicated in the study schedule (Protocol Attachment 1). Selected study procedures should be performed before administration of the investigational product, as applicable, according to the study schedule. Protocol Section 10.4 describes collection of laboratory samples; Protocol Attachment 2 lists the specific laboratory tests that will be performed for this study.

Patients discontinuing from the study who have received at least 1 dose of investigational product should complete the early termination visit (ETV) before proceeding to the post-treatment follow-up period (Period 4). For the management of patient safety, all patients should be monitored through the post-treatment follow-up period at least as frequently as indicated on the study schedule (Protocol Attachment 1).

All treatment groups are described in Protocol Section 9.1. Details of the administration of the investigational product are described in Protocol Section 9.1.1, special treatment considerations are outlined in Protocol Section 9.5.1, and the use of the study drug administration log is detailed in Protocol Section 9.5.2.

Excluded and restricted therapies are detailed in Protocol Section 9.8.

Pharmacokinetic sampling is detailed in Protocol Section 10.4.4.



Figure RHBF.5.1. Illustration of study design for Clinical Protocol I1F-MC-RHBF.

Abbreviations: LV = date of last visit; LY = LY2439821 (ixekizumab); MDA = minimal disease activity; n = number of patients; Q2W = every 2 weeks; RW = randomized withdrawal; V = study visit; w = study week.

- <sup>a</sup> The initial open-label treatment period (Period 2) encompasses Week 0 up to Week 36. During Period 2, all patients will receive open-label ixekizumab 80 mg Q2W.
- b Between Week 36 and Week 64 (inclusive), patients who have been treated with ixekizumab 80 mg Q2W for at least 36 weeks and have achieved 4 consecutive visits of meeting Coates criteria for MDA will be eligible for randomization at the visit at which these criteria are met. Eligible patients will be randomized in a 1:1 ratio to 1 of 2 treatment arms: ixekizumab 80 mg Q2W or placebo Q2W. Patients will remain in their RW treatment arms until they no longer meet Coates criteria for MDA, at which point they will receive ixekizumab 80 mg Q2W. Patients who do not meet Coates criteria for MDA at Week 52 are not eligible for randomization.
- c Patients who do not meet the RW eligibility criteria by Week 64 will remain on ixekizumab 80 mg Q2W uninterrupted for the duration of Period 3.
- d Patients who no longer meet Coates criteria for MDA during Period 3 (the RW period) will be switched to ixekizumab 80 mg Q2W. Patients who continue to meet Coates criteria for MDA during Period 3 (the RW period) will continue treatment until Week 104 and move to Period 4 (the post-treatment follow-up period).

#### 5.2. Determination of Sample Size

Approximately 400 patients will enter the initial open-label treatment period. It is expected that approximately 34% of the patients will meet the randomization criteria for the randomized double-blind withdrawal period. Approximately 136 patients will be randomized in a 1:1 ratio into ixekizumab 80 mg Q2W and placebo treatment groups (68 patients per treatment group). This assumption is based on Study RHAP Week 24 results and estimating the number of patients achieving Coates criteria for MDA for 3 consecutive months over 4 consecutive visits of meeting MDA.

It is assumed that approximately 60% and 20% of patients in the placebo and ixekizumab groups, respectively, who enter the randomized double-blind withdrawal period will relapse (no longer meet Coates criteria for MDA). According to these assumptions, a total of 39 patients must meet relapse criteria in the combined treatment groups to achieve 95% power to test the superiority of ixekizumab 80 mg Q2W to placebo for time-to relapse at a 2-sided  $0.05~\alpha$  significance level. The dropout rate before relapse for patients randomized in the randomized double-blind withdrawal period is assumed to be 10%. Sample size and power calculations were calculated using nQuery+nTerim 3.0.

Randomization and relapse rates will be monitored to assess whether the number of patients who enter the initial open-label treatment period should be increased to ensure sufficient sample size and power for the randomized withdrawal period.

## 5.3. Method of Assignment to Treatment

Patients who meet the eligibility criteria for randomization any time from Week 36 through Week 64 will be randomized to double-blind treatment groups as determined by a computer-generated random sequence using an interactive web-response system (IWRS). The IWRS will be used to assign double-blind investigational product to each patient. Site personnel will confirm that they have located the correct assigned investigational product package by entering a confirmation number found on the package into the IWRS. Patients will be stratified by geographic region and cDMARD use (past use, current use) at the time of randomization in Period 3.

#### 6. A Priori Statistical Methods

#### 6.1. General Considerations

Statistical analysis of this study will be the responsibility of Eli Lilly and Company (hereafter Lilly). The statistical analyses will be performed using SAS® Version 9.2 or higher.

Continuous data will be summarized in terms of the number of observations, mean, standard deviation (SD), minimum, median, and maximum. The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database. The mean and median will be reported to 1 more decimal place than the raw data recorded in the database. The SD will be reported to 2 more decimal places than the raw data recorded in the database. In general, the maximum number of decimal places reported shall be 4 for any summary statistic.

Categorical data will be summarized in terms of the number of patients in the analysis population, the number of patients providing data at the relevant time point, frequency counts, and the percentages corresponding to the appropriate method. Percentages will be presented to 1 decimal place. Percentages will not be presented for zero counts.

Change from baseline will be calculated as the post-baseline value minus the baseline value. Percent change from baseline is defined as (100 x [post-baseline – baseline] / baseline). Percent improvement from baseline is calculated as the positive percent change from baseline if a higher value at postbaseline means improvement from baseline. Similarly, percent improvement from baseline is calculated as the negative percent change from baseline if a lower value at postbaseline means improvement from baseline.

Data collected at ETVs will be mapped to the next planned visit number for that patient. For by-visit and by-treatment-week summaries, only visits in which a measure was scheduled to be collected will be summarized. Unplanned/unscheduled measurements will be excluded from the mixed-effects model of repeated measures (MMRM) analysis. However, the data will still be used in other analyses as indicated in the SAP. Such analyses will include, but are not limited to, shift analyses and change from baseline to last-observation (e.g., mBOCF) endpoint analyses.

All confidence intervals (CIs) and statistical tests will be 2-sided with an  $\alpha$  level of 0.05 unless otherwise specified. P-values that are greater than or equal to 0.001, and less than or equal to 0.999, will be presented to 3 decimal places. All other p-values which are less than 0.001 will be presented as <0.001, while p-values greater than 0.999 will be presented as >0.999. Confidence intervals will be presented to one more decimal place than the raw data.

Age, sex, and race will be reported on all by-patient listings unless otherwise specified. Sex will be abbreviated as follows: female (F) and male (M). Race will be abbreviated as follows: American Indian or Alaska Native (AI), Asian (AS), Black or African American (BL), Native Hawaiian or other Pacific Islander (NH), White (WH), and Multiple (MU).

# 6.1.1. General Considerations for Analyses during Period 2 (Initial Open-Label Treatment Period)

#### 6.1.1.1. Initial Open-Label Treatment Period Population

Efficacy, health outcomes, and safety data collected in Period 2 will be summarized for ixekizumab 80 mg Q2W without inferential statistics.

Baseline for Period 2 is defined as the last available value on or before the first injection of ixekizumab 80 mg Q2W in Period 2 and in most cases will be the value recorded at Week 0 (Visit 2). For patients who do not take any injections of ixekizumab 80 mg Q2W in Period 2, the last available value prior to Week 0 (Visit 2) will be their baseline. The baseline period is defined as the start of screening and ends prior to the first injection of ixekizumab 80 mg Q2W at Week 0 (Visit 2). If the date of first injection is missing, the date of Visit 2 will be used.

Period 2 starts at the time of first injection of ixekizumab 80 mg Q2W (or after the date of Visit 2, if the date of first injection is missing) and ends for the following study events:

- Prior to the first injection of study treatment in the randomized double-blind withdrawal period (Period 3) for patients who meet the randomization criteria,
- Week 64 (Visit 19) for patients who do not meet the randomization criteria, or
- Visit of early discontinuation of study treatment in the initial open-label treatment.

Kaplan-Meier estimates will be used to estimate the survival curve for time-to variables.

For longitudinal continuous and categorical efficacy and health outcome variables, summaries will be performed by treatment week through the last observation during the study period. The last observation is defined as the value reported for the last visit prior to the first injection of randomized study treatment for patients who randomize or the value reported for Week 64 (Visit 19) for patients who do not meet randomization criteria or the last observation prior to discontinuation for patients who discontinue early.

# 6.1.2. General Considerations for Analyses during Period 3 (Randomized Double-Blind Withdrawal Period)

# 6.1.2.1. Randomized Withdrawal ITT and Randomized Withdrawal Safety Populations

Efficacy, health outcomes, and safety data collected in Period 3 will be summarized and treatment group comparisons (ixekizumab 80 mg Q2W versus placebo) will be performed for randomized patients.

Period 3 starts at the first injection of study treatment after randomization (or at randomization if missing the first injection of study treatment) and ends at the following study events:

- Relapse (no longer meeting Coates criteria for MDA),
- Week 104 (Visit 29) for patients who do not relapse, or

• Visit of early discontinuation of study treatment in the randomized double-blind withdrawal period.

For the efficacy and health outcome analyses, baseline is defined as the last available value on or before the first injection of study treatment in Period 2 and in most cases will be the value recorded at Week 0 (Visit 2). If the date of first injection is missing, the date of Week 0 (Visit 2) will be used. For the safety analysis, baseline is defined as the last available value on or before the first injection of randomized study treatment in Period 3. If the date of first injection is missing, the date of randomization will be used.

The Kaplan-Meier product limit method will be used to estimate the survival curves for time-to variables. Treatment comparisons will be performed using a log-rank test with treatment, geographic region, and cDMARD use (past use, current use) at the time of randomization in Period 3, in the model. Time-to analyses will be calculated in weeks from the date of first injection on the randomized study treatment in Period 3 (see Section 6.11.1).

For longitudinal continuous and categorical efficacy and health outcome variables, the analysis will be summarized by randomized treatment week through 40 weeks of randomized treatment. For the proportion of patients who relapse, additional descriptive summaries will be provided by randomized treatment week beyond 40-week without inferential statistics.

The primary analysis of the categorical efficacy and health outcome variables will use a logistic regression with treatment, geographic region, and cDMARD use (past use, current use) at the time of randomization in Period 3, in the model. Secondary analysis of the categorical efficacy and health outcome variables will be conducted using the Fisher's exact test. In general, missing data will be imputed using the nonresponder imputation (NRI) method. For relapse analysis, the cumulative relapse will be provided at each randomized treatment week and is defined as a relapse on or before the randomized treatment week or a study treatment discontinuation. If a patient has missing components for Coates criteria for MDA that results in missing MDA at a particular visit, the patient will not be considered as relapse.

The primary analyses for all continuous efficacy and health outcome variables, change from baseline to endpoint, and percent improvement from baseline analyses, will be made using MMRM. Secondary analyses will be performed using an analysis of covariance (ANCOVA) model.

The MMRM includes treatment group, baseline measure, geographic region, cDMARD use (past use, current use), treatment week, baseline measure-by-treatment week interaction term, and treatment week-by-treatment interaction term as fixed factors. The covariance structure to model the within-patient errors will be unstructured. If the unstructured covariance matrix results in a lack of convergence, the heterogeneous Toeplitz covariance structure, followed by the heterogeneous autoregressive covariance structure will be used. The Kenward-Roger method will be used to estimate the denominator degrees of freedom. For each treatment comparison performed, the least squares (LS) mean for each treatment group, an estimate of the difference between treatments, corresponding 95% CI and p-value will be presented. The estimate, 95% CI, and p-value for the overall difference between treatments over Period 3 will also be presented

for each treatment comparison. Type III tests for the LS means will be used for the statistical comparison.

The ANCOVA model includes treatment as a factor and baseline value, geographic region, and cDMARD use (past use, current use) as covariates. Missing data will be imputed using the mBOCF. Type III sums of squares for the LS means will be used for the statistical comparison. For each treatment comparison performed, the LS mean for each treatment group, an estimate of the difference between treatments, corresponding 95% CI and p-value will be presented. Type III sums of squares for the LS means will be used for the statistical comparison.

The Fisher's exact test will be used for all adverse event (AE), baseline, discontinuation, and other categorical data. Adverse event data will be analyzed using exposure-adjusted incidence rates (per 100 patient years). Summary tables comparing exposure-adjusted incidence rate (that is, person-time-adjusted incidence rates) over the entire time period will be generated where total number of patients who experienced the TEAE for each PT will be divided by the sum of all patients' time (in 100 years) of exposure during the treatment period. The entire time on study during the treatment period will be used instead of the time up to the first event (for those patients that have an event) due to implementation and display considerations. These tables will include the total number of patients in each treatment group, the total person years, the incidence rate ([number of patients with the event / total person years]\*100), the relative risk (all ixekizumab in numerator), and p-value. Both the relative risk and p-value will be derived from a Poisson regression model with treatment as explanatory variable. The p-value will be based on the likelihood ratio test. Statistical comparisons will be applied at each MedDRA level (that is, SOC, and PT).

Continuous vital sign and laboratory values will be analyzed by an ANCOVA model with treatment and baseline value as independent variables. Other continuous variables will be analyzed by t-tests unless otherwise stated.

#### 6.1.2.2. Relapse Population

For patients who randomize and subsequently relapse in Period 3, efficacy, health outcomes, and safety data collected between relapse and the end of Period 3 will be summarized by the randomized treatment group (ixekizumab 80 mg Q2W or Placebo) without inferential statistics for the relapse period.

For the efficacy and health outcomes analyses, baseline is defined as the last available value on or before the initial first injection of ixekizumab 80 mg Q2W in Period 2 and in most cases will be the value recorded at Week 0 (Visit 2). If the date of first injection is missing, the date of Visit 2 will be used. For the safety analysis, baseline is defined as the last available value on or before relapse in Period 3.

The relapse period, for the relapse population, starts at the time of first injection of ixekizumab 80 mg Q2W following relapse and ends on the date of Week 104 (Visit 29) or the visit of early discontinuation.

A subset of the efficacy and health outcomes (refer to Section 6.11.2) will be summarized after the re-treatment of ixekizumab 80 mg Q2W for:

- the relapse population
- the relapse population who, following relapse, were re-treated with ixekizumab 80 mg Q2W after relapse for at least 16 weeks.

Categorical safety measures will be summarized with incidence rates.

For longitudinal continuous and categorical efficacy and health outcome variables, summaries will be performed by treatment week through the last observation during the study period. The last observation is defined as the value reported for Week 104 (Visit 29) or the last observation prior to discontinuation for patients who discontinue early.

# 6.1.3. General Considerations for Analyses during Period 2 and Period 3 Combined (Initial Open-Label Treatment and Randomized Double-Blind Withdrawal Periods)

# 6.1.3.1. Ixekizumab 80 mg Q2W-Treated Patients from the Randomized Withdrawal ITT Population

For patients who are randomized in Period 3, efficacy, health outcomes, and safety data collected in Period 2 and Period 3 combined will be summarized for ixekizumab 80 mg Q2W without inferential statistics.

For efficacy, health outcomes, and safety analyses, baseline is defined as the last available value on or before the first initial injection of ixekizumab in Period 2 and in most cases will be the value recorded at Week 0 (Visit 2). If the date of first injection is missing, the date of Visit 2 will be used.

For patients who are randomized in Period 3, the combined Period 2 and Period 3 will start after the first initial injection of ixekizumab 80 mg Q2W in Period 2 (or after the date of Visit 2, if the date of first injection is missing) and ends at the following study events:

- Relapse (no longer meeting Coates criteria for MDA),
- Week 104 (Visit 29) for patients who do not relapse, or
- Visit of early discontinuation of study treatment in the randomized double-blind withdrawal period.

That is, Period 2 and Period 3 combined will end prior to the first injection of placebo for patients who randomize to placebo in Period 3.

A subset of the efficacy and health outcomes (refer to Section 6.11.2) will be summarized.

Categorical safety measures will be summarized with incidence rates.

For longitudinal continuous and categorical efficacy and health outcome variables, summaries will be performed by treatment week through the last observation during the study period. The last observation is defined as follows:

- the value reported for the last visit prior to the first injection of placebo for patients who randomize to placebo in Period 3,
- the value reported for the relapse visit for patients randomized to ixekizumab 80 mg Q2W and who relapse,
- the value reported at Week 104 (Visit 29) for patients randomized to ixekizumab 80 mg Q2W and who do not relapse, or
- the last observation prior to discontinuation for patients who discontinue early and for patients who do not relapse.

#### 6.1.3.2. Nonrandomized Population

For patients who are not randomized in Period 3, efficacy, health outcomes, and safety data collected in Period 2 and Period 3 combined will be summarized for ixekizumab 80 mg Q2W without inferential statistics.

For efficacy, health outcomes, and safety analyses, baseline is defined as the last available value on or before the first injection of ixekizumab 80 mg Q2W in Period 2 and in most cases will be the value recorded at Week 0 (Visit 2). If the date of first injection is missing, the date of Visit 2 will be used.

Period 2 and Period 3 combined, for the nonrandomized patients, starts at the first injection of ixekizumab 80 mg Q2W in Period 2 (or after the date of Visit 2, if the date of first injection is missing) and ends at the following study events: Week 104 (Visit 29) or Visit of early discontinuation of study treatment in the Initial Open-Label Treatment period or randomized double-blind withdrawal period.

A subset of the efficacy and health outcomes (refer to Section 6.11.2) will be summarized.

Categorical safety measures will be summarized with incidence rates.

For longitudinal continuous and categorical efficacy and health outcome variables, summaries will be performed by treatment week through the last observation during the study period. The last observation is defined as the value reported for Week 104 (Visit 29) or the last observation prior to discontinuation for patients who discontinue early.

# 6.1.4. General Considerations for Analyses during Period 4 (Post-Treatment Follow-up Period)

Safety data collected in Period 4 will be summarized by treatment group without inferential statistics. Patients will be analyzed according to the treatment they were taking before entering Period 4

Baseline is defined as the last available value on or before entering Period 4. Period 4 starts at Visit 801 and ends at the last visit prior to study discontinuation.

Categorical safety measures will be summarized with incidence rates.

#### **6.2.** Adjustments for Covariates

The randomization at the beginning of the Period 3 (randomized double-blind withdrawal period) is stratified by geographic region and cDMARD use (past use, current use) at the time of randomization in Period 3. Unless otherwise specified, all categorical efficacy and health outcome analyses during Period 3 on the randomized withdrawal intent-to-treat (ITT) population will include geographic region in the analysis model. Unless otherwise specified, all continuous efficacy and health outcome analyses during Period 3 on the randomized withdrawal ITT population will include geographic region and cDMARD use (past use, current use) at the time of randomization in Period 3, in the analysis model.

In general for Period 3, when an MMRM is to be used for analyses, baseline value, and baseline-by-treatment week interactions will be included as covariates; when an ANCOVA is to be used for analyses, baseline value will be included as a covariate.

## 6.3. Handling of Dropouts or Missing Data

# 6.3.1. Nonresponder Imputation (NRI) for Clinical Response

For secondary analyses assessed during Period 3, patients will be considered a nonresponder for the NRI analysis if they do not meet the clinical response criteria or have missing clinical response data at any specified analysis time point. All nonresponders at any specified time point as well as all patients who discontinue study treatment before the specified analysis time point, for any reason, will be defined as a nonresponder for the NRI analysis. Patients without at least 1 observation on study treatment will also be defined as a nonresponder for the NRI analysis. The NRI analyses will be performed on categorical efficacy and health outcome variables.

# 6.3.2. Modified Baseline Observation Carried Forward (mBOCF)

A mBOCF analysis for Period 3 through 40 weeks of randomized treatment will be performed on all continuous efficacy and health outcome variables. In this approach the baseline observation will be carried forward to the corresponding endpoint for evaluation for patients who discontinue study treatment due to an AE or death. The last non-missing observation before discontinuation of study treatment will be carried forward to the corresponding primary endpoint for evaluation for patients who discontinue study treatment for any reason other than due to an AE. Patients without at least 1 post-baseline observation will not be included for evaluation with the exception of patients who discontinue study treatment due to an AE.

Period 2, combined periods 2 and 3, and Relapse Period summaries will also include a mBOCF summary. Summaries will be performed on all continuous efficacy and health outcome variables.

#### 6.4. Multicenter Studies

This study will be conducted by multiple investigators at multiple sites internationally. The countries will be categorized into geographic regions, as described in Table RHBF.6.1, for analysis.

Table RHBF.6.1. Geographic Regions

| Geographic Region | Country |
|---|---|
| Africa | South Africa |
| Central America | Mexico |
| North America | United States |
| Eastern Europe | Bulgaria, Czech Republic, Estonia, Poland, Russia, Slovak Republic, and Ukraine |
| Western Europe | Spain and United Kingdom |

Unless otherwise specified, the statistical analysis models will adjust for geographic region at the time of randomization.

For analysis of the primary endpoint, the presence of a treatment-by-region interaction will be tested at 10% significance level for the randomized withdrawal ITT population. Where there is evidence of an interaction (p<.10), descriptive statistics will be used to assess whether the interaction is quantitative (that is, the treatment effect is consistent in direction but not the size of effect is not consistent) or qualitative (the treatment is beneficial for some but not other regions).

#### 6.5. Multiple Comparisons/Multiplicity

There will be no adjustment for multiple comparisons in this study.

# 6.6. Use of an "Efficacy Subset" of Patients

The per protocol set (PPS) is defined below in Section 6.6.1 and is an Efficacy Subset of patients. Analysis details for the PPS can be found in Section 6.11.1.

# 6.6.1. Analysis Populations

Unless otherwise specified, efficacy, health outcomes, and safety summaries for Period 2 (initial open-label treatment period) will be conducted on the **initial open-label treatment period population**, defined as all patients who receive at least 1 injection of ixekizumab in Period 2. Efficacy and health outcomes analyses for Period 3 (randomized double-blind withdrawal period) will be conducted on the **randomized withdrawal intent-to-treat (ITT) population**, defined as all randomized patients, even if the patient does not receive the correct treatment or otherwise does not follow the protocol. Patients will be analyzed according to the treatment to which they were assigned.

The primary analyses will be repeated using the **PPS**. The PPS is defined as patients included in the randomized withdrawal ITT population who are compliant with therapy, who do not have significant protocol deviations (refer to Section 6.17), and whose investigator's site did not have significant good clinical practice (GCP) issues that occurred during the randomized, double-blind withdrawal period which would require reporting to regulatory agencies. Compliance with

therapy is defined to be missing no more than 20% of expected doses and not missing 2 consecutive doses (all injections at a visit are counted as 1 dose) during the randomized double-blind treatment period. Patients will be analyzed according to the treatment to which they were assigned.

Safety analyses for Period 3 will be conducted on the **randomized withdrawal safety population**, defined as all randomized patients who receive at least 1 injection of study treatment after randomization. Patients will be analyzed according to the treatment to which they were assigned.

Efficacy and health outcomes summaries for Period 2 and Period 3 combined will be conducted on the **Ixekizumab 80 mg Q2W-Treated Patients: Nonrandomized Population and Randomized Withdrawal ITT Population**, defined as all patients who were not randomized and who receive at least 1 injection of ixekizumab and all randomized patients who receive at least 1 injection of study treatment after randomization, respectively.

Safety summaries for Period 2 and Period 3 combined will be conducted on the **Ixekizumab 80 mg Q2W-Treated Patients: Nonrandomized Population and Randomized Withdrawal Safety Population**, defined as all patients who were not randomized and who receive at least 1 injection of ixekizumab and all randomized patients who receive at least 1 injection of study treatment after randomization, respectively. Efficacy, health outcomes, and safety summaries will be conducted on the **relapse population**, defined as all randomized patients who relapsed (no longer met Coates criteria for MDA) after randomization and who receive at least 1 injection of ixekizumab after relapse.

Safety analyses for Period 4 (post-treatment follow-up period) will be conducted on the **follow-up period population**, defined as all patients who receive at least 1 injection of study treatment at any time during Period 2 and Period 3 and have entered the post-treatment follow-up period. Patients will be analyzed according to the treatment they were taking before entering Period 4.

# 6.7. Patient Disposition

Patient flow will be summarized from entered to randomized to completion.

Analysis populations will be listed and summarized by treatment group for all entered patients.

Patient disposition from study and study treatment will be listed for all entered patients.

Patient disposition from study treatment will be summarized with reasons for disposition for:

- Period 2 (initial open-label treatment period population),
- Period 3 (randomized withdrawal ITT population),
- Relapse period (relapse population), and
- Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal ITT population, and nonrandomized population).

Patient disposition for Period 3 will be compared between treatment groups using the Fisher's exact test for the randomized withdrawal ITT population.

Patient disposition from study treatment by visit will be summarized with reasons for:

• Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal ITT population, and nonrandomized population).

Patient disposition from study by visit will be summarized with reasons for disposition for:

• Period 4 (post-treatment follow-up period population).

Time-to study treatment discontinuation due to an AE (in weeks) will be summarized by treatment group and graphically presented using Kaplan-Meier technique. The log-rank test will be used to compare time-to study treatment discontinuation between treatment groups for randomized withdrawal ITT population.

Time-to study treatment discontinuation will be calculated as:

$$\frac{\textit{Date of study treatment discontinuation} - \textit{Date of first injection} + 1}{7}$$

The date of first injection varies across the period and the analysis populations. Table RHBF.6.2 defines the date of first injection for each period and analysis population.

Table RHBF.6.2. Date of First Injection by Period and Analysis Population

| Period | Analysis Population | Date of First Injection |
|---|---|---|
| Period 2 | initial open-label treatment population | date of the first injection of ixekizumab<br>80 mg Q2W in Period 2 |
| Period 3 | randomized withdrawal ITT population | date of the first injection of study treatment after randomization in Period 3 |
| Relapse Period | relapse population | date of the first injection of ixekizumab 80 mg Q2W after relapse |
| Combined Periods 2 and 3 | ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal IIT population | date of the first injection of ixekizumab<br>80 mg Q2W in Period 2 |
| Combined Periods 2 and 3 | nonrandomized population | date of the first injection of ixekizumab<br>80 mg Q2W in Period 2 |

Abbreviations: ITT = intent-to-treat; Q2W = every 2 weeks.

Patient allocation by region, country, and center/site will be summarized with number of patients who entered the study, number of patients who entered the initial open-label treatment period, number of patients discontinued from study treatment, and number of patients discontinued from study.

#### 6.8. Patient Characteristics

Patient characteristics will be listed for all entered patients and summarized for the following populations:

- initial open-label treatment period population
- randomized withdrawal ITT population
- relapse population
- nonrandomized population

The continuous variables will be summarized using descriptive statistics and the categorical variables will be summarized using frequency counts and percentages.

For the randomized withdrawal ITT population, comparisons between treatment groups will be conducted using an analysis of variance (ANOVA) model with treatment group as a factor for continuous data, and using the Fisher's exact test for categorical data. (For categorical variables that have more than 2 categories, Monte Carlo estimates of exact p-values will be used.)

The following patient characteristics will be summarized:

• Age (in years): calculated using an imputed date of birth of July 1 in the year of birth collected in the electronic case report form (eCRF). Age will be calculated as:

```
Age = floor((intck('month', brthdtc, rfstdtc) - (day(rfstdtc) < day(brthdtc)))/12)
where brthdtc = Imputed date of birth, and rfstdtc = patient reference start date (that is, the date when patient is first exposed to study treatment)
```

- Age group: <65 years,  $\ge65$  years to <75 years,  $\ge75$  years
- Age group: <40 years,  $\ge40$  years
- Gender
- Age groups within gender
- Race: AI, AS, BL, NH, WH, MU
- Ethnicity: Hispanic or Latino, Not Hispanic or Latino, Not Applicable
- Country: South Africa, Mexico, Bulgaria, Czech Republic, Estonia, Poland, Russia, Slovak Republic, Ukraine, United States (US), Spain, and United Kingdom (UK)
- Geographic region: Europe, US, Rest of the World
- Geographic region:
  - o Africa (South Africa)
  - o Central America (Mexico)
  - o North America (US)

- Eastern Europe (Bulgaria, Czech Republic, Estonia, Poland, Russia, Slovak Republic, and Ukraine)
- Western Europe (Spain and UK)
- Geographic region at the time of randomization for the randomized withdrawal ITT population:
  - o Africa (South Africa)
  - o Central America (Mexico)
  - o North America (US)
  - o Eastern Europe (Bulgaria, Czech Republic, Estonia, Poland, Russia, Slovak Republic, and Ukraine)
  - Western Europe (Spain and UK)
- Height (cm): last non-missing result before first study treatment injection
- Weight (kg): last non-missing result before first study treatment injection
- Weight category: <100 kg, ≥100 kg
- Weight category:  $<80 \text{ kg}, \ge80 \text{ kg}$  and  $<100 \text{ kg}, \ge100 \text{ kg}$
- Body mass index (BMI) (kg/m<sup>2</sup>): BMI will be calculated as:

$$BMI (kg / m^2) = \frac{Weight (kg)}{(Height (m))^2}$$

- BMI category: underweight (<18.5 kg/m²); normal (≥18.5 and <25 kg/m²); overweight (≥25 and <30 kg/m²); obese (≥30 and 40 kg/m²); extreme obese (≥40 kg/m²)
- Waist circumference (cm)
- Alcohol use: never, current, former
- Caffeine use: never, current, former
- Tobacco use: never, current, former
- Number of pipefuls, cigarettes, cigars, and smokeless (pinches) tobacco consumed per day
- Time since PsA onset (years) calculated as

$$(date\ of\ informed\ consent-date\ of\ PsA\ onset+1)/365.25$$

Patients who have a completely missing date of onset will have a missing value for the time since PsA onset, otherwise, "January" and "01" will be imputed for the missing month and day respectively in cases where these 2 date components are missing.

• Time since PsA diagnosis (years) – calculated as

Patients who have a completely missing date of diagnosis will have a missing value for the time since diagnosis, otherwise "January" and "01" will be imputed for the missing month and day respectively in cases where for these 2 date components are missing.

• Time since plaque psoriasis (Ps) onset (years) – calculated as

```
(date of informed consent – date of Ps onset + 1) / 365.25
```

Patients who have a completely missing date of onset will have a missing value for the time since Ps onset, otherwise, "January" and "01" will be imputed for the missing month and day respectively in cases where these 2 date components are missing.

• Time since Ps diagnosis (years) – calculated as

```
(date of informed consent – date of Ps diagnosis + 1) / 365.25
```

Patients who have a completely missing date of diagnosis will have a missing value for the time since diagnosis, otherwise "January" and "01" will be imputed for the missing month and day respectively in cases where for these two date components are missing.

- Previous cDMARD use (none, past use, current use) for:
  - o methotrexate (MTX)
  - o sulfasalazine (SSZ)
  - o leflunomide (LEF)
  - hydroxychloroquine (HCQ)
  - o cyclosporine (CSA)
  - o apremilast
- Previous cDMARD use (past use, current use)
- Previous cDMARD use at the time of randomization for the randomized withdrawal ITT and safety populations:
  - o Previous cDMARD use (yes, no) for:
    - methotrexate
    - sulfasalazine
    - leflunomide
    - hydroxychloroquine
    - cyclosporine
    - apremilast
  - Previous cDMARD use; yes or no

- Methotrexate dose at baseline (weekly)
- Methotrexate dose at the time of randomization for the randomized withdrawal ITT and safety populations
- Tender joint count (TJC) based on 68 joints
- Swollen joint count (SJC) based on 66 joints
- Physician's global assessment of disease activity (mm)
- Patient's global assessment of disease activity (mm)
- Patient's assessment of joint pain (mm)
- Health Assessment Questionnaire–Disability Index total score
- C-reactive protein (mg/L)
- C-reactive protein categories; >6 mg/L or ≤6 mg/L
- classification for psoriatic arthritis (CASPAR) total score (see Appendix 1 for additional details)
- Rheumatoid Factor Positive (RF+); yes or no
- Anti-cyclic citrullinated peptide positive (Anti-CCP +); yes or no
- Disease Activity Score modified to include the 28 diarthrodial joint count, based on C-reactive protein
- Enthesitis (based on 18 point entheseal point assessment); yes or no
- Enthesitis (Spondyloarthritis Research Consortium of Canada [SPARCC] >0); yes or no
- Spondyloarthritis Research Consortium of Canada for patients with baseline Enthesitis (SPARCC>0)
- Enthesitis (Leeds Enthesitis Index [LEI]>0); yes or no
- Leeds Enthesitis Index for patients with baseline enthesitis (LEI >0)
- Dactylitis (as reported on the eCRF); yes or no
- Dactylitis (Leeds Dactylitis Index Basic [LDI-B] >0); yes or no
- Leeds Dactylitis Index Basic for patients with baseline dactylitis (LDI-B >0)
- Modified CPDAI without the spinal disease assessment (Ankylosing Spondylitis Quality of Life Questionnaire [AsQoL] and Bath Ankylosing Spondylitis Disease Activity Index [BASDAI])
- Psoriasis Area and Severity Index (PASI) total score for patients who have baseline plaque psoriasis (PASI >0)
- Psoriasis Area and Severity Index total score for patients who have baseline psoriatic lesion(s) involving BSA ≥3%

- Psoriasis Area and Severity Index total score ≥12 for patients who have baseline plaque psoriasis (PASI >0); yes or no
- Psoriasis Area and Severity Index total score ≥12 for patients who have baseline psoriatic lesion(s) involving BSA ≥3%: yes or no
- Static Physician Global Assessment (sPGA) score for patients who have baseline plaque psoriasis (sPGA >0)
- Static Physician Global Assessment ≥3 for patients who have baseline plaque psoriasis (sPGA >0); yes or no
- Moderate to severe psoriasis (defined as PASI ≥12, sPGA ≥3, and BSA ≥10%); yes or no
- Percentage of BSA for patients who have baseline plaque psoriasis (BSA >0)
- Body surface area  $\ge 3\%$ ; yes or no for patients with baseline plaque psoriasis (BSA > 0)
- Body surface area ≥10%; yes or no for patients with baseline plaque psoriasis (BSA >0)
- Itch NRS score for patients who have baseline psoriatic lesion(s) involving BSA >3%
- Fatigue Severity NRS score
- Quick Inventory of Depressive Symptomatology-self report 16 items total score
- Medical Outcomes Study 36-Item Short Form Health Survey PCS score
- Medical Outcomes Study 36-Item Short Form Health Survey MCS score
- Dermatology Life Quality Index total score for patients who have baseline psoriatic lesion(s) involving BSA ≥3%
- Latent tuberculosis (TB); yes or no.

# 6.8.1. Previous Therapy for Psoriatic Arthritis

The number and percentage of patients who received previous therapy for PsA (as recorded on the *Previous Therapy: Psoriatic Arthritis* eCRF page) will be summarized by treatment group, overall and Preferred Term (PT). The number and percentage of patients with each reason for discontinuing previous therapy for PsA will also be presented by treatment group.

Previous therapy for PsA will be summarized for the following populations:

- initial open-label treatment period population
- randomized withdrawal ITT population
- nonrandomized population

Treatment group comparisons for the randomized withdrawal ITT population will be conducted using the Fisher's exact test.

Listing of previous therapy for PsA will be provided for the initial open-label treatment period population.

## 6.8.2. Historical Illness and Preexisting Conditions

Historical illnesses and preexisting conditions will be classified using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) dictionary. Preexisting conditions for the Open-label Treatment Period (Period 2) are defined as those conditions recorded on the *Preexisting Conditions and AEs or the Historical Events* eCRF pages with a start date prior to the date of informed consent and no end date (that is, the event is ongoing) or an end date after the date of informed consent. Adverse events occurring prior to the date of first study injection will also be reported as preexisting condition for the open-label treatment period (Period 2). Preexisting conditions for subsequent treatment periods are defined as those preexisting conditions and AEs which are ongoing at the treatment period baseline. If a preexisting condition worsens in severity on or after date of informed consent, it will be considered an AE from the date of worsening onwards. Note that conditions with a partial or missing start date will be assumed to be "not preexisting" unless there is evidence, through comparison of partial dates, to suggest otherwise. Patients will only be counted once, regardless of how many conditions are included under the same System Organ Class (SOC) and PT.

The number and percentage of patients with historical illnesses and preexisting conditions will be provided by treatment group, overall and by SOC and PT for each treatment period.

Preexisting conditions will be summarized for the following periods and populations:

- initial open-label treatment period population;
- randomized withdrawal ITT population

Historical illnesses will be summarized for the following populations:

- initial open-label treatment period population
- randomized withdrawal ITT population
- nonrandomized population

Treatment group comparisons for randomized withdrawal ITT Population will be conducted using Fisher's exact test.

Listing of historical illnesses and preexisting conditions will be provided for initial open-label treatment period population.

# 6.9. Treatment Compliance

The randomization schedule will be listed by center for the randomized withdrawal ITT population. Study treatment dispensed will be listed (including the clinical trial [CT] Lot

number) for all entered patients. Study treatment administration and compliance will be listed for all entered patients.

Throughout Period 2 and Period 3, patients will record information in a Study Drug Administration Log (captured in the *Exposure* eCRF page), including the date, time, and anatomical location of administration of investigational product, syringe number, who administered the investigational product, and the reason if the investigational product was not fully administered.

Treatment compliance (%) for each patient will be calculated as:

$$100 \times \frac{Total\ number\ of\ injections\ administered}{Total\ number\ of\ injections\ prescribed}$$

- o Number of injections prescribed (that is, expected) will be calculated as:
  - For Period 2:

$$2 + \frac{Number\ of\ weeks\ in\ the\ study\ period}{2}$$

• For Period 3:

$$\frac{Number\ of\ weeks\ in\ the\ study\ period}{2}$$

Note that the number of injections dispensed will vary across patients for each study period by analysis population, refer to Section 6.1 for the study period duration definitions by analysis populations.

Note there are 2 ixekizumab 80 mg injections at Week 0 and there is 1 ixekizumab 80 mg or placebo injection every 2 weeks, thereafter, starting at Week 2.

- For patients who discontinue during Period 2 or Period 3, the number of injections prescribed can be derived from the IWRS study drug dispense dataset.
- The total number of injections administered will be derived using the response to the question "Was dose administered?" on the Exposure eCRF page.

A patient will be considered overall compliant for Period 2 or Period 3 if he/she is missing no more than 20% of the expected doses, does not miss 2 consecutive doses, and does not over-dose (that is, take more injections at the same time point than specified in the protocol) within the respective study period.

Treatment compliance with investigational product will be summarized for the following periods:

- Period 2 (initial open-label treatment period population)
- Period 3 (randomized withdrawal safety population)

Treatment group comparisons will be conducted for Period 3 for the randomized withdrawal safety population using the Fisher's exact test.

## 6.10. Concomitant Therapy

Previous therapy is defined as therapy that starts and ends before the first day of study treatment in Period 2.

Concomitant therapy for each treatment period (Period 2, Period 3, and Period 2 and Period 3 combined) is defined as the therapy that starts before, on, or after the first day of study treatment in the treatment period and before the last visit date in the treatment period, and has either no end date (the therapy is ongoing) or an end date on or after the first day of study treatment in the treatment period. Notice, concomitant therapy will belong to a period if the therapy starts and ends on the exact same day as the first day of study treatment in the study period.

Concomitant therapy for the post-treatment follow-up period (Period 4) is defined as the therapy that starts before, on, or after the last visit date of Period 3 or ETV and continues into Period 4, that is, either no end date (the therapy is ongoing) or an end date after the last visit date of Period 3 or ETV.

The following summaries will be provided:

- Previous therapy by World Health Organization (WHO) Anatomical Therapeutic Chemical (ATC) Level 4 and WHO PT
  - o Initial Open-Label Treatment Period Population
- Concomitant therapy by WHO ATC Level 4 and WHO PT for:
  - o Period 2 (initial open-label treatment period population)
  - o Period 3 (randomized withdrawal safety population)
  - o Relapse Period (relapse population)
  - Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population, and nonrandomized population).

Comparisons between treatment groups will be conducted for Period 3 for the randomized withdrawal safety population using the Fisher's exact test.

A by-patient listing of all prior and concomitant medications will be provided for the initial open-label treatment period population.

If a partial or completely missing medication start date/time or end date/time is present, the following imputation rules will be utilized in the analysis:

- For the start date:
  - o If year, month, and day are missing, then use the consent date.
  - o If either month or month and day are missing, then use January 1.
- o If only day is missing, impute the first day of the month.
- For the start time:
  - o Impute as 23:59.
- For the end date:
  - o If year, month, and day are missing, then use the patient's last visit date.
  - o If either month or month and day are missing, then use December 31.
  - o If only day is missing, then use the last day of the month.
  - The imputed date will not be beyond the patient's last visit date.
- For the end time:
  - o Impute as 23:59.
- If there is any doubt, the medication will be flagged as concomitant.

## 6.11. Efficacy Analyses

Table RHBF.6.3 includes the description and derivation of the primary and secondary efficacy outcomes.

Table RHBF.6.4 provides the detailed analyses including analysis type, method and imputation, population, time point, and comparisons for primary and secondary efficacy analyses.

 Table RHBF.6.3.
 Description and Derivation of Primary and Secondary Efficacy Outcomes

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| Coates Criteria for<br>Minimal Disease<br>Activity (MDA) | Uses a composite of 7 key outcome measures (includes PASI) used in PsA to encompass all of the domains of the disease to measure the overall state of a patients' disease (Coates et al. 2010; Coates and Helliwell 2010). | MDA Flag | Patients are classified as achieving MDA if they fulfill 5 of 7 outcome measures: 1. TJC ≤1 2. SJC ≤1 3. PASI total score ≤1 or BSA ≤3 4. patient pain VAS score of ≤15 5. patient global VAS score of ≤20 6. HAQ-DI score ≤0.5 7. tender entheseal points (of 18 entheseal points) ≤1 See Appendix 2 for complete details. | If the patient achieves MDA with the non- missing measures, then impute as achieving MDA; otherwise, the result is missing. |
| Modified Coates<br>Criteria for<br>Minimal Disease<br>Activity (MDA) | Uses a composite of 7 key outcome measures (includes sPGA) used in PsA to encompass all of the domains of the disease to measure the overall state of a patients' disease (Mease et al. 2013). | MDA-sPGA<br>Flag | Patients are classified as achieving MDA if they fulfill 5 of 7 outcome measures: 1. TJC ≤1 2. SJC ≤1 3. sPGA (0,1) or BSA ≤3 4. patient pain VAS score of ≤15 5. patient global VAS score of ≤20 6. HAQ-DI score ≤0.5 7. tender entheseal points (of 18 entheseal points) ≤1 See Appendix 2 for complete details. | If the patient achieves MDA with the non-missing measures, then impute as achieving MDA; otherwise, the result is missing. |
| Tender Joint Count (TJC) | The number of tender and painful joints will be determined by examination of 68 joints (34 joints on each side of the patient's body). The 68 joints to be assessed and classified as tender or not tender. | TJC total score | Adjusted sum of the pain/tenderness for all 68 joints: $\left(\frac{sum\ of\ the\ evaluable\ individual\ tender\ joints}{number\ of\ evaluable\ joints}\right) X\ 68$ See Appendix 3 for complete details. | If more than half<br>of the joints are<br>nonevaluable, the<br>total score will<br>be missing. |

| Measure<br>Swollen Joint | Description The number of swollen joints will be determined | Variable SJC total score | Derivation / Comment Adjusted sum of the pain/tenderness for all 66 | Imputation Approach if with Missing Components If more than half |
|---|---|---|---|---|
| Count (SJC) | by examination of 66 joints (33 joints on each side of the patient's body). The 66 joints to be assessed and classified as swollen or not swollen. | | joints. $ \left( \frac{sum\ of\ the\ evaluable\ individual\ swollen\ joints}{number\ of\ evaluable\ joints} \right) X\ 66 $ See Appendix 3 for complete details. | of the joint s are<br>nonevaluable, the<br>total score will<br>be missing. |
| Patient's<br>Assessment of Pain<br>Visual Analog<br>Scale (VAS) | Assesses the patient's current level of joint pain by marking a vertical tick on a 100-mm horizontal VAS. | Patient Pain<br>VAS | Range: 0 to 100 mm | Single item,<br>missing if<br>missing |
| Patient's Global<br>Assessment of<br>Disease Activity<br>Visual Analog<br>Scale (VAS) | Assesses the patient's overall assessment of his or her PsA activity by marking a 100-mm horizontal VAS. | Patient Global<br>VAS | Range: 0 to 100 mm 0 represents no disease activity 100 represents extremely active disease activity | Single item,<br>missing if<br>missing |
| Patient's Assessment of Physical Function Health Assessment Questionnaire— Disability Index (HAQ-DI) | Patient-reported standardized questionnaire that is commonly used in PsA total measure disease-associated disability (assessment of physical function). It consists of 24 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other daily activities | HAQ-DI score | Sum of the highest sub-category scores within 8 categories and adjusted for aids/devices and/or help from another person. See Appendix 4 for complete details. | The patient must have a score for at least 6 of the 8 categories. If there are <6 categories completed, a HAQ-DI will be missing |
| American College<br>of Rheumatology<br>Responder Index<br>(ACR) | ACR Responder Index: a composite of clinical, laboratory, and functional measures in PsA to assess relief of signs and symptoms; responses are presented as the minimal numeric disease assessment criteria. | ACR20 Flag ACR50 Flag ACR70 Flag | See Appendix 5 for details. | See Appendix 5 for details. |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| C-Reactive Protein (CRP) | The ACR Core Set measure of acute phase reactant. It will be measured with a high sensitivity assay at the central laboratory to help assess the effect of ixekizumab on the patient's PsA | <ul> <li>CRP (mg/L)</li> <li>Change from baseline in CRP (mg/L)</li> <li>% improvemen t in CRP (mg/L)</li> </ul> | Raw laboratory result, no derivation will be applied with the exception of converting the units to mg/L when the results are reported in units other than mg/L | Single lab<br>measure, missing<br>if missing |
| Static Physician<br>Global Assessment<br>(sPGA) | For patients with plaque psoriasis, the physician's global assessment of the patient's psoriasis (Ps) lesions at a given time point (European Medicines Agency [EMA] 2004 [WWW]). Plaques are assessed for induration, erythema, and scaling, and an overall rating of psoriasis severity is given. | sPGA score | Range from 0 to 5: clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). | Single item,<br>missing if<br>missing |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| Psoriasis Area and Severity Index (PASI) | For patients with plaque psoriasis, combines assessments of the extent of body-surface involvement in 4 anatomical regions (head and neck, trunk, arms, and legs) and the severity of scaling (S), redness (R), and plaque induration/infiltration thickness (T) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease (Fredriksson and Pettersson 1978). Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none 1 = slight 2 = moderate 3 = severe 4 = very severe The body is divided into 4 anatomical regions comprising the head (h), upper limb (u), trunk (t), and lower limb (l). In each of these areas, the fraction of total BSA affected is graded on a 0-6 scale (0 for no involvement; up to 6 for 90% - 100% involvement): 0 = 0% (clear) 1 = >0% to <10% 2 = 10% to <30% 3 = 30% to <50% 4 = 50% to <70% 5 = 70% to <90% 6 = 90% to 100% The various body regions are weighted to reflect | PASI total score | The composite PASI score is calculated by multiplying the sum of the individual-severity scores for each area by the weighted area-of-involvement score for that respective area, and then summing the 4 resulting quantities as follows: $PASI = 0.1(R_h + T_h + S_h)A_h + 0.2(R_u + T_u + S_u)A_u + 0.3(R_t + T_t + S_t)A_t + 0.4(R_l + T_l + S_l)A_l$ Where, $R_h, R_u, R_t, R_l = \text{redness score of plaques}$ on the head, upper limb, trunk, and lower limb, scored 0-4 respectively; $T_h, T_u, T_t, T_l = \text{thickness score of plaques}$ on the head, upper limb, trunk, and lower limb, scored 0-4 respectively; $S_h, S_u, S_t, S_l = \text{scaliness score of plaques}$ on the head, upper limb, trunk, and lower limb, scored 0-4 respectively; $A_h, A_u, A_t, A_l = \text{numerical value}$ translation of % area of psoriatic involvement score for the head, upper limb, trunk, and lower limb, respectively. $PASI \text{ scores are treated as a continuous score, with 0.1 increments within these values.}$ | If any individual score is missing, the PASI score will not be calculated, hence missing. |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| Percentage of Body<br>Surface Area | The investigator will evaluate the percentage involvement of psoriasis on each patient's BSA | BSA | Collected as a single scale. Range from 0% to 100%. | Single item,<br>missing if |
| (BSA) | on a continuous scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the patient's hand (including the palm, fingers, and thumb) (National Psoriasis Foundation [NPF] 2009). | | | missing |

Abbreviations: ACR20/50/70 = 20%, 50%, or 70% improvement in American College of Rheumatology criteria; PsA = psoriatic arthritis; PGA = static physician global assessment.

 Table RHBF.6.4.
 Description of Primary and Secondary Efficacy Analyses

| | | Analysis Method | Population | Comparison/Time | |
|---|---|---|---|---|---|
| Measure | Variable | (Section 6.1) | (Section 6.6.1) | Point | Analysis Type |
| Coates Criteria | Time-to achieve | Descriptive Statistics | Initial open-label treatment | Assessed Period 2 | Secondary analysis: |
| for Minimal | Coates criteria for | (including Kaplan Meier | period population | | 1. Time-to achieve |
| Disease | MDA | estimates of the survival | | | Coates criteria for |
| Activity | | curve) | | | MDA |
| (MDA) | | | | | 2. Time-to achieve |
| | | | | | Coates criteria for |
| | | | | | MDA for 3 |
| | | | | | consecutive months |
| | | | | | over 4 consecutive |
| | | | | | visits |
| | | | Relapse population | Assessed during | Secondary analysis: |
| | | | | Relapse Period | Time-to achieve Coates |
| | | | | | criteria for MDA |
| | | | Relapse population who have | Assessed during | Secondary analysis: |
| | | | completed 16 weeks on | Relapse Period | Time-to achieve Coates |
| | | | relapse treatment | | criteria for MDA for 3 |
| | | | | | consecutive months over |
| | | | | | 4 consecutive visits |
| | Proportion of patients | Descriptive Statistics | Initial open-label treatment | Assessed Period 2 | Secondary analysis |
| | achieving MDA | | period population | | |
| | | | Relapse population | Assessed during | Secondary analysis |
| | | | | Relapse Period | |
| | | | Relapse population who have | Assessed during | Secondary analysis |
| | | | completed 16 weeks on | Relapse Period | |
| | | | relapse treatment | | |
| | Time-to relapse (no | Log-Rank Test. Kaplan- | Randomized withdrawal ITT | Assessed during Period 3 | Primary analysis |
| | longer meeting Coates | Meier product limit method | population and PPS | | comparing IXE80Q2W |
| | criteria for MDA) | | | | vs. placebo (see Section |
| | | | | | 6.11.1) |

| | | Analysis Method | Population | Comparison/Time | |
|---|---|---|---|---|---|
| Measure | Variable | (Section 6.1) | (Section 6.6.1) | Point | Analysis Type |
| | Proportion of relapse patients | Logistic regression analysis and Fisher's exact test with cumulative rate Descriptive statistics | Randomized withdrawal ITT population | Assessed during Period 3 (by Treatment Week) through 40 weeks of randomized treatment, then descriptive beyond 40 weeks | Secondary analysis assessed during Period 3 |
| Modified<br>Coates Criteria<br>for Minimal<br>Disease<br>Activity | Time-to achieve<br>modified Coates<br>criteria for MDA | Descriptive statistics for IXE80Q2W | Initial open-label treatment period population | Assessed during Period 2 | Sensitivity analysis: 1. Time-to achieve Coates criteria for MDA 2. Time-to achieve Coates criteria for MDA for 3 consecutive months over 4 consecutive visits |
| | Time-to relapse of modified Coates criteria for MDA | Log-Rank Test. Kaplan-<br>Meier product limit method | Randomized withdrawal ITT population who met modified Coates Criteria for MDA at time of randomization | Assessed during Period 3 | Sensitivity analysis |
| | Proportion of relapse<br>patients of modified<br>Coates criteria for<br>MDA | Logistic regression (primary) and Fisher's exact test (secondary) with cumulative rate Descriptive statistics | Randomized withdrawal ITT population who met modified Coates Criteria for MDA at time of randomization | Assessed during Period 3<br>(by Treatment Week)<br>through 40 weeks of<br>randomized treatment,<br>then descriptive beyond<br>40 weeks | Sensitivity analysis |
| Tender Joint<br>Count (TJC) | Time-to TJC >1 (loss of response) | Log-Rank Test. Kaplan-<br>Meier product limit method | Randomized withdrawal ITT population who had TJC ≤1 at time of randomization | Assessed during Period 3 | Secondary analysis |
| | Time-to Achieve TJC ≤1 | Descriptive statistics<br>(including Kaplan Meier<br>estimates of the survival<br>curve) | Relapse population who had TJC >1 at time of relapse | Assessed during Relapse<br>Period | Secondary analysis |

| | | Analysis Method | Population | Comparison/Time | |
|---|---|---|---|---|---|
| Measure | Variable | (Section 6.1) | (Section 6.6.1) | Point | Analysis Type |
| Swollen Joint | Time-to SJC >1 (loss | Log-Rank Test. Kaplan- | Randomized withdrawal ITT | Assessed during Period 3 | Secondary analysis |
| Count (SJC) | of response) | Meier product limit method | population who had a SJC ≤1 at time of randomization | | |
| | Time-to SJC Achieve ≤1 | Descriptive statistics<br>(including Kaplan Meier<br>estimates of the survival<br>curve) | Relapse population who had a SJC >1 at time of relapse | Assessed during Relapse<br>Period | Secondary analysis |
| Patient's<br>Assessment of<br>Pain Visual<br>Analog Scale | Time-to Pain VAS<br>score >15 (loss of<br>response) | Log-Rank Test. Kaplan-<br>Meier product limit method | Randomized withdrawal ITT population who had a Pain VAS score ≤15 at time of randomization | Assessed during Period 3 | Secondary analysis |
| (VAS) | Time-to Achieve Pain<br>VAS score ≤15 | Descriptive statistics<br>(including Kaplan Meier<br>estimates of the survival<br>curve) | Relapse population who had<br>a Pain VAS score >15 at time<br>of relapse | Assessed during Relapse<br>Period | Secondary analysis |
| Patient's<br>Global Visual<br>Analog Scale<br>(VAS) | Time-to patient global<br>disease activity VAS<br>score >20 (loss of<br>response) | Log-Rank Test. Kaplan-<br>Meier product limit method | Randomized withdrawal ITT population who had a global disease activity VAS score ≤20 at time of randomization | Assessed during Period 3 | Secondary analysis |
| | Time-to Achieve patient global disease activity VAS score ≤20 | Descriptive statistics<br>(including Kaplan Meier<br>estimates of the survival<br>curve) | Relapse population who had<br>a global disease activity scale<br>VAS score >20 at time of<br>relapse | Assessed during Relapse<br>Period | Secondary analysis |

| | | Analysis Method | Population | Comparison/Time | |
|---|---|---|---|---|---|
| Measure | Variable | (Section 6.1) | (Section 6.6.1) | Point | Analysis Type |
| Patient's<br>Assessment of | Change from baseline in HAQ-DI total score | Descriptive statistics | Initial open-label treatment period population | Assessed during Period 2 | Secondary analysis |
| Physical<br>Function | Percent improvement | | Relapse population | Assessed during Relapse<br>Period | Secondary analysis |
| Health Assessment Questionnaire— Disability | in HAQ-DI total score | | Ixekizumab-treated patients:<br>nonrandomized population<br>and randomized withdrawal<br>ITT population | Assessed during Period 2 and Period 3 combined | Secondary analysis |
| Index (HAQ-<br>DI) | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3<br>through 40 Weeks of<br>Randomized Treatment | Secondary analysis |
| | HAQ-DI total score improvement ≥0.35 | Descriptive statistics | Initial open-label treatment period population - Patients with baseline HAQ-DI ≥0.35 | Assessed during Period 2 | Secondary analysis |
| | | | Relapse population- Patients with baseline HAQ-DI $\geq$ 0.35 | Assessed during Relapse<br>Period | Secondary analysis |
| | | | Ixekizumab-treated patients: nonrandomized population and randomized withdrawal ITT population- Patients with baseline HAQ-DI ≥0.35 | Assessed during Period 2 and Period 3 combined | Secondary analysis |
| | | Logistic regression analysis with NRI; Fisher's exact test with NRI | Randomized withdrawal ITT population | Assess during Period 3<br>through 40 weeks of<br>Randomized Treatment | Secondary analysis |
| | Time-to HAQ-DI<br>score >0.5 (loss of<br>response) | Log-Rank Test. Kaplan-<br>Meier product limit method | Randomized withdrawal ITT population who had a HAQ-DI score ≤0.5 at time of randomization | Assessed during Period 3 | Secondary analysis |
| | Time-to Achieve<br>HAQ-DI score ≤0.5 | Descriptive statistics<br>(including Kaplan Meier<br>estimates of the survival<br>curve) | Relapse population who had<br>a HAQ-DI score >0.5 at time<br>of relapse | Assessed during Relapse<br>Period | Secondary analysis |

| Measure | Variable | Analysis Method<br>(Section 6.1) | Population (Section 6.6.1) | Comparison/Time<br>Point | Analysis Type |
|---|---|---|---|---|---|
| American<br>College of | Time-to achieve<br>ACR20 | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 | Secondary analysis |
| Rheumatology<br>Responder<br>Index (ACR) | Time-to achieve<br>ACR50<br>Time-to achieve<br>ACR70 | (including Kaplan Meier estimates of the survival curve) | Ixekizumab-treated patients:<br>nonrandomized population<br>and randomized withdrawal<br>ITT population | Assessed during Period 2 and Period 3 combined | Secondary analysis |
| | Proportion of patients achieving ACR20 | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment population | Assessed during Period 2 | Secondary analysis |
| | Proportion of patients achieving ACR50 | | Ixekizumab-treated patients nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined | Secondary analysis |
| | Proportion of patients achieving ACR70 | Logistic regression analysis with NRI; Fisher's exact test with NRI | Randomized withdrawal ITT population | Assess during Period 3<br>through 40 weeks of<br>Randomized Treatment | Secondary analysis |
| C-Reactive<br>Protein (CRP) | CRP (mg/L) | Descriptive statistics | Initial open-label treatment period population | Assessed during Period 2 | Secondary analysis |
| | Change from baseline in CRP (mg/L) | | Relapse population | Assessed during Relapse<br>Period | Secondary analysis |
| | % improvement in CRP (mg/L) | | Ixekizumab-treated patients:<br>nonrandomized population<br>and randomized withdrawal<br>ITT population | Assessed during Period 2 and Period 3 combined | Secondary analysis |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3<br>through 40 weeks of<br>Randomized Treatment | Secondary analysis |
| Static<br>Physician's<br>Global<br>Assessment | Time-to sPGA ≥2 (loss of response) | Log-Rank Test. Kaplan-<br>Meier product limit method | Randomized withdrawal ITT population who were sPGA (0,1) at time of randomization | Assessed during Period 3 | Secondary analysis |

| | | Analysis Method | Population | Comparison/Time | |
|---|---|---|---|---|---|
| Measure | Variable | (Section 6.1) | (Section 6.6.1) | Point | Analysis Type |
| (sPGA) | Time-to Achieve<br>sPGA (0,1) | Descriptive statistics<br>(including Kaplan Meier<br>estimates of the survival<br>curve) | Relapse population who were sPGA ≥2 at time of relapse | Assessed during Relapse<br>Period | Secondary analysis |
| Psoriasis Area<br>and Severity<br>Index (PASI) | Time-to PASI total<br>score >1 (loss of<br>response) | Log-Rank Test. Kaplan-<br>Meier product limit method | Randomized withdrawal ITT population who were PASI total score ≤1 at time of randomization | Assessed during Period 3 | Secondary analysis |
| | Time-to Achieve PASI total score ≤1 | Descriptive statistics<br>(including Kaplan Meier<br>estimates of the survival<br>curve) | Relapse population who were PASI total score >1 at time of relapse | Assessed during Relapse<br>Period | Secondary analysis |
| Percentage of<br>Body Surface<br>Area (BSA) | Time-to-BSA >3% (loss of response) | Log-Rank Test. Kaplan-<br>Meier product limit method | Randomized withdrawal ITT population who were BSA ≤3% at time of randomization | Assessed during Period 3 | Secondary analysis |
| | Time-to Achieve BSA ≤3% | Descriptive statistics<br>(including Kaplan Meier<br>estimates of the survival<br>curve) | Relapse population who were BSA >3% at time of relapse | Assessed during Relapse<br>Period | Secondary analysis |
| Tender Entheseal Points (defined using the 18 | Time-to tender<br>entheseal points >1<br>(loss of response) | Log-Rank Test. Kaplan-<br>Meier product limit method | Randomized withdrawal ITT population who had a tender entheseal points ≤1 at time of randomization | Assessed during Period 3 | Secondary analysis |
| entheseal points) | Time-to Achieve tender entheseal points ≤1 | Descriptive statistics (including Kaplan Meier estimates of the survival curve) | Relapse population who had a tender entheseal points >1 at time of relapse | Assessed during Relapse<br>Period | Secondary analysis |

Abbreviations: ACR20/50/70 = 20%, 50%, or 70% improvement in American College of Rheumatology criteria; ANCOVA = analysis of covariance; ITT = intent-to-treat; IXE80Q2W = ixekizumab 80 mg every 2 weeks; mBOCF = modified baseline observation carried forward; MMRM = mixed-effects model of repeated measures; NRI = nonresponder imputation; PPS = per-protocol set; Q2W = every 2 weeks.

## 6.11.1. Primary Outcome and Methodology

The primary analysis is the time-to relapse (no longer meeting Coates criteria for MDA) for the randomized withdrawal ITT population. Time-to relapse will be calculated in weeks as follows:

(Date of Relapse - Date of First injection of Randomized study treatment in Period 3) + 1

7

If the date of first injection is missing, the date of randomization will be used. Patients completing Period 3 without relapsing will be censored at the date of completion (that is, the date of the last visit in the period). Patients without a date of completion or discontinuation for Period 3 will be censored at the latest non-missing date out of the following dates: date of last dose and date of last attended visit in Period 3.

Treatment comparison between ixekizumab 80 mg Q2W and placebo in time-to relapse for the randomized withdrawal ITT population and the PPS will be analyzed using a log-rank test with treatment, geographic region, and cDMARD use (past use, current use) at the time of randomization in Period 3, in the model. The Kaplan-Meier product limit method will be used to estimate the survival curves for time-to relapse. Time-to relapse will also be summarized graphically by treatment group using Kaplan-Meier techniques.

## 6.11.2. Secondary Efficacy Analyses

There will be no adjustment for multiple comparisons for other secondary analyses. The secondary analyses are detailed in Table RHBF.6.3 and Table RHBF.6.4.

## 6.11.3. Sensitivity Analyses

Sensitivity analyses will be performed for the primary analysis using the modified Coates criteria for MDA. For the modified criteria for MDA, sPGA "skin clear" or "skin almost clear" (as MDA-sPGA [0,1]) is substituted for PASI ≤1 (Mease et al. 2013). The modified Coates criteria for MDA is described in Table RHBF.6.3 and the sensitivity analyses are detailed in Table RHBF.6.4.

## 6.12. Bioanalytical and Pharmacokinetic/Pharmacodynamic Methods

Pharmacokinetic, PD, and biomarker analyses to address secondary and exploratory objectives of this study will be described by Lilly in separate PK/PD and biomarker analysis plans.

## 6.13. Safety Analyses

Safety will be assessed by summarizing and analyzing SAEs, AEs, AEsIs, QIDS-SR16, vital signs, other measures of cardiovascular function, laboratory evaluations (including chemistry, calculated creatinine clearance, hematology [including (WBC) count and differential], urinalysis [dipstick and microscopic], thyroid-stimulating hormone and free T4, and immunogenicity testing [TE-ADAs]).

Primary safety analyses will focus on comparison of ixekizumab 80 mg Q2W to placebo for the randomized withdrawal safety population in Period 3. Treatment group comparisons will be

analyzed using the methods described in Section 6.1.2. the Period 2 (initial open-label treatment population), Period 2 and Period 3 combined (ixekizumab-treated patients within the randomized withdrawal safety population and nonrandomized population), and for Relapse Period (relapse population), the above safety variables will be summarized as described in Sections 6.1.1, 6.1.2, and 6.1.3, respectively.

Summaries of safety data collected during the Period 4 (post-treatment follow-up period) will be presented separately.

For safety analyses, the following baselines will be used:

- Treatment-emergent adverse events: baseline will be all results recorded during the baseline period (see Section 6.1 for definitions of the baseline period).
- Treatment-emergent abnormal laboratory and vital signs: baseline will be all results recorded during the baseline period (see Section 6.1 for definitions of the baseline period).
- Change from baseline to minimum and maximum: baseline will be all results recorded during the baseline period (see Section 6.1 for definitions of the baseline period).

## 6.13.1. Extent of Exposure

Duration of exposure to study drug will be summarized by treatment group for Period 2, Period 3, and the Period 2 and Period 3 combined using descriptive statistics.

A by-patient listing of exposure duration with number of active injections and total dose will be provided.

The duration of exposure for Period 2 (initial open-label treatment period population) will be calculated:

For randomized patients:

```
Duration of exposure (days)
= (Date of randomization
- Date of first injection of ixekizumab 80 mg Q2W in Period 2) + 1
```

For nonrandomized patients:

```
\begin{aligned} \textit{Duration of exposure (days)} \\ &= (\textit{Date of last visit (scheduled or unscheduled)} \textit{on or prior to Visit 19}) \\ &- \textit{Date of first injection of ixekizumab 80 mg Q2W in Period 2)} + 1 \end{aligned}
```

The duration of exposure for Period 3 (randomized withdrawal safety population) will be calculated for the randomized patients as:

```
Duration of exposure (days)
= (Date of last visit (scheduled or unscheduled) or relapse in Period 3
- Date of first injection of study treatment after randomization in Period 3) + 1
```

Note that patients who experience a relapse during Period 3 will only have their Period 3 exposure calculated up until the date of relapse.

The duration of exposure for Relapse Period (relapse population) will be calculated as:

*Duration of exposure (days)* 

- = (Date of last visit (scheduled or unscheduled) in Period 3
- Date of first injection of ixekizumab 80 mg Q2W in Period 3 following relapse) + 1

The duration of exposure for Period 2 and Period 3 combined (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population) will be calculated for randomized patients as:

Duration of exposure (days)

- = (Date of last visit (scheduled or unscheduled) or relapse in Period 3
- Date of first injection of inital ixekizumab 80 mg Q2W treatment in Period 2) + 1

The duration of exposure for Period 2 and Period 3 combined (nonrandomized safety population) will be calculated for nonrandomized patients as:

Duration of exposure (days)

- = (Date of last visit (scheduled or unscheduled) in periods 2 or 3
- Date of first injection of inital ixekizumab 80 mg Q2W treatment in Period 2) + 1

The number and percentage of patients in each of the following categories will be included in the summaries (as applicable for the treatment period summarized):

- >0, ≥7 days, ≥14 days, ≥30 days, ≥60 days, ≥90 days, ≥120 days, ≥183 days, and ≥365 days, ≥548, and ≥730. Note that patients may be included in more than 1 category.
- >0 to <7 days, ≥7 to <14 days, ≥14 to <30 days, ≥30 to <60 days, ≥60 days to <90 days, >90 to <120 days, >120 to <183 days, >183 to <365 days, and >365 days.

The summaries will also include the following information:

• Total exposure in patient years, calculated as:

```
= \frac{\textit{Sum of duration of exposures for all patients in the study period in the treatment group}}{365.25}
```

- Number of active injections taken; derived using the response to the question "Was dose administered?" on the Exposure eCRF page and the actual dose description from IWRS study drug dispense dataset.
- Total dose (in mg); calculated by the number of active injections taken multiplied by a dose of 80 mg.

#### 6.13.2. Adverse Events

Adverse events will be classified based upon the latest version of Medical Dictionary for Regulatory Activities (MedDRA). Adverse events will be recorded at every study visit.

Condition starting on or after the date of informed consent will be considered an AE. A preexisting condition that worsens in severity on or after the date of informed consent will be considered and recorded as an AE on the AE eCRF page from the date of worsening onwards.

A TEAE is defined as an event that first occurred or worsened in severity after baseline and on or prior to the date of the last visit within the defined treatment period. Both the date/time of the event and the date/time of the dose (that is, injection) are considered when determining TEAEs. Treatment-emergent adverse events will be assigned to the study period to which it's considered treatment-emergent.

- The MedDRA Lowest Level Term (LLT) will be used when classifying AEs as treatment-emergent.
- The maximum severity recorded for each LLT prior to the first dose date/time in the treatment period will be used as the pretreatment severity for that LLT. If an event during the baseline period has missing severity, and the event persists during the treatment period, then it will be considered as treatment-emergent, regardless of the post-baseline level of severity. Events with a missing severity during the treatment period will be considered treatment-emergent.
- Adverse events with a particular LLT will be classified as treatment-emergent if they first start on or after the first dose date/time in the treatment period (that is, a patient has no preexisting conditions with that LLT), or if the severity is greater than the pretreatment severity for that LLT.

A follow-up emergent adverse event (FEAE) is defined as an event that first occurred or worsened in severity after the date of Visit 29 (that is, Week 104) or the ETV:

- The MedDRA LLT will be used when classifying AEs as follow-up emergent.
- For AEs that are ongoing at the date of Visit 29 (Week 104) or ETV, the
  maximum severity recorded for each LLT on or prior to the date of Visit 29
  (Week 104) or ETV will be used as the follow-up baseline severity for that LLT.

If a partial or completely missing AE start date/time or end date/time is present the following imputation rules will be utilized in the analysis:

- For the start date:
  - o If year, month, and day are missing, then use the consent date.
  - o If either month or month and day are missing, then use January 1.
  - o If only day is missing, impute the first day of the month.
- For the start time:
  - o Impute as 23:59
- For the end date:
  - o If year, month, and day are missing, then use the patient's last visit date.

- o If either month or month and day are missing, then use December 31.
- o If only day is missing, then use the last day of the month.
- The imputed date will not be beyond the patient's last visit date in the follow-up period.
- If there is any doubt, the event will be flagged as treatment-emergent or follow-up emergent according the corresponding study period. If a follow-up emergent event was already counted as treatment-emergent during the prior treatment period, it will not be counted as a follow-up emergent event.

Adverse events and TEAEs will be listed for all entered patients and summarized for the following periods:

- Period 2 (initial open-label treatment period population)
- Period 3 (randomized withdrawal safety population)
- Relapse Period (relapse population)
- Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population and nonrandomized population).

Adverse events and TEAEs for Period 3 will be compared between treatment groups using a Fisher's exact test for the randomized withdrawal safety population.

The following summaries/analyses will be performed:

- An overall summary of AEs including the number and percentage of patients who experienced TEAE, TEAE by maximum severity, death, SAE, TEAE related to study drug, discontinuations from the treatment due to an AE, and TEAEs of special interest.
- treatment-emergent adverse event by System Organ Class (SOC) and PT
- treatment-emergent adverse event by maximum severity, SOC, and PT

Follow-up emergent adverse events will be summarized for the follow-up population for the post-treatment follow-up period (Period 4):

• Follow-up emergent adverse event by SOC and PT

In general, for all AE related summaries, the number and percentage of patients experiencing the events will be presented by treatment group. The events will be ordered by decreasing frequency in the ixekizumab treatment group, within SOC and/or PT for sorting. For events that are gender-specific (as defined by MedDRA), the denominator and computation of the percentage will include only patients from the given gender.

# 6.13.3. Deaths, Other Serious Adverse Events, and Other Notable Adverse Events

#### 6.13.3.1. Deaths

A listing of deaths will be provided for all entered patients. All deaths will be included, regardless of the Investigator's or the Sponsor's judgment about causality, including (1) any deaths occurring during participation in the study, (2) any deaths occurring after a patient leaves (is discontinued from the study or completes the study) any of the studies in the database for which data are being presented if the death is (a) the result of a process initiated during the study, regardless of when it actually occurs, or (b) occurs during the post-treatment follow-up period after discontinuation of study drug. The actual rule used for including deaths will be provided in a footnote to the table. Any discrepancies between what is in the Lilly Safety System (LSS) and what is in the clinical study report (CSR) for individual studies will be explained in the footnote. The information from the LSS listing is used to create a hand-generated listing. Each listing will include study ID, investigator ID, patient ID, treatment group, baseline age, sex, associated AE, whether or not the death and Lilly's assessment of whether the process leading to death (NOT the death itself) began:

- "On study Drug": on study drug or within 14 days after study drug discontinuation
- "During the post-treatment follow-up period": >14 days after study drug discontinuation through the end of the post-treatment follow-up period
- "After the post-treatment follow-up period": any time after the end of the post-treatment follow-up period.

#### 6.13.3.2. Serious Adverse Event Analyses

An SAE is any AE that results in 1 of the following outcomes: death, life-threatening, initial or prolonged hospitalization, disability or permanent damage, congenital anomaly or birth defect, or any other serious/important medical events that may jeopardize the patient or may require intervention to prevent 1 of the other outcomes listed in the definition above.

Exposure-adjusted incidence rates (per 100 patient years) for SAEs will be presented by treatment group using MedDRA PT nested within SOC.

Serious adverse events will be listed for all entered patients and summarized for the following periods:

- Period 2 (initial open-label treatment period population)
- Period 3 (randomized withdrawal safety population)
- Relapse Period (relapse population)
- Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population and nonrandomized population).

Serious adverse events for Period 3 will be compared between treatment groups using the Fisher's exact test for the randomized withdrawal safety population.

A summary table of SAEs by SOC and PT will be provided.

A follow-up emergent serious adverse event (FESAE) is defined as an SAE that first occurred or worsened in severity after the date of Visit 29 (that is, Week 104) or the ETV. The baseline severity for SAEs occurring during the post-treatment follow-up period will be the maximum severity from the preceding visit before entering the post-treatment follow up period. A summary table of FESAEs by SOC and PT will be provided for the follow-up population for Period 4

The events will be ordered by decreasing frequency in the ixekizumab treatment group, within SOC and/or PT for sorting. For events that are gender-specific, the denominator and computation of the percentage will include only patients from the given gender.

#### 6.13.3.3. Other Significant Adverse Events

Adverse events that lead to treatment discontinuation (including death) will be listed for all entered patients and summarized for the following periods:

- Period 2 (initial open-label treatment period population)
- Period 3 (randomized withdrawal safety population)
- Relapse Period (relapse population)
- Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population and nonrandomized population).

Adverse events that lead to treatment discontinuation (including death) for Period 3 will be compared between treatment groups using the Fisher's exact test for the randomized withdrawal safety population.

A summary table of AEs that lead to treatment discontinuation (including death) by SOC and PT will be provided:

A summary table of FEAEs that lead to study discontinuation (including death) by SOC and PT will be provided for Period 4:

Events will be ordered by decreasing frequency in the combined ixekizumab group within SOC. For events that are gender-specific, the denominator and computation of the percentage will include only patients from the given gender.

# 6.13.4. Depression and Suicide-Related Patient Reported Outcomes

The QIDS-SR16, the C-SSRS, and the Self-Harm Supplement Form will be administered to patients at baseline and post-baseline to assess depression and the risk of suicide.

The QIDS-SR16 is a self-administered 16-item instrument intended to assess the existence and severity of symptoms of depression as listed in the American Psychiatric Association's (APA's)

Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) (APA 1994). Refer to Table RHBF.6.11 and Table RHBF.6.12 for further details.

The C-SSRS (Posner et al. 2007; Columbia University Medical Center [WWW]) is a scale that captures the occurrence, severity, and frequency of suicide-related ideations and behaviors during the assessment period.

The C-SSRS was added after study enrollment had been initiated. Given that few or no suicidal ideation or behaviors are anticipated, C-SSRS will be listed by patient and visit. Only patients that show suicidal ideation/behavior or self-injurious behavior without suicidal intent will be displayed (that is, if a patient answers are all 'no' for the C-SSRS, then that patient will not be displayed). However, if a patient reported any suicidal ideation/ behavior or self-injurious behavior without suicidal intent at any time point then all their ideation and behavior will be displayed, even if not positive.

The Self-Harm Supplement Form is a 1-question form that is completed, at any visit, including baseline visits, that asks for the number of suicidal or nonsuicidal self-injurious behaviors the patient has experienced since the last assessment. For each unique event identified, a questionnaire (Self-Harm Follow-up Form) which collects supplemental information on the self-injurious behavior is to be completed. Supplemental information collected will be listed by patient and visit for only the patients that have a number of suicidal or nonsuicidal self-injurious behaviors greater than 0 at any visit.

## 6.13.5. Clinical Laboratory Evaluation

Clinical laboratory assessments include hematology, serum chemistry, urinalysis, and safety-related immune markers such as neutrophil counts.

By-patient listing of laboratory test values will be provided for all entered patients. Listing of laboratory tests reference ranges (both large clinical trial population based reference limits and Covance reference ranges) will be provided. By-patient listing of abnormal laboratory test results (criteria defined in the shift tables excluding the normal category) for parameters of special interest (hepatic, immunoglobulins, leukocytes and platelets) will be provided.

Laboratory results will be summarized for (unless otherwise noted):

- Period 2 (initial open-label treatment period population);
- Period 3 (randomized withdrawal safety population);
- Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population and nonrandomized population)

Continuous laboratory tests will be summarized as changes from baseline for patients who have both baseline and at least 1 post-baseline result.

• The scheduled visits/measurements will be included. The unscheduled visits and the repeat measurements will be excluded.

- Both international system of unit (SI) and conventional unit will be summarized when different.
- Data will be analyzed based on original scale.

Change from minimum value during the baseline period to the minimum value during the treatment period, as well as change from the maximum value during the baseline period to the maximum value during the treatment period will be summarized for patients who have both a baseline and at least 1 post-baseline result.

For the randomized withdrawal safety population for Period 3, the comparisons between treatment groups will be conducted using an ANCOVA with treatment group and baseline value in the model.

The number and percentage of patients with a treatment-emergent or follow-up emergent abnormal, high, or low for laboratory tests will be summarized by treatment group. These will be displayed for (unless otherwise noted):

- Period 2 (initial open-label treatment period population)
- Period 3 (randomized withdrawal safety population)
- Relapse Period (relapse population)
- Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population and nonrandomized population); and Period 4 (post-treatment follow-up period population)
- Period 4 (post-treatment follow-up period population)

The comparisons between treatment groups will be conducted using the Fisher's exact test for the randomized withdrawal safety population for Period 3.

- All scheduled, unscheduled, and repeated measurements will be included.
- In general, large clinical trial population based reference limits (that is, Lilly reference ranges) will be used to define the low and high limits since it is generally desirable for limits used for analyses to have greater specificity (identify fewer false positive cases) than reference limits used for individual subject management. In the case when the reference limits based on the large clinical trial population is not available for a laboratory measure, Covance reference ranges will be used. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, and alkaline phosphatase (ALP) will not be included in the treatment-emergent abnormal, high, or low summary as a separate analysis addressing the risk of liver injury is described in Section 6.13.7 in which Covance Reference Ranges are used.
- Note that the ranges are defined by a lower limit of normal (LLN) and an upper limit of normal (ULN). A result that is greater than or equal to the LLN and less than or equal to the ULN is considered to be within the normal ranges.

- For categorical laboratory tests:
  - Treatment-emergent abnormal value is defined as a change from normal at all baseline visits to abnormal at any time post-baseline during the treatment period.
  - o Follow-up emergent **abnormal** result is defined as a change from normal at baseline to abnormal at any time during the follow-up period.
- For continuous laboratory tests:
  - Treatment-emergent high value is defined as a change from a value less than
    or equal to the ULN at all baseline visits to a value greater than the ULN at
    any time post-baseline during the treatment period.
  - Treatment-emergent low value is defined as a change from a value greater than or equal to the LLN at all baseline visits to a value less than the LLN at any time post-baseline during the treatment period.
  - Follow-up emergent high value is defined as a change from a value less than
    or equal to the ULN at baseline to a value greater than the ULN at any time
    post-baseline during the follow-up period.
  - o Follow-up emergent **low** value is defined as a change from a value greater than or equal to the LLN at baseline to a value less than the LLN at any time post-baseline during the follow-up period.

Shift tables will be produced using the following categories:

- Neutrophils:  $\ge 1 \times LLN$  (Normal), < LLN to  $\ge 1.5 \times 10^{9}/L$  (Grade 1),  $< 1.5 \times 10^{9}/L$  to  $\ge 1.0 \times 10^{9}/L$  (Grade 2),  $< 1.0 \times 10^{9}/L$  to  $\ge 0.5 \times 10^{9}/L$  (Grade 3), and  $< 0.5 \times 10^{9}/L$  (Grade 4)
- Leukocytes:  $\ge 1 \times LLN$  (Normal), < LLN to  $\ge 3.0 \times 10^9/L$  (Grade 1),  $< 3.0 \times 10^9/L$  to  $\ge 2.0 \times 10^9/L$  (Grade 2),  $< 2.0 \times 10^9/L$  to  $\ge 1.0 \times 10^9/L$  (Grade 3), and  $< 1.0 \times 10^9/L$  (Grade 4)
- Platelets: ≥1 × LLN (Normal), < LLN to ≥75.0 × 10^9/L (Grade 1), <75.0 × 10^9/L to ≥50.0 × 10^9/L (Grade 2), <50.0 × 10^9/L to ≥25.0 × 10^9/L (Grade 3), and <25.0 × 10^9/L (Grade 4)
- Lymphocytes:  $\ge 1 \times LLN$  (Normal), < LLN to  $\ge 0.8 \times 10^9/L$  (Grade 1),  $< 0.8 \times 10^9/L$  to  $\ge 0.5 \times 10^9/L$  (Grade 2),  $< 0.5 \times 10^9/L$  to  $\ge 0.2 \times 10^9/L$  (Grade 3), and  $< 0.2 \times 10^9/L$  (Grade 4)

The following LLN will be defined for analyses:

• Leukocytes: LLN=4.0 ×10^9/L

• Neutrophils: LLN=2.0×10^9/L

• Lymphocytes: LLN=1.1×10^9/L

• Platelets: LLN=150×10^9/L

In addition, for the above parameters (neutrophils, leukocytes, platelets and lymphocytes), the number and percentage of patients with minimum post-baseline results will be presented overall and by treatment group within the following groups using the categories as defined above:

- Decreased; post-baseline category < baseline category
- Increased; post-baseline category > baseline category
- Same; post-baseline category = baseline category

The number and percentages of patients with treatment-emergent low laboratory results at any time will be summarized for these 4 measures by treatment group for each treatment period. Shift tables will be produced showing the number and percentage of patients with a minimum post-baseline result for these 4 measures and will be summarized overall, and by treatment group and baseline result.

### 6.13.5.1. Leukocytes (WBC) and Platelets

Leukocytes (WBC) and platelets results will be summarized for (unless otherwise noted):

- Period 2 (initial open-label treatment period population)
- Period 3 (randomized withdrawal safety population)
- Relapse period (relapse population)
- Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population and nonrandomized population).

Change from minimum value and maximum value for total leukocytes, neutrophils, platelets, lymphocytes, monocytes, eosinophils, and basophils will be included in summaries described in Section 6.13.5. Unless otherwise specified, neutrophils will be summarized for absolute neutrophils (defined as the sum of segmented neutrophil count and the band neutrophil count). Laboratory values at each visit (starting at baseline) and change from baseline to each scheduled visit for these laboratory tests will be included in box plots (with outliers displayed) described in Section 6.13.5.

## 6.13.5.2. Neutrophil Follow-Up

Neutrophil counts will be followed throughout the study. Patients will continue in Period 4 until their neutrophil counts have recovered.

The neutrophil follow-up analysis will be conducted on the neutrophil follow-up population defined as patients who have an absolute neutrophil count <1500 cells/ $\mu$ L (SI units: <1.5× 10^9/L) at the last scheduled visit or early termination visit prior to entering the post-treatment follow-up period (Period 4) and less than the patient's baseline absolute neutrophil count (that is, prior to first injection at Week 0). These patients are monitored during the Period 4 until neutrophil recovery.

Neutrophil clinical recovery is defined as an absolute neutrophil count  $\geq 1500$  cells/ $\mu$ L (SI units:  $\geq 1.5 \times 10^{9}$ L) or greater than or equal to a patient's absolute neutrophil count prior to first study drug injection at Week 0.

If a patient's neutrophil count has not recovered, within 12 weeks after entering the follow-up period (Visit 802), the patient will return for Visit 803 (12 weeks after Visit 802). Additional visits may be required for appropriate patient management depending upon the degree of neutropenia. If at Visit 802, a patient has met the criteria for neutrophil recovery, the patient's participation in the study will be considered complete unless the investigator deems additional follow-up may be necessary.

The number and percentage of patients achieving neutrophil clinical recovery will be presented by treatment group and week interval for neutrophil follow-up population for post-treatment follow-up period (Period 4). The number and percentage of patients with an absolute neutrophil cell count that is at least 25%, 50%, 75%, or 100% of the patient's baseline absolute neutrophil count (that is, prior to first injection at Week 0), irrespective of absolute neutrophil minimum, will be included in the summary.

The time to neutrophil recovery will be calculated (for patients entering the Post-Treatment Follow-up Period) as follows:

Time to neutrophil recovery (in weeks) =  $(Date\ of\ neutrophil\ recovery-Date\ of\ last\ visit\ prior\ to\ entering\ the\ follow-up\ period)$  / 7.

Kaplan-Meier estimates of the proportion of patients not yet experiencing absolute neutrophil recovery at selected time points will be provided by treatment group. A Kaplan-Meier plot of the time to neutrophil recovery will be presented by treatment group.

If a patient has not experienced neutrophil recovery, he/she will be censored at the date of the last neutrophil count assessment. If they did not have a neutrophil count assessment, they will be censored at the date of last follow-up visit.

# 6.13.6. Vital Signs and Other Physical Findings

Analyses will be conducted on vital signs and physical characteristics including systolic blood pressure (mmHg), diastolic blood pressure (mmHg), pulse (bpm), weight (kg), and BMI (kg/m²). By-patient listing of vital signs and physical characteristics will be provided.

Vital signs and other physical finding results will be summarized for (unless otherwise noted):

- Period 2 (initial open-label treatment period population)
- Period 3 (randomized withdrawal safety population)
- Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population and nonrandomized population).

Change from baseline for vital signs and other physical findings will be summarized for patients who have both baseline and at least one post-baseline result.

• The scheduled visits/measurements will be included. The unscheduled visits and the repeat measurements will be excluded.

- For the randomized withdrawal safety population for Period 3, the comparisons between treatment groups will be conducted using an ANCOVA with treatment group and baseline value in the model.
- Data will be analyzed based on original scale.

Change from minimum value during the baseline period to the minimum value during the treatment period, as well as change from the maximum value during the baseline period to the maximum value during the treatment period will be summarized for patients who have both a baseline and at least 1 post-baseline result.

The number and percentage of patients with treatment-emergent or follow-up emergent high or low vital sign and weight at any time will be summarized. These will be displayed for (unless otherwise noted):

- Period 2 (initial open-label treatment period population)
- Period 3 (randomized withdrawal safety population)
- Relapse Period (relapse population)
- Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population and nonrandomized population)
- Period 4 (post-treatment follow-up period population)

The comparisons between treatment groups will be conducted using the Fisher's exact test for the randomized withdrawal safety population for Period 3.

Table RHBF.6.5 defines the high and low baseline values as well as the limits that are specified as treatment-emergent and follow-up emergent. Note that weight does not have an abnormal baseline; therefore, the treatment-emergent and follow-up emergent values are determined by change from baseline.

- All post-baseline scheduled, unscheduled and repeated measurements will be included.
- To assess increases, change from the maximum value during the baseline period or baseline to the maximum value during each study period will be used.
- To assess decreases, change from the minimum value during the baseline period or baseline to the minimum value during each study period will be used.
- For treatment-emergent high and low:
  - A treatment-emergent high result is defined as a change from a value less than
    or equal to the high limit at baseline to a value greater than the high limit at
    any time that meets the specified change criteria during the treatment period.
  - o A treatment-emergent **low** result is defined as a change from a value greater than or equal to the low limit at baseline to a value less than the low limit at any time that meets the specified change criteria during the treatment period.

- For follow-up emergent high and low:
  - A follow-up emergent high result is defined as a change from a value less than or equal to the high limit at baseline to a value greater than the high limit at any time that meets the specified change criteria during the follow-up period.
  - A follow-up emergent low result is defined as a change from a value greater than or equal to the low limit at baseline to a value less than the low limit at any time that meets the specified change criteria during the follow-up period.

Table RHBF.6.5. Categorical Criteria for Abnormal Treatment-Emergent Blood Pressures and Pulse Measurement, and Categorical Criteria for Weight Changes for Adults

| Parameter | Low | High |
|-------------------------|-----------------------|------------------------|
| Systolic BP (mm Hg) a | ≤90 and decrease from | ≥140 and increase from |
| (supine or sitting – | baseline ≥20 | baseline ≥20 |
| forearm at heart level) | | |
| Diastolic BP (mm Hg) a | ≤50 and decrease from | ≥90 and increase from |
| (supine or sitting – | baseline ≥10 | baseline ≥10 |
| forearm at heart level) | | |
| Pulse (bpm) a | <50 and decrease from | >100 and increase from |
| (supine or sitting) | baseline ≥15 | baseline ≥15 |
| Weight (kg) | (Loss) decrease from | (Gain) increase from |
| | baseline ≥7% | baseline ≥7% |

Abbreviations: BP = blood pressure; bpm = beats per minute; kg = kilogram; mm Hg = millimeters of mercury.

To assess the effect of administration of study drug on vital signs (blood pressures and pulse rate) among patients, at Week 0, vital signs will be measured before the first injection and 1 hour after the injection. The box plots will be produced for pre-dose and post-dose vital signs at Week 0 (Visit 2) for the initial open-label treatment period population.

# 6.13.7. Special Safety Topics including Adverse Events of Special Interest

Safety information on special topics including AESIs will be presented by treatment group and by study period. Table RHBF.6.6 provides the definitions/derivations and analyses methods (including analyses, summaries and by-patient listings) of special safety topics including AESIs.

Potential AESIs will be identified by a standardized MedDRA query (SMQ) or a Lilly-defined MedDRA PT listing. Preferred terms within an SMQ will be classified as broad and narrow. In the Lilly-defined MedDRA PT listings, Lilly has provided the broad and narrow classification. The Lilly-defined broad terms are for a more sensitive search of potential events of interest and the Lilly-defined narrow terms are for a more specific search. Therefore, the summaries will include the classifications of broad term (same as pooling narrow and broad terms together) and narrow term. In the event that the listing of terms or analysis changes for a special safety topic,

a Baseline abnormal values are defined by the value presented.

it will be documented in the program safety analysis plan (PSAP) which will supersede this document; it will not warrant an amendment to the individual study SAP.

Table RHBF.6.6. Definitions and Analyses of Special Safety Topics Including Adverse Events of Special Interest

| Special Safety<br>Topic | Definition / Derivation | Analysis / Summary / Listing |
|---|---|---|
| Hepatic | Hepatic AE analysis will include events that are potentially drug-related hepatic disorders by using the MedDRA PTs contained in any of the following SMQs or sub-SMQs as defined in MedDRA: • Broad and narrow terms in the Liver related investigations, signs and symptoms (20000008) • Broad and narrow terms in the Cholestasis and jaundice of hepatic origin (20000009) • Broad and narrow terms in the Hepatitis, non-infectious (20000010) • Broad and narrow terms in the Hepatic failure, fibrosis and cirrhosis and other liver damage (20000013) • Narrow terms in the Liver-related coagulation and bleeding disturbances (20000015) | Period 2, Period 3, and Combined Periods 2 and 3 (Summary): Period 3 randomized withdrawal safety population (Fisher's exact test): TEAE by PT within SMQ or sub-SMQ, SAE by PT within SMQ or sub-SMQ, AE leading to treatment discontinuation by PT within SMQ or sub-SMQ Listing: TEAE |
| | Elevations in hepatic laboratory tests (ALT, AST, ALP, total bilirubin) using Performing lab ULN during the treatment period are defined as: • Include scheduled visits, unscheduled visits, and repeat measurements. • ALT or AST: maximum post-baseline measurement ≥3 times (3×), 5×, 10×, and 20× the Covance ULN for all patients with a post-baseline value. ○ The analysis of 3×ULN will contain 4 subsets: patients whose non-missing maximum baseline value is ≤1×ULN, >1×ULN to <3×ULN, ≥3×ULN, or missing. ○ The analysis of 5×ULN will contain 5 subsets: patients whose non-missing maximum baseline value is ≤1×ULN, >1×ULN to <3×ULN, ≥3×ULN to <5×ULN, ≥5×ULN, or missing. ○ The analysis of 10×ULN will contain 6 subsets: patients whose non-missing maximum baseline value is ≤1×ULN, >1×ULN to <3×ULN, ≥3×ULN to <5×ULN, ≥5×ULN to <10×ULN, ≥10×ULN, or missing. ○ The analysis of 20×ULN will contain 7 subsets: patients whose non-missing maximum baseline value is ≤1×ULN, >1×ULN to <3×ULN, ≥3×ULN to <5×ULN, ≥5×ULN to <10×ULN, ≥10×ULN to <20×ULN, ≥20×ULN, or missing. • Total bilirubin: maximum post-baseline measurement greater ≥2× the Performing lab ULN for all patients with a post-baseline value, and divided into 4 subsets: patients whose non-missing maximum baseline value is ≤1×ULN, >1×ULN to <1.5×ULN, ≥1.5×ULN to <2×ULN, ≥2×ULN, or missing. • ALP: maximum post-baseline measurement >1.5× the Covance ULN for all patients with a | Period 2, Period 3, and Combined Periods 2 and 3 (Summary): Elevations in hepatic laboratory tests: maximum baseline category to abnormal maximum post-baseline category |

| Special Safety | D. C. Hiller / Device the | And Livin / Samura and / Living |
|---|---|---|
| Topic | Definition / Derivation | Analysis / Summary / Listing |
| | post-baseline value, and divided into 4 subsets: patients whose non-missing maximum | |
| | baseline value is $\le 1 \times ULN$ , $>1 \times ULN$ to $\le 1.5 \times ULN$ , $>1.5 \times ULN$ , or missing. | D : 14 D : 14 1C 1: 1 |
| | Shift for ALT, AST, and total bilirubin from maximum baseline to maximum post-baseline will | Period 2, Period 3, and Combined |
| | be produced with the requirements using Performing lab ULN during the treatment period: | Periods 2 and 3 (Summary): |
| | Include scheduled visits, unscheduled visits, and repeat measurements. | Shifts from maximum baseline to |
| | Use the maximum non-missing value in the baseline period. Here the maximum non-missing value in the baseline period. | maximum post-baseline category |
| | Use the maximum non-missing post-baseline value within each study period. | |
| | • Categories are: | |
| | o ALT: ≤1×ULN, >1 to <3×ULN, ≥3 to <5×ULN, ≥5 to <10×ULN, ≥10 to <20×ULN, | |
| | and ≥20×ULN | |
| | o AST: ≤1×ULN, >1 to <3×ULN, ≥3 to <5×ULN, ≥5 to <10×ULN, ≥10× to <20×ULN | |
| | and ≥20×ULN | |
| | o Total bilirubin: ≤1×ULN, >1 to <1.5×ULN, ≥1.5 to <2×ULN, ≥2×ULN | |
| | o ALP; ≤1× ULN, >1 to ≤1.5× ULN, >1.5× ULN. | |
| | With additional categories: | |
| | o Decreased: post-baseline category < baseline category | |
| | o Increased: post-baseline category > baseline category | |
| | Same: post-baseline category = baseline category | |
| | Elevated hepatic criteria: maximum ALT $\ge 3 \times ULN$ and maximum total bilirubin $\ge 2 \times ULN$ , | Listing: |
| | using Performing lab Reference Ranges. | Elevations in hepatic laboratory tests |
| | Listing of patients who meet any of the following criteria: | |
| | • Elevated hepatic criteria: defined as maximum ALT ≥3×ULN and maximum total bilirubin | |
| | ≥2×ULN | |
| | An ALT or AST ≥3×ULN | |
| | • An alkaline phosphatase (ALP) ≥1.5×ULN | |
| | A total bilirubin ≥2×ULN | |
| | The listing will include: patient demographics, concomitant medications, ALT/AST/ALP/total | |
| | bilirubin/gamma-glutamyl transferase (GGT) by visit, treatment start and stop dates, and reason | |
| | for treatment discontinuation. | |
| | eDISH plot: use maximum ALT measurement and maximum total bilirubin measurement after | <b>Period 2, 3, and 4 combined</b> : eDISH plot |
| | the first injection of study treatment with patients having at least one post-baseline ALT and | |
| | total bilirubin, which contributes one point to the plot. The measurements do not need to be | |
| | taken at the same blood draw. | |

| Special Safety<br>Topic | Definition / Derivation | Analysis / Summary / Listing |
|---|---|---|
| Cytopenias | Cytopenias are defined using the PTs from the following 2 sub-SMQs of the Haematopoietic cytopenias SMQ (20000027) as specified in MedDRA: • Broad and narrow terms in the Haematopoietic leukopenia (20000030) • Broad and narrow terms in the Haematopoietic thrombocytopenia (20000031) | Period 2, Period 3, and Combined Periods 2 and 3 (Summary): Period 3 randomized withdrawal safety population (Fisher's exact test): TEAE by PT within sub-SMQ, SAE by PT within sub-SMQ, AE leading to treatment discontinuation by PT within sub-SMQ |
| | | Listing:<br>TEAE |
| Infections | Infections are events including all infections (defined using all the MedDRA PTs from the Infections and infestations SOC), serious infections, potential OIs, and infections resulting in anti-infective medication adminstration (i.e., antibacterial, antiviral, antifungal, antiparasitic treatment.). | Period 2, Period 3, and Combined Periods 2 and 3 (Summary): Period 3 randomized withdrawal safety population (Fisher's exact test): TEAE by PT, TEAE by maximum severity by PT, SAE by PT, AE leading to treatment discontinuation by PT |
| | | Listing: TEAE |
| | Anti-infective medications are defined in Appendix 7 including antibacterial, antiviral, antifungal, and antiparasitic treatment. Listing of patients experiencing a TEAE of infections will be provided including the following additional information: anti-infective medications use (if treated) with medication start/end dates, indication for use, and route; minimum post-baseline value within treatment Period 2 for leukocytes, platelets, lymphocytes, and absolute neutrophils. | Listing: TEAE with anti-infective medications |
| | <ul> <li>The list of MedDRA terms used to identify infections that are defined as potential OIs are<br/>found in Appendix 12. This list contains PTs with Categories (narrow or broad) from the<br/>Infections and Infestations SOC and from the Investigations SOC which can assist in<br/>indentifying potential OIs. The narrow terms are considered OIs unless medical review</li> </ul> | Period 2, Period 3, and Combined<br>Periods 2 and 3 (Summary):<br>Period 3 randomized withdrawal safety<br>population (Fisher's exact test): |

| Special Safety | | |
|---|---|---|
| Topic | Definition / Derivation | Analysis / Summary / Listing |
| | determines that the reported term is not consistent with the patient's clinical | TEAE of OIs by maximum severity by PT |
| | history/presentation/course. Medical review of broad terms is needed for final | |
| | determination of patients meeting the program definition of OIs. | Listing: |
| | Listing of patients experiencing a TEAE of potential OIs will be provided including the | TEAE of OIs |
| | following additional information: source of identification (CRF or Lilly-defined list), | |
| | primary/secondary site of infection, primary/secondary infection type, primary/secondary | |
| | identified by a laboratory diagnostic test (Yes/No), acquired in a health care setting (Yes/No). | |
| | The duration of each common ( $\geq$ 1% of total ixekizumab) TEAE PT of Infections is defined as: | Period 2, Period 3, and Combined |
| | Duration of treatment-emergent AE Infections (in weeks) = (End date of AE – Start date of AE | Periods 2 and 3 (Summary): |
| | + 1) / 7. Only TEAEs of infections beginning during treatment Period 3 will be included in the | Period 3 randomized withdrawal safety |
| | summary. If an AE has not ended by the date of completion of the treatment Period 3, or date of | population (Summary): |
| | early discontinuation, it will be censored as of that date (last visit within the treatment Period 3, | Duration of Common TEAE – Infections |
| | or date of early discontinuation). If a patient has multiple episodes of the same TEAE, the | |
| | episode with the greatest severity will be used for the duration of event calculation. If a patient | |
| | has multiple episodes of the same TEAE with the same severity, the episode with the longest | |
| | duration will be used for the duration of event calculation. | |

| Reactions/ Hypersensitivities or non-anaphylaxis events (these will refer to events that are not localized to the site of injection) and summarized separately. Medical reviews are needed for final determination of patients with allergic reactions/hypersensitivities. Allergic Reactions/Hypersensitivities Events, Potential Anaphylaxis: Anaphylaxis has been broadly defined as "a serious allergic reaction that is rapid in onset and may cause death" (Sampson et al. 2006). Identification of cases of potential anaphylaxis from the clinical trial data involves 2 criteria: 1) designed to specifically identify cases (following Criterion 1) based on narrow terms from the MedDRA SMQ for anaphylactic reaction (20000021). Criterion 1 for anaphylaxis is defined by the presence of a TEAE based on the following MedDRA PTs from the anaphylactic reaction SMQ: • Anaphylactic reaction • Anaphylactic reaction • Anaphylactic disock • Anaphylactic is hock • Anaphylactic is the complete of the sevents should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | Special Safety<br>Topic | Definition / Derivation | Analysis / Summary / Listing |
|---|---|---|---|
| of patients with allergic reactions/hypersensitivities. Allergic Reactions/Hypersensitivity Events. Potential Anaphylaxis: Anaphylaxis has been broadly defined as "a serious allergic reaction that is rapid in onset and may cause death" (Sampson et al. 2006). Identification of cases of potential anaphylaxis from the clinical trial data involves 2 criteria: 1) designed to specifically identify cases (following Criterion 1) based on narrow terms from the MedDRA SMQ for anaphylactic reaction (20000021). Criterion 1 for anaphylaxis is defined by the presence of a TEAE based on the following MedDRA PTs from the anaphylactic reaction (20000021). Criterion 1 for anaphylactic shock • Anaphylactoid shock • Anaphylactoid shock • Anaphylactoid reaction • Anaphylactoid reaction • Anaphylactoid shock • Anaphylactoid and evelop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category A: Involvement of the skin-mucosal tissue • Category C: Reduced blood pressure or associated symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | - | | Period 2, Period 3, and Combined Periods 2 and 3: |
| Allergic Reactions/Hypersensitivity Events, Potential Anaphylaxis: Anaphylaxis has been broadly defined as "a serious allergic reaction that is rapid in onset and may cause death" (Sampson et al. 2006). Identification of cases of potential anaphylaxis from the clinical trial data involves 2 criteria: 1) designed to specifically identify cases (following Criterion 1) based on narrow terms from the MedDRA SMQ for anaphylactic reaction (20000021). Criterion 1 for anaphylaxis is defined by the presence of a TEAE based on the following MedDRA PTs from the anaphylactic reaction SMQ: • Anaphylactic reaction • Anaphylactic shock • Anaphylactic identify cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Ccriterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Category and device to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | • • | | |
| Allergic Reactions/Hypersensitivity Events, Potential Anaphylaxis: Anaphylaxis has been broadly defined as "a serious allergic reaction that is rapid in onset and may cause death" (Sampson et al. 2006). Identification of cases of potential anaphylaxis from the clinical trial data involves 2 criteria: 1) designed to specifically identify cases (following Criterion 1) based on narrow terms from the MedDRA SMQ for anaphylactic reaction (20000021). Criterion 1 for anaphylaxis is defined by the presence of a TEAE based on the following MedDRA PTs from the anaphylactic reaction SMQ: • Anaphylactic is shock • Anaphylactic is shock • Anaphylactoid reaction • Anaphylactoid reaction • Anaphylactoid reaction • Anaphylactoid reaction • Anaphylactoid reaction • Anaphylactoid shock • Anaphylactoid reaction • Kounis Syndrome 2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | ities | of patients with allergic reactions/hypersensitivities. | • |
| (Sampson et al. 2006). Identification of cases of potential anaphylaxis from the clinical trial data involves 2 criteria: 1) designed to specifically identify cases (following Criterion 1) based on narrow terms from the MedDRA SMQ for anaphylactic reaction (20000021). Criterion 1 for anaphylaxis is defined by the presence of a TEAE based on the following MedDRA PTs from the anaphylactic reaction SMQ: • Anaphylactic reaction • Anaphylactic shock • Anaphylactoid shock • Anaphylactoid shock • Anaphylactoid shock • Anaphylactic treatment • Kounis Syndrome 2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | Allergic Reactions/Hypersensitivity Events, Potential Anaphylaxis: Anaphylaxis has been | = = · |
| data involves 2 criteria: 1) designed to specifically identify cases (following Criterion 1) based on narrow terms from the MedDRA SMQ for anaphylactic reaction (20000021). Criterion 1 for anaphylaxis is defined by the presence of a TEAE based on the following MedDRA PTs from the anaphylactic reaction SMQ: • Anaphylactic reaction • Anaphylactic shock • Anaphylactic deaction • Anaphylactic treatment • Kounis Syndrome 2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | broadly defined as "a serious allergic reaction that is rapid in onset and may cause death" | TEAE by maximum severity by PT within |
| 1) designed to specifically identify cases (following Criterion 1) based on narrow terms from the MedDRA SMQ for anaphylactic reaction (20000021). Criterion 1 for anaphylaxis is defined by the presence of a TEAE based on the following MedDRA PTs from the anaphylactic reaction SMQ: • Anaphylactic reaction • Anaphylactic shock • Anaphylactoid reaction • Anaphylactoid shock • Anaphylactic treatment • Kounis Syndrome 2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | (Sampson et al. 2006). Identification of cases of potential anaphylaxis from the clinical trial | Category, |
| from the MedDRA SMQ for anaphylactic reaction (20000021). Criterion 1 for anaphylaxis is defined by the presence of a TEAE based on the following MedDRA PTs from the anaphylactic reaction SMQ: • Anaphylactic reaction • Anaphylactic shock • Anaphylactic di shock • Anaphylactic treatment • Kounis Syndrome 2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | data involves 2 criteria: | SAE by PT within Category, |
| anaphylaxis is defined by the presence of a TEAE based on the following MedDRA PTs from the anaphylactic reaction SMQ: • Anaphylactic reaction • Anaphylactic shock • Anaphylactoid reaction • Anaphylactoid shock • Anaphylactoid shock • Anaphylactic treatment • Kounis Syndrome 2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | 1) designed to specifically identify cases (following Criterion 1) based on narrow terms | AE leading to treatment discontinuation by |
| PTs from the anaphylactic reaction Anaphylactic reaction Anaphylactic shock Anaphylactoid reaction Anaphylactoid shock Anaphylactoid shock Anaphylactic treatment Kounis Syndrome 2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: Category A: Involvement of the skin-mucosal tissue Category B: Respiratory compromise Category C: Reduced blood pressure or associated symptoms Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | from the MedDRA SMQ for anaphylactic reaction (20000021). Criterion 1 for | PT within Category |
| <ul> <li>Anaphylactic reaction</li> <li>Anaphylactoid reaction</li> <li>Anaphylactoid shock</li> <li>Anaphylactoid shock</li> <li>Anaphylactic treatment</li> <li>Kounis Syndrome</li> <li>to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection.</li> <li>The 4 categories to be considered in Criterion 2 are:</li> <li>Category A: Involvement of the skin-mucosal tissue</li> <li>Category C: Reduced blood pressure or associated symptoms</li> <li>Category D: Persistent gastrointestinal symptoms</li> <li>The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in</li> </ul> | | anaphylaxis is defined by the presence of a TEAE based on the following MedDRA | |
| <ul> <li>Anaphylactic shock</li> <li>Anaphylactoid reaction</li> <li>Anaphylactoid shock</li> <li>Anaphylactic treatment</li> <li>Kounis Syndrome</li> <li>to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection.</li> <li>The 4 categories to be considered in Criterion 2 are: <ul> <li>Category A: Involvement of the skin-mucosal tissue</li> <li>Category B: Respiratory compromise</li> <li>Category C: Reduced blood pressure or associated symptoms</li> <li>Category D: Persistent gastrointestinal symptoms</li> </ul> </li> <li>The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in</li> </ul> | | | |
| <ul> <li>Anaphylactoid reaction</li> <li>Anaphylactoid shock</li> <li>Anaphylactic treatment</li> <li>Kounis Syndrome</li> <li>2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection.</li> <li>The 4 categories to be considered in Criterion 2 are: <ul> <li>Category A: Involvement of the skin-mucosal tissue</li> <li>Category B: Respiratory compromise</li> <li>Category C: Reduced blood pressure or associated symptoms</li> <li>Category D: Persistent gastrointestinal symptoms</li> </ul> The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in</li> </ul> | | | TEAE |
| <ul> <li>Anaphylactoid shock</li> <li>Anaphylactic treatment</li> <li>Kounis Syndrome</li> <li>2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection.</li> <li>The 4 categories to be considered in Criterion 2 are: <ul> <li>Category A: Involvement of the skin-mucosal tissue</li> <li>Category B: Respiratory compromise</li> <li>Category C: Reduced blood pressure or associated symptoms</li> <li>Category D: Persistent gastrointestinal symptoms</li> </ul> The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in</li> </ul> | | ± * | |
| <ul> <li>Anaphylactic treatment</li> <li>Kounis Syndrome</li> <li>2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection.</li> <li>The 4 categories to be considered in Criterion 2 are: <ul> <li>Category A: Involvement of the skin-mucosal tissue</li> <li>Category B: Respiratory compromise</li> <li>Category C: Reduced blood pressure or associated symptoms</li> <li>Category D: Persistent gastrointestinal symptoms</li> </ul> The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in</li> </ul> | | | |
| <ul> <li>Kounis Syndrome</li> <li>to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection.</li> <li>The 4 categories to be considered in Criterion 2 are: <ul> <li>Category A: Involvement of the skin-mucosal tissue</li> <li>Category B: Respiratory compromise</li> <li>Category C: Reduced blood pressure or associated symptoms</li> <li>Category D: Persistent gastrointestinal symptoms</li> </ul> The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in</li> </ul> | | 1 7 | |
| <ul> <li>2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in</li> </ul> | | | |
| Criterion 2 for anaphylaxis requires having TEAEs from 2 or more of 4 categories of AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | | |
| AEs as described by Sampson et al. (2006). Occurrence of these events should be nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | | |
| nearly coincident and develop rapidly after exposure to the most recent injection; based on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | | |
| on recording of events on CRFs, all qualifying events must be within 1 day of study drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | | |
| drug injection. The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | | |
| The 4 categories to be considered in Criterion 2 are: • Category A: Involvement of the skin-mucosal tissue • Category B: Respiratory compromise • Category C: Reduced blood pressure or associated symptoms • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | | |
| <ul> <li>Category A: Involvement of the skin-mucosal tissue</li> <li>Category B: Respiratory compromise</li> <li>Category C: Reduced blood pressure or associated symptoms</li> <li>Category D: Persistent gastrointestinal symptoms</li> <li>The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in</li> </ul> | | | |
| <ul> <li>Category B: Respiratory compromise</li> <li>Category C: Reduced blood pressure or associated symptoms</li> <li>Category D: Persistent gastrointestinal symptoms</li> <li>The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in</li> </ul> | | | |
| <ul> <li>Category C: Reduced blood pressure or associated symptoms</li> <li>Category D: Persistent gastrointestinal symptoms</li> <li>The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in</li> </ul> | | | |
| • Category D: Persistent gastrointestinal symptoms The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | | |
| The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in | | | |
| L Appendix 8 | | Appendix 8. | |

| Special Safety | | |
|---|---|---|
| Topic | Definition / Derivation | Analysis / Summary / Listing |
| | Summaries of Criterion 2 anaphylactic TEAEs will be provided by the specific | |
| | combination of categories as follows: | |
| | AB: events based on meeting Category A and Category B (but no other category) | |
| | • AC: events based on meeting Category A and Category C (but no other category) | |
| | AD: events based on meeting Category A and Category D (but no other category) | |
| | BC: events based on meeting Category B and Category C (but no other category) | |
| | BD: events based on meeting Category B and Category D (but no other category) | |
| | CD: events based on meeting Category C and Category D (but no other category) | |
| | <ul> <li>ABC: events based on meeting Category A, Category B and Category C (but no<br/>other category)</li> </ul> | |
| | ABD: events based on meeting Category A, Category B and Category D (but no other category) | |
| | <ul> <li>ACD: events based on meeting Category A, Category C and Category D (but no other category)</li> </ul> | |
| | BCD: events based on meeting Category B, Category C and Category D (but no | |
| | other category) | |
| | ABCD: events based on meeting each of the 4 Criterion 2 categories | |
| | Summaries of treatment-emergent anaphylactic AEs will be provided for patients meeting | |
| | each of the 2 criteria and for patients who meet either criteria overall. Severity of treatment- | |
| | emergent Criterion 2 anaphylactic AEs will be based on the maximum severity of the | |
| | specific events met by the patient. Maximum severity of an (or overall) treatment-emergent | |
| | anaphylactic AE will be based on the maximum severity within Criterion 1 and/or Criterion | |
| | 2. | |
| | Allergic Reactions/Hypersensitivity Events, Non-Anaphylaxis: TEAEs of allergic | |
| | reaction/hypersensitivity categorized as non-anaphylaxis events are defined by the narrow | |
| | terms within Hypersensitivity SMQ (20000214) excluding the PTs noted in Appendix 9 and | |
| | excluding the anaphylactic events as defined above. | |
| | A by-patient listing will be provided for all patients experiencing TEAE of allergic | Listing: |
| | reactions/hypersensitivities at any time, including status/criterion of anaphylaxis or non- | TEAE including information collected on |
| | anaphylaxis, and the associated information collected on <i>Allergic/Hypersensitivity Reaction</i> | Allergic/Hypersensitivity Reaction Follow- |
| | Follow-Up eCRF page if identified by the investigator. | Up eCRF page |
| Injection Site | Injection site reaction is defined using the PTs from the MedDRA HLT of Injection site | Period 2, Period 3, and Combined Periods |

| Special Safety | | |
|---|---|---|
| Topic | Definition / Derivation | Analysis / Summary / Listing |
| Reactions | reactions as specified by MedDRA excluding the following 10 PTs: | 2 and 3: (Summary): |
| | 1) Embolia cutis medicamentosa | Period 3 randomized withdrawal safety |
| | 2) Injection site joint discomfort | population (Fisher's exact test): |
| | 3) Injection site joint effusion | TEAE by maximum severity by PT within |
| | 4) Injection site joint inflammation | HLT, |
| | 5) Injection site joint movement impairment | SAE by PT within HLT, |
| | 6) Injection site joint pain | AE leading to treatment discontinuation by |
| | 7) Injection site joint redness | PT within HLT |
| | 8) Injection site joint swelling | |
| | 9) Injection site joint warmth | TEAE identified by the investigator PT |
| | 10) Injection site joint infection | within HLT: |
| | | by maximum severity, |
| | The <i>Injection Site Reaction</i> eCRF page captures the injection site reactions identified by the | by maximum redness category, |
| | investigator. These TEAEs will be summarized within the MedDRA HLT by maximum | by maximum swelling category, |
| | severity or category. If more than 1 TEAE of injection site reaction occurs, the event with | by maximum pain category |
| | the worst value (within the individual categories: redness, swelling and pain) will be used. | |
| | Redness (Scored 0-4) | Listing: |
| | [0] Subject's normal skin color, no increased redness | TEAE including information collected on |
| | [1] Noticeable, but very mild redness | Injection Site Reaction eCRF page |
| | [2] Clearly red | |
| | [3] Bright red | |
| | [4] Dark with some scar formation | |
| | Swelling (Scored 0-4 after running a finger over injected area) | |
| | [0] No bump | |
| | [1] Barely noticeable | |
| | [2] Clear bump but very thin | |
| | [3] Clear bump 1 mm thick | |
| | [4] Clear bump 2 mm thick or more | |
| | Pain (including burning) (Scored 0-3) | |
| | [0] None | |
| | [1] Mild | |
| | [2] Moderate | |
| | [3] Severe | |

| Special Safety | | A 1 : (6 /T: r: |
|---|---|---|
| Topic Cerebro- | Definition / Derivation Cerebro-cardiovascular events will be externally adjudicated by the CEC at the Cleveland | Analysis / Summary / Listing |
| | | Period 2, Period 3, and Combined Periods |
| cardiovascular | Clinic, as outlined in the Manual of Operations. The CEC will adjudicate investigator- | 2 and 3 (Summary): |
| Events | reported events selected for adjudication and render an assessment as to whether the event | Period 3 randomized withdrawal safety |
| | represents a confirmed event (meeting the event definition with all necessary | population (Fisher's exact test): |
| | documentation), a non-event (does not meet the event definition and likely represents an | TEAE by PT within Subcategory, |
| | alternative or nonevent diagnosis), or lacks sufficient documentation for confirmation of an | |
| | event. All events which qualify for CEC adjudication will be used for the analysis of | T |
| | cerebro-cardiovascular events. The categories and subcategories of adjudicated events used | Listing: |
| | for the analysis will include the following: • Cardiovascular | TEAE |
| | o Death (Cardiovascular) | |
| | Cardiac Ischemic Event: Myocardial Infarction and Hospitalization for Unstable | |
| | Angina | |
| | Serious Arrhythmia Heavitalization for Heavit Failure | |
| | Hospitalization for Heart Failure Hospitalization for Hypertension | |
| | <ul> <li>Hospitalization for Hypertension</li> <li>Resuscitated Sudden Death</li> </ul> | |
| | Cardiogenic Shock | |
| | Coronary Revascularization | |
| | Neurologic Combined to French Transient Ladennia Attach on Strake (Harmandania) | |
| | <ul> <li>Cerebrovascular Event: Transient Ischemic Attack or Stroke (Haemorrhagic,<br/>Ischemic and Undetermined)</li> </ul> | |
| | / | |
| | Peripheral Vascular Events Peripheral Actorial Events | |
| | Peripheral Arterial Event Peripheral Review Visit (1988) | |
| | Peripheral Revascularization Figure will be analyzed using MedDBA BT nested within the CEC assessment (confirmed). | |
| | Events will be analyzed using MedDRA PT nested within the CEC assessment (confirmed event, no event, or insufficient documentation for event determination) and the subcategory. | |
| | The state of the s | |
| | Subtypes of stroke (Hemorrhagic Stroke, Ischemic Stroke, and Undetermined Stroke Type) will be displayed in the analyses nested within Cerebrovascular Event. Subtypes of Serious | |
| | Arrhythmia (Atrial Arrhythmia, Ventricular Arrhythmia, Heart Block, Other, Unknown) | |
| | will be displayed nested within Serious Arrhythmia. | |
| Major | | Donied 2 Donied 2 and Combined Donied 1 |
| Major | MACE (requiring adjudication as defined above) is defined as: | Period 2, Period 3, and Combined Periods |
| Adverse | Vascular Death (including cardiovascular and cerebro-vascular causes excluding) | 2 and 3 (Summary): |

| Special Safety | | |
|---|---|---|
| Topic | Definition / Derivation | Analysis / Summary / Listing |
| Cerebro- | hemorrhagic deaths outside of the central nervous system) | Period 3 randomized withdrawal safety |
| Cardiovascular | Non-fatal myocardial infarction | population (Fisher's exact test): |
| Events | Non-fatal stroke (subtypes: hemorrhagic stroke, ischemic stroke, undetermined stroke) | TEAE by maximum severity by PT within |
| (MACE) | type) | Category |
| | Where, | |
| | Vascular death should be captured as an Event on Adjudication - Death eCRF page with | |
| | Adjudication Death Type = 'Cardiovascular'. | Listing: |
| | Non-fatal myocardial infarction should be captured as an Event on Adjudication - | TEAE |
| | Cardiac Ischemic Event eCRF page with Type of Ischemic Event = "Myocardial | |
| | Infarction" and the Event is NOT on Adjudication - Death eCRF page. | |
| | Non-fatal strokes (ischemic, hemorrhagic) should be captured as an Event on | |
| | Adjudication - Cerebrovascular Event eCRF page with Stroke Cerebrovascular Event | |
| | Subtype in one of the following categories: hemorrhagic stroke, ischemic stroke, | |
| | undetermined stroke type, and the Event is NOT on Adjudication - Death eCRF page. | |
| | Subcategories of non-fatal stroke (Hemorrhagic Stroke, Ischemic Stroke, and | |
| | Undetermined Stroke Type) will be displayed nested within non-fatal stroke category. | |
| Malignancies | Malignancy is defined using PTs from the Malignant or unspecified tumors SMQ as | Period 2, Period 3, and Combined Periods |
| | specified in MedDRA (SMQ: 20000091, which includes the sub-SMQs: | 2 and 3 (Summary): |
| | • 20000195 [Tumors of unspecified malignancy], including sub-SMQs of 20000229 | Period 3 randomized withdrawal safety |
| | [Haematological tumours of unspecified malignancy] and 20000230 [Non- | population (Fisher's exact test): |
| | haematological tumours of unspecified malignancy] and | TEAE by PT within Category, |
| | • 20000194 [Malignant tumors], including sub-SMQs of 20000227 [Haematological | SAE by PT within Category, |
| | malignant tumours] and 20000228 [Non-haematological malignant tumours]). | AE leading to treatment discontinuation by |
| | Events will be summarize by the following categories: | PT within Category |
| | Nonmelanoma Skin Cancer (NMSC) | |
| | o Basal Cell Carcinoma, PTs include: | Listing: |
| | <ul> <li>Basal cell carcinoma</li> </ul> | TEAE |
| | <ul> <li>Basosquamous carcinoma</li> </ul> | |
| | <ul> <li>Basosquamous carcinoma of skin</li> </ul> | |
| | o Squamous Cell Carcinoma, PTs include: | |
| | <ul> <li>Squamous cell carcinoma of skin</li> </ul> | |
| | <ul> <li>Bowen's disease</li> </ul> | |
| | <ul> <li>Lip squamous cell carcinoma</li> </ul> | |
| Special Safety | | |
|---|---|---|
| Topic | Definition / Derivation | Analysis / Summary / Listing |
| | <ul> <li>Skin squamous cell carcinoma metastatic</li> </ul> | |
| | <ul> <li>Keratoacanthoma</li> </ul> | |
| | Malignancies excluding NMSC: all PTs in the Malignant or unspecified tumors SMQ | |
| | excluding the 8 defined NMSC PTs. | |
| Depression and | Depression and suicide/self-injury is defined using the PTs from the Depression and | Period 2, Period 3, and Combined Periods |
| Suicide/self- | suicide/self-injury SMQ as specified in MedDRA (SMQ: 20000035, which includes the sub- | 2 and 3 (Summary): |
| injury | SMQs: 20000037 [Suicide/self-injury] and 20000167 [Depression (excluding suicide and | Period 3 randomized withdrawal safety |
| | self injury)]). | population (Fisher's exact test): |
| | | TEAE by PT within SMQ and sub-SMQ, |
| | | SAE by PT within SMQ and sub-SMQ, |
| | | AE leading to treatment discontinuation by |
| | | PT within SMQ and sub-SMQ |
| | | Listing: |
| | | TEAE (including QIDS-SR16 total scores) |
| | The Quick Inventory of Depressive Symptomology-Self Report 16 items (QIDS-SR16) is a | Period 2, Period 3, and Combined Periods |
| | self-administered 16-item instrument intended to assess the existence and severity of | 2 and 3 |
| | symptoms of depression as listed in the American Psychiatric Association's (APA's) | Period 3 randomized withdrawal safety |
| | Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) (APA 1994). | population |
| | Refer to Table RHBF.6.11 and Table RHBF.6.12 for further details. | Shift in QIDS-SR16 total score categories |
| | The following groups are based upon the maximum post-baseline QIDS-SR16 total score | Similar Que de como de |
| | category (none, mild, moderate, severe, very severe) score: | |
| | ■ Improved; maximum post-baseline < baseline | |
| | <ul> <li>Worsened; post-baseline &gt; baseline</li> </ul> | |
| | <ul><li>Same; post-baseline = baseline</li></ul> | |
| Inflammatory | Inflammatory Bowel Disease (IBD) will be identified by medical review using the following | Period 2, Period 3, and Combined Periods |
| Bowel Disease | Category and MedDRA PTs. The narrow terms are considered IBD. Medical reviews of | 2 and 3 (Summary): |
| | patients with identified broad terms are needed for final determination of patients with IBD. | Period 3 randomized withdrawal safety |
| | IBD Specific Terms (Narrow terms) | population (Fisher's exact test): |
| | Inflammatory Bowel Disease: Inflammatory bowel disease Contra's Disease: Contra's disease. | TEAE by PT by maximum severity by PT |
| | Crohn's Disease: Crohn's disease Ula practice Colities: A part has properly a circula practice colities of colities and constitute colities. | within Category |
| | Ulcerative Colitis: Acute haemorrhagic ulcerative colitis; Colitis ulcerative; Proctitis ulcerative | Listing: |
| | IBD Non-Specific Terms: The PTs in this category are listed in Appendix 11 | TEAE |
| | 1 100 Non-openic Terms. The FF3 in this category are listed in Appendix 11 | |

| Special Safety | | |
|---|---|---|
| Topic | Definition / Derivation | Analysis / Summary / Listing |
| Interstitial | Interstitial lung disease is defined using the following terms: | Listing: |
| Lung Disease | Narrow terms in the interstitial lung disease SMQ (20000042) | TEAE |
| | • The following 6 PTs from eosinophilic pneumonia SMQ (20000157): | |
| | <ul> <li>Angiolymphoid hyperplasia with eosinophilia (Narrow)</li> </ul> | |
| | <ul> <li>Eosinophilic bronchitis (Narrow)</li> </ul> | |
| | Hypereosinophilic syndrome (Narrow) | |
| | o Loeffler's syndrome (Narrow) | |
| | o Pulmonary eosinophilia (Narrow) | |
| | o Pulmonary vasculitis (Narrow) | |

Abbreviations: AE = adverse event; ALT = alanine aminotransferase; AST = aspartate aminotransferase; CEC = Central Events Committee; eCRF = electronic case report form; eDISH = Evaluation of Drug-Induced Serious Hepatotoxicity; HLT = High Level Term; MedDRA = Medical Dictionary for Regulatory Activities; OI = opportunistic infection; PT = preferred term; SAE = serious adverse event; SMQ = standardized MedDRA query; SOC = System Organ Class; TB = tuberculosis; TEAE = treatment-emergent adverse event; ULN = upper limit of normal.

# 6.13.8. Immunogenicity

#### 6.13.8.1. Definitions and Terms

The following sample- and patient-related definitions and parameters will be used to describe the immunogenicity data.

#### 6.13.8.1.1. Sample Category Definitions

Samples are classified into the following categories:

- Unevaluable sample: Sample could not be tested for anti-drug antibody (ADA) due to sample loss, mishandling, or errors in collection, processing, storage, etc.
- Antidrug antibody (ADA) Positive sample: The presences of ADA is detected and confirmed. The samples are reported as positive. If the sample is positive, a titer value is reported.
- Neutralizing anti-drug antibody (NAb) Positive sample: NAb are reported as detected
- Antidrug antibody (ADA) Negative sample: The presence of ADA is not detected and the assay drug tolerance level is not exceeded.
- Neutralizing anti-drug antibody (Nab) Negative sample: The presence of NAb is not detected and the assay drug tolerance level is not exceeded.
- **Inconclusive sample:** when ADA/NAb is not detected in a sample but drug is present in the same sample at a level that can cause interference in the ADA/NAb detection method. The negative ADA/NAb result cannot be confirmed and the sample was considered inconclusive.
  - Confirmation of a negative ADA result was based on ixekizumab concentrations.

Figure RHBF.6.1 illustrates the relationship of some of the above terms.



Abbreviation: ADA = anti-drug antibody.

Figure RHBF.6.1. Sample definitions.

#### 6.13.8.1.2. Patient Category Definitions

The following categories are applied to patients based on the classification of their samples:

- Unevaluable patient: a) a patient with no evaluable baseline sample and/or no evaluable postbaseline samples; b) a patient with an evaluable baseline sample but no evaluable postbaseline sample; c) a patient with no evaluable baseline sample, but whose evaluable postbaseline values are all ADA positive or a mix of positive and negative. (Note: If all post-baseline samples are negative, the patient is considered 'evaluable' and will be classified as ADA-negative.)
- Evaluable patient: a) Patient with an evaluable baseline sample and at least 1 evaluable post-baseline sample (that is, sample after administration of study drug); b) patient with no evaluable baseline sample whose evaluable post-baseline samples are all ADA negative.

Figure RHBF.6.2 illustrates the relationship of the above terms.



Figure RHBF.6.2. Patient categories (evaluable/unevaluable) based on sample status at baseline and post-baseline.

## 6.13.8.1.3. Definitions for Clinical Interpretation of Assay Results

- **Baseline:** For immunogenicity analyses during Period 2, Period 3, and Period 4, baseline is the last nonmissing observation on, or prior to, the date of the first injection of study treatment of ixekizumab (Week 0).
- Baseline ADA positive (preexisting antibody): ADA detected in a sample collected at baseline.
- Treatment-emergent antidrug antibody positive: a) a patient with a ≥4-fold increase over a positive baseline antibody titer (Tier 3); or b) for a negative baseline titer, a patient with an increase from the baseline to a level of ≥1:10.
- Baseline ADA-negative: ADA is not detected in a sample collected at baseline.
- Treatment-emergent antidrug antibody inconclusive patient: A patient without a TE-ADA positive sample and with at least one sample for which drug levels may interfere with the ADA assay.
- Treatment-emergent antidrug antibody negative patient: A patient who is evaluable for TE-ADA and is not either TE-ADA positive or TE-ADA inconclusive.

Figure RHBF.6.3 illustrates the relationship of some of these terms.



Abbreviation: ADA = anti-drug antibody.

Figure RHBF.6.3. Relationship of terms for clinical interpretation of assay results for evaluable patients.

• **Incidence of TE-ADA:** Patients with TE-ADA as a proportion of the evaluable patient population during the treatment period. This excludes unevaluable patients.

All ADA positive samples will be evaluated for NAb. Definitions for NAb patient status will be defined as follows:

- Neutralizing anti-drug antibody-positive patient: A patient where a NAb positive result is detected for ≥1 TE-ADA positive samples.
- Neutralizing anti-drug antibody-inconclusive patient: A patient without a NAb positive sample and with at least one sample for which drug levels may interfere with the NAb assay.
- **Neutralizing anti-drug antibody-negative patient:** A patient who is evaluable for NAb and is not either NAb positive or NAb inconclusive.

A flow chart that reflects the connection between the analytical test results and the clinical interpretation based on the definitions is shown in Figure RHBF.6.4.



Abbreviation: ADA = anti-drug antibody; NAb = neutralizing anti-drug antibody; PK = pharmacokinetic.

Figure RHBF.6.4. Flow chart of ADA assessment with clinical interpretation of the various result possibilities.

# 6.13.8.2. Immunogenicity Analyses

Immunogenicity will be summarized for evaluable patients for (unless otherwise noted):

- Period 2 (initial open-label treatment period population)
- Period 3 (randomized withdrawal safety population)
- Relapse period (relapse population)

- Combined Period 2 and Period 3 (ixekizumab 80 mg Q2W-treated patients from the randomized withdrawal safety population and nonrandomized population)
- Period 4 (post-treatment follow-up period population).

Immunogenicity evaluable patients will be identified as TE-ADA positive, TE-ADA negative, or TE-ADA inconclusive, according to the definitions provided in Section 6.13.8.1.2 and further grouped into TE-ADA status groups and time-varying TE-ADA status groups:

#### **TE-ADA Status Groups:**

- **Treatment-emergent antidrug antibody** status (positive, negative, or inconclusive);
- Neutralizing anti-drug antibody status (positive, negative, or inconclusive) for TE-ADA positive patients
- **Treatment-emergent antidrug antibody** titer groups for TE-ADA positive patients:
  - o Low Titer: TE-ADA titer value (LOCF) < 1:160
  - o Moderate Titer: TE-ADA titer value (LOCF) ≥1:160 and < 1:1,280
  - o High Titer: TE-ADA titer value (LOCF) ≥1:1,280

#### **Time-varying TE-ADA Status Groups:**

Individual ADA samples will be ascribed into 3 different dichotomous variables as explained in Table RHBF.6.7. Each variable has possible values of a 'greater-TE-ADA status' or a 'lesser-TE-ADA status,' in the sense that the level of TE-ADA detected in the greater-TE-ADA category is higher than in the lesser-TE-ADA category.

**Table RHBF.6.7.** TE-ADA Status Dichotomous Variables for AE analysis

| TE-ADA Status Dichotomous<br>Variable | Greater-TE-ADA Status | Lesser-TE-ADA Status |
|---|---|---|
| TE-ADA positive | TE-ADA positive | not TE-ADA positive |
| TE-ADA moderate-to-high | TE-ADA positive with moderate titer or high titer | not TE-ADA positive, or TE-ADA positive with low titer |
| TE-ADA high status | TE-ADA positive with high titer | not TE-ADA positive, or TE-ADA positive with low or moderate titer |

#### TE-ADA Status Dichotomous Variables for AE analysis (Abbreviations and Footnotes)

Abbreviations: AE = adverse events; ADA = antidrug antibody; TE-ADA = treatment-emergent antidrug antibody. Note: For purpose of this analysis, TE-ADA Inconclusive is taken to be "not TE-ADA positive."

Note: A TE-ADA low is defined as a TE-ADA positive with a titer value < 1:160; a TE-ADA moderate is defined as a TE-ADA positive with a titer value ≥1:160 and < 1:1,280; and a TE-ADA high is defined as a TE-ADA positive with a titer value ≥1:1,280.

For each TE-ADA status dichotomous variable, a time-varying TE-ADA status will be computed. At time *t* the TE-ADA status is taken to be the highest of the TE-ADA values bracketing time *t*. More formally, the TE-ADA status at time *t* is given by the greater of (a) the TE-ADA status at the most-recent postbaseline measurement prior to *t*, and (b) the TE-ADA status at the first TE-ADA postbaseline measurement at or after time *t*. In this computation, 'greater' is given by the greater-TE-ADA status of Table RHBF.6.7. If there is no value satisfying criterion (a), then the value (b) is used. Similarly, if there is no value (b), then the value (a) is used.

For each TE-ADA status dichotomous variable, patients will be categorized according to whether they were (i) always in lesser-TE-ADA status postbaseline or (ii) at some point postbaseline, were in greater-TE-ADA status.

#### 6.13.8.2.1. Analyses of Characteristics of ADA Immune Response

The analyses of characteristics of ADA response will be conducted on all immunogenicity evaluable patients within the Initial Open-Label Treatment, Randomized Double-Blind Withdrawal Period, Combined Open-Label Treatment Period and Randomized Double-Blind Withdrawal Periods, Relapse Period, and the Post-Treatment Follow-up Period. Patients will be analyzed according to the treatment to which they were assigned.

The overall frequency and percentage (incidence) of patients will be summarized for the TE-ADA status groups and the time-varying TE-ADA status groups. Scheduled visits, unscheduled visits, and repeat measurements will be included.

The time to the development of TE-ADAs (TE-ADA positive, low titer, moderate titer, high titer, and NAb positive) will be calculated as follows:

Time to development of TE-ADAs/NAb (in weeks) = (Date of development of TE-ADAs/NAb – Date of first injection of study treatment + 1) / 7.

If a patient has not developed TE-ADAs/NAbs, they will be censored at the date of the last immunogenicity assessment. If a patient does not have any postbaseline assessments for immunogenicity, they will be censored at the date of randomization.

Descriptive statistics, including 25th percentile, 50th percentile (median), 75th percentile, and corresponding 95% CIs as well as probability of TE-ADA/NAb positive by endpoint summarized by treatment group, will also be provided if sufficient data is present. A Kaplan-Meier plot of the time to development of treatment-emergent ADA/NAb will be presented by treatment group, also if sufficient data is present. The log-rank test will be used to test the null

hypothesis against the alternate hypothesis that the time to TE-ADA/NAb is not equal between ixekizumab and placebo. Caution should be exercised in the interpretation of time-to event analyses, and related statistics, given the limited sampling scheme for immunogenicity testing.

For each TE-ADA status dichotomous variable (as defined in Table RHBF.6.7), summaries will be provided of the total postbaseline time in the greater-TE-ADA status for patients who were at some point postbaseline in the greater-TE-ADA status group. Postbaseline time in greater-TE-ADA status for each patient will be aggregated.

A by-patient listing to include treatment, visit date, visit, ADA result, TE-ADA result, NAb result, ADA titer value, ixekizumab concentration, ADA and NAb inconclusive results will also be provided, for patients with any one sample of ADA (or NAb) positive or inconclusive.

### 6.13.8.2.2. Analyses of Treatment-Emergent ADA Effects on Efficacy

Analyses will be performed to examine how patient TE-ADA effects time-to relapse in the randomized withdrawal ITT population by the TE-ADA status groups. The Kaplan-Meier product limit method will be used to estimate the survival curves for time-to relapse. A Coxproportional hazards model with treatment group, TE-ADA status group and the interaction of treatment group-by-TE-ADA status group included as factors in the model will be used to test the interaction of treatment group-by-TE-ADA status group. Additionally, the Kaplan-Meier product limit method will be used to estimate the survival curves for time-to relapse.

Analyses will also be performed to examine how patient TE-ADA effects the proportion of patients who relapse by 40 weeks of randomized treatment in the randomized withdrawal ITT population by the TE-ADA status groups. A logistic regression model with treatment group, TE-ADA status group and the interaction of treatment group-by-TE-ADA status group included as factors in the model will be used to test the interaction of treatment group-by-TE-ADA status group.

Analyses will also be performed to examine how patient TE-ADA effects the proportion of patients with 20% and 50% improvement in American College of Rheumatology criteria (ACR20 and ACR50) at the last observation in the initial open-label treatment period population and at 40 weeks of randomized treatment in the randomized withdrawal ITT population by the TE-ADA status groups. For the initial open-label treatment period population, the TE-ADA status groups will be summarized for the ixekizumab 80 mg Q2W treatment group. For the randomized withdrawal ITT population, a logistic regression model with treatment group, TE-ADA status group and the interaction of treatment group-by-TE-ADA status group included as factors in the model will be used to test the interaction of treatment group-by-TE-ADA status group.

The p-value associated with the interaction terms will be used to assess if the treatment group effect is consistent across TE-ADA status group. When the interaction term is statistically significant, the association between responder status and the treatment group depends, in some manner, on the status group. The interaction will be tested at the 10% significance level. If any group within the subgroup (for example, yes, no) is <10% of the total population, only

descriptive statistics will be provided for that subgroup (that is, no inferential testing). Treatment group differences will be evaluated within each subgroup regardless of whether the interaction is statistically significant.

#### 6.13.8.2.3. Analyses of Treatment-Emergent ADA on Specific Adverse Events

The analyses of TE-ADA effects on safety will be conducted on all immunogenicity evaluable patients within the Initial Open-Label Treatment Period, Randomized Double-Blind Withdrawal Period, and the Combined Open-Label Treatment and Randomized Double-Blind Withdrawal Periods. Patients will be analyzed according to the treatment to which they were assigned.

Adverse events of special interest of allergic reaction/hypersensitivity (anaphylaxis and nonanaphylaxis) and of injection-site reactions will be included in an assessment of AE to TE-ADA over time. See Table RHBF.6.6 for the definitions of the AESIs. Timing of an AE will be taken to be the reported AE start date.

For each TE-ADA status dichotomous variable (as defined in Table RHBF.6.7), patients will be categorized according to whether they were (i) always in lesser-TE-ADA status postbaseline or (ii) at some point postbaseline, were in greater-TE-ADA status. For each AESI, within the time-varying TE-ADA status groups, a summary will be provided of the number of patients who had no event, events only while in lesser-TE-ADA status for group (i), or – for group (ii) – at least one event while in greater-TE-ADA status.

Additionally, summaries will be provided of the total number of AESI events (with unique start dates) by time-varying TE-ADA status groups at the event date. The summaries will aggregate time respectively in greater-TE-ADA status and in lesser-TE-ADA status, along with the event rates (rates per 100 patient-years) relative to those aggregate times.

By-patient listings will be provided of patients with TE-ADA who experience a treatmentemergent allergic reaction/hypersensitivity reaction or an injection site reaction.

# 6.14. Subgroup Analyses

# 6.14.1. Efficacy Subgroup Analysis

Subgroup analyses will be conducted for time-to relapse and the proportion of patients who relapse by 40 weeks of randomized treatment in the randomized withdrawal ITT population during Period 3.

For the time-to-relapse, the Kaplan-Meier product limit method will be used to estimate the survival curves for time-to relapse. Analyses will be performed using a Cox-proportional hazards model with treatment group, subgroup, and the interaction of treatment group-by-subgroup included as factors in the model.

For the proportion of patients who relapse, a logistic regression model with treatment, subgroup, and the interaction of treatment group-by-subgroup included as factors will be used.

The treatment group-by-subgroup interactions will be tested at the significance level of 0.10. If any group within the subgroup (for example, yes, no) is <10% of the total population, only

descriptive statistics will be provided for that subgroup (that is, no inferential testing). Treatment group differences will be evaluated within each category of the subgroup using log-rank test without stratifications or Fisher's exact test, regardless of whether the interaction is statistically significant.

Subgroups to be evaluated include:

- Demographic subgroups:
  - Age group: <65 years,  $\ge65$  years to <75 years,  $\ge75$  years
  - o Age group: <40 years, ≥40 years
  - o Gender (male, female)
  - o Race: AI, AS, BL, NH, WH, MU
  - o Ethnicity: Hispanic or Latino, Not Hispanic or Latino
  - o Weight category: <100 kg, ≥100 kg
  - Weight category:  $<80 \text{ kg}, \ge80 \text{ kg to } <100 \text{ kg}, \ge100 \text{ kg}$
  - O BMI category: underweight (<18.5 kg/m²); normal (≥18.5 to <25 kg/m²); overweight (≥25 to <30 kg/m²); obese (≥30 to 40 kg/m²); extreme obese (≥40 kg/m²)</p>
- Geographic region subgroups:
  - o Geographic region: US, Europe, Rest of the World
- Baseline severity subgroups:
  - o C-reactive protein (mg/dL):  $\leq 6, > 6$
  - o Duration of PsA (years): 0 to  $<5, \ge 5$
  - o Baseline psoriatic lesion(s) involving BSA  $\geq$ 3%: yes or no)
  - o Moderate to severe psoriasis (defined as PASI  $\geq$ 12, sPGA  $\geq$ 3, and BSA  $\geq$ 10%): yes, no
  - o Enthesitis (LEI score >0 or SPARCC >0): yes or no
  - o Dactylitis (LDI-B score >0): yes or no
- Psoriatic arthritis therapy subgroups:
  - o Previous cDMARD use at the time of randomization (past use, current use) for the randomized withdrawal ITT population
  - Methotrexate use at the time of randomization (none, past use, current use) for the randomized withdrawal ITT population

Additional subgroup analyses on efficacy may be performed as deemed appropriate and necessary.

# 6.14.2. Safety Subgroup Analysis

Subgroup analyses will be conducted for common TEAEs and AESIs of allergy/hypersensitivity, infections, and injection site reactions for the initial open-label treatment period population during Period 2 and the randomized withdrawal safety population during Period 3.

The most common TEAEs and AESIs will be presented by MedDRA PT nested within SOC (SMQ or High Level Term where specified in Section 6.13.7). A logistic regression model will be used to test the treatment group-by-subgroup interaction for the randomized withdrawal safety population. The model will include explanatory variables of treatment group, subgroup, and treatment group by-subgroup interaction. The interaction test will be evaluated at the 0.10 significance level. If any group within the subgroup (for example, yes, no) is <10% of the total population, only descriptive statistics will be provided for that subgroup (that is, no inferential testing). Treatment group differences will be evaluated within each category of the subgroup, regardless of whether the interaction is statistically significant. Treatment differences will be assessed within the subgroups using the Fisher's exact test.

Subgroups to be evaluated include:

- Demographic subgroups:
  - o Age group: <65 years,  $\ge65$  years to <75 years,  $\ge75$  years
  - o Age group: <40 years, ≥40 years
  - o Gender (male, female)
  - o Race: AI, AS, BL, NH, WH, MU
  - o Ethnicity: Hispanic or Latino, Not Hispanic or Latino
  - o Weight category: <100 kg, ≥100 kg
  - $\circ$  Weight category:  $<80 \text{ kg}, \ge80 \text{ kg to } <100 \text{ kg}, \ge100 \text{ kg}$
  - o Body mass index category: underweight (<18.5 kg/m²); normal (≥18.5 and <25 kg/m²); overweight (≥25 to <30 kg/m²); obese (≥30 to 40 kg/m²); extreme obese (≥40 kg/m²)
- Geographic region subgroups:
  - Geographic region at baseline for the initial open-label treatment period population: Europe, US, Rest of the World
- Psoriatic arthritis therapy subgroups:
  - Previous cDMARD use at the time of randomization (past use, current use) for the randomized withdrawal safety population
  - Methotrexate use at the time of randomization (none, past use, current use) for the randomized withdrawal safety population.

# 6.15. Analysis for Australian Submission

Efficacy analysis may be conducted if needed to meet the Pharmaceutical Benefits Advisory Commission (PBAC) criteria for a regulatory submission or request. The time-to relapse and proportion of patients with relapse will be analyzed using a PBAC randomized withdrawal ITT population for Period 3. Data will be analyzed using the analysis methods defined in Section 6.1.2.1 for the time-to analysis and categorical analyses.

The PBAC randomized withdrawal ITT population is a subset of the randomized withdrawal population and is defined as all randomized patients in Period 3 with:

- 1. An elevated CRP > 15 mg/L
- 2. An active joint count of at least 20 active (swollen and tender) joints or at least 4 major active joints: elbow, wrist, knee, ankle, shoulder and/or hip
- 3. Psoriatic arthritis that has not responded to adequate trials of at least 2 cDMARDs, administered either individually or in combination for a minimum of 3 months

# 6.16. Analysis for United Kingdom National Institute for Health and Care Excellence Submission

Efficacy analysis will be conducted to meet the UK's National Institute for Health and Care Excellence (NICE) criteria. The time-to relapse and proportion of patients with relapse will be analyzed using a NICE randomized withdrawal ITT population for Period 3. Data will be analyzed using the analysis methods defined in Section 6.1.2.1 for the time-to analysis and categorical analyses.

The NICE randomized withdrawal ITT population is a subset of the randomized withdrawal population and is defined as all randomized patients in Period 3 with:

- 1. Peripheral arthritis with  $\geq 3$  tender joints and  $\geq 3$  swollen joints
- 2. Psoriatic arthritis that has not responded to adequate trials of at least 2 cDMARDs, administered either individually or in combination.

#### 6.17. Protocol Deviations

Protocol deviations will be identified throughout the study. Important protocol deviations are defined as those deviations from the protocol likely to have a significant impact on the completeness, accuracy, and/or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being. All important protocol deviations identified are reviewed by the study team prior to database lock.

Table RHBF.6.8 includes the categories and subcategories of important protocol deviations, the source of identification for the deviation, and the statistical programming guidance for the CSR.

A by-patient listing of important protocol deviations will be provided for all entered patients.

The number and percentage of patients having important protocol deviation(s) will be summarized within category and subcategory of deviations by treatment group for:

- Period 2 (initial open-label treatment period population)
- Period 3 (randomized withdrawal ITT population).

In addition, other protocol deviations considered important for reporting purposes derived from manual review of study records as recorded via monitoring reports or other site compliance monitoring will be summarized. These may include

- Ethics review board (ERB) approval not obtained
- Follicle-stimulating hormone (FSH) not assessed
- Good Clinical Practice guidelines not followed by principal investigator (PI)
- Hepatitis monitoring not done
- Improper consent/re-consent (not timely, wrong version, not signed)
- Physical examination not performed
- Postbaseline pregnancy test not performed
- Quick Inventory of Depressive Symptomatology not assessed
- Serious adverse events not reported on time
- Tuberculosis test collected late
- Tuberculosis test not performed
- Temperature excursion at site
- Unqualified study personnel performing procedures
- One hour post-dose vitals not performed at Visit 2
- Assessment not performed by Independent Assessor
- Unauthorized use of electronic patient reported outcomes (ePRO) device credentials
- Vital signs not performed.

This list is not conclusive and additional other important protocol deviations may be identified.

 Table RHBF.6.8.
 Identification and Action of Important Protocol Deviations

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| Patient did not give written consent | | | |
| Informed consent form must be signed before any protocol procedures begin (Proper order of informed consent signature, randomization, and therapy start dates). Failed to meet study inclusion criteria but was e | Monitor and Stats | Either from monitor's list, or, If patient informed consent date is after Visit 1 date | Yes |
| [1] Age <18 years | Monitor and Stats | From monitor's list. Stats may program preliminarily based on data for age <18 at Visit 1, but deviation must be confirmed and sourced by monitor. This is because only birth year is collected, and age is calculated by imputation. | Yes |
| [1a] Male patients did not use a reliable method of birth control | Monitor | From monitor's list. | Yes |
| [1b] Lack of confirmation of non-pregnant status prior to randomization at visit 2 | Monitor | From monitor's list. | Yes |
| [2] No confirmed diagnosis of PsA of at least 6 months prior to baseline or did not meet CASPAR criteria | Monitor and Stats | Review monitor's list. Check time since PsA diagnosis and CASPAR criteria. | Yes |
| [3] <3 tender or <3 swollen joints at Visit 1 or Visit 2 | Monitor and Stats | Review monitor's list. Check if TJC68 <3 or SJC66 <3 either at Visit 1 or at Visit 2 | Yes |
| [4] Never been treated with a cDMARD or has been treated with a cDMARD and no documentation of inadequate response with a minimum of 12 weeks or intolerance | Monitor | From monitor's list. | Yes |
| [5] No active or history of plaque psoriasis | Monitor and Stats | Review monitor's list. Check if the answer to current Psoriasis is No AND patient contains no record in medical history where: 1. (the reported term for medical history = "PSORIASIS DISEASE" and category for medical history = "PRIMARY DIAGNOSIS") or 2. (the dictionary derived term = "PSORIASIS" and category for medical history = "PRE-EXISTING") | Yes |

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| | | CONDITION") or 3. (reported term for medical history = "PLAQUE PSORIASIS" and category for medical history = "PRE-EXISTING CONDITION")] | |
| Met study exclusion criteria but was enrolled in | to the study | | |
| [7] Prior or current use of bDMARDs or biologics | Monitor | Monitor's list | Yes |
| [8] Previous or current medication exposure at Visit 1 to LY2439821 or IL-17 antagonists or previous participation in the current study. (Note: See protocol for patients who may be allowed to re-screen.) | Monitor | Monitor's list | Yes |
| [9] Have history of drug-induced Ps | Monitor | Monitor's list | Yes |
| [10] Inadequate response to ≥4 cDMARDs prescribed alone or in combination for 3 months | Monitor and Stats | Either from monitor's list, or, If a patient used for least 90 days any 4 or more of the following previous therapies category or non-biologic systemic agent subcategory: MTX, Leflunomide, Azathioprine, Cyclosporine, Hydroxychloroquine, Gold Salts, Sulfasalazine | Yes |
| [11] & [12] Use of cDMARDs within the washout periods or using >1 at entry into the study, or using DMARDs at doses outside of specified range | Monitor | Monitor's list | Yes |
| [13] Have discontinued leflunomide within 4 weeks prior to baseline or from 4 to 12 weeks prior without drug elimination procedure | Monitor and Stats | Monitor's list, or, If the difference between Visit 2 date and medication end date <28 days for previous therapy, Leflunomide | Yes |
| [14] Use of oral corticosteroids >10 mg/day of prednisone or equivalent, use of variable doses within 4 weeks prior to baseline | Monitor | Monitor's list | Yes |
| [15] Have received parenteral glucocorticoids within 6 weeks prior to baseline or if use is anticipated during initial open-label treatment period (Period 2) of the study | Monitor and Stats | Monitor's list, or, If a patient has a reported previous therapy of parenteral glucocorticoids with and end date <42 days prior to the Visit 2 date | Yes |
| [16] Concomitant use of NSAIDs or | Monitor | Monitor's list | Yes |

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| cyclooxygenase -2 inhibitors unless on a stable dose for at least 2 weeks prior to baseline | | | |
| [17] Use of opiate analgesics >30 mg/day of morphine or equivalent or variable doses within 6 weeks prior to baseline | Monitor and Status | Monitor's list, or, If a patient has either a reported previous therapy of opiate analgesics or a concomitant medication with ATC codes of N02AA with a start or end date of <42 days prior to Visit 2 date. | Yes |
| [18] Received systemic non-biologic psoriasis therapy (including, but not limited to, oral psoralens and ultraviolet A [PUVA] light therapy; cyclosporine; corticosteroids; MTX; oral retinoids; mycophenolate mofetil; thioguanine; hydroxyurea; sirolimus; azathioprine; fumaric acid derivatives; or 1, 25 dihydroxy vitamin D3 and analogues) or phototherapy (including either oral and topical PUVA light therapy, ultraviolet B [UVB] or self-treatment with tanning beds or therapeutic sunbathing) within 4 weeks prior to baseline (Visit 2). or had topical psoriasis treatment (including, but not limited to, corticosteroids, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, emollients and other non-prescription topical products containing urea, >3% salicylic acid, or alpha- or beta-hydroxyl acids, and medicated shampoos [for example those that contain >3% salicylic acid, corticosteroids, coal tar, or vitamin D3 analogues]) within the previous 2 weeks prior to baseline (Week 0; Visit 2). Note WHO Group 1 weak potency (such as hydrocortisone) topical TRT are allowed. | Monitor and Stats | Monitor's list, or, If the patient has any record with an end date ≤28 days of the Visit 2 date for Phototherapy for previous therapy If the patient has any concomitant medications with an end date that is on or prior to Visit 2 date, and ≤28 days prior to the Visit 2 date for oral medications with the following ATC codes: D05B, D05BA, D05BB, D05BX). If the patient has any concomitant medications with an end date that is on or prior to Visit 2 date, and ≤14 days prior to the Visit 2 date for topical medications with the following ATC codes: D07AC, D07AD, D07BC, D07BD, D07CC, D07CD, D07XC, D07XD, A11CC, D05AA, D05AC, D05AD, D05AX, D05BB, L04AD, D11AC, D07AB, D02AF, D02BB. | Yes |

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| [19] Use of tanning beds/booths for at least 4 weeks (or 28 days) prior to Visit 2 for patients with plaque psoriasis. | Monitor | Monitor's list | Yes |
| [20] Have a known allergy or hypersensitivity to any biologic therapy that would pose an unacceptable risk to the patient if participating in this study. | Monitor | Monitor's list | Yes |
| [21] Ever received natalizumab or other agents that target alpha-4-integrin | Monitor | Monitor's list | Yes |
| [22] Have been exposed to a live vaccine within 12 weeks prior to Visit 2 or intend to have a live vaccination during the course of the study, or participated in a BCG (12 months prior to baseline) or other vaccine clinical study within 12 weeks prior to Visit 2 | Monitor | Monitor's list | Yes |
| [23] Had a BCG (12 months prior to baseline), or intent to have this vaccine during the study or within 12 months of completion of the study | Monitor | Monitor's list | Yes |
| [24] Have diagnosis of other inflammatory arthritic syndrome | Monitor | Monitor's list | Yes |
| [25] Have active Crohn's disease or active ulcerative colitis | Monitor | Monitor's list | Yes |
| [26] Have current diagnosis of fibromyalgia | Monitor | Monitor's list | Yes |
| [27] Have a chronic pain condition what would confound evaluation of the patient | Monitor | Monitor's list | Yes |
| [28] Evidence of active vasculitis or uveitis | Monitor | Monitor's list | Yes |
| [29] Surgical treatment of joint within 8 weeks prior to baseline or will require such up to Week 24 | Monitor | Monitor's list | Yes |
| [30] Had any major surgery within 8 weeks prior to baseline (Week 0; Visit 2), or will require such during the study that, in the opinion of the | Monitor | Monitor's list | Yes |

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| investigator in consultation with Lilly or its designee, would pose an unacceptable risk to the patient. | | | |
| [31] Have current or a history of lymphoproliferative disease | Monitor | Monitor's list | Yes |
| [32] Have active or history of malignant disease within the 5 years prior to baseline (Visit 2). Patients with successfully treated basal-cell carcinoma [no more than 3], squamous-cell carcinoma of the skin (no more than 2), within the 5 years prior to Visit 2 may participate in the study. | Monitor | Monitor's list | Yes |
| [33] Presence of significant uncontrolled cerebro-<br>cardiovascular (for example, MI, unstable angina,<br>unstable arterial hypertension, moderate-to-severe<br>NYHA class III/IV heart failure, or<br>cerebrovascular accident [CVA]), respiratory,<br>hepatic, renal, gastrointestinal, endocrine,<br>hematologic, neurologic or neuropsychiatric<br>disorders, or abnormal laboratory values at<br>screening that, in the opinion of the investigator,<br>pose an unacceptable risk to the patient if<br>participating in the study or of interfering with the<br>interpretation of data. | Monitor | Monitor's list | Yes |
| [34] Have had fluid overload, MI, or new-onset ischemic heart disease, uncompensated heart failure, or in the opinion of the investigator other serious cardiac disease within 12 weeks prior to Visit 2. | Monitor | Monitor's list | Yes |
| [35] Have history of a suicide attempt, have a score of 3 on Item 12 (Thoughts of Death or Suicide) of the QIDS-SR16 at screening (Visit 1) | Monitor and Stats | Monitor's list, or, If a patient has a score of 3 for the 'thoughts of death or suicide' on the QIDS-SR16 at Visits 1 or 2. | Yes |

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| or baseline (Week 0; Visit 2), or are clinically judged by the investigator to be at risk for suicide. | | | |
| [36] Have serious infection (for example, pneumonia, cellulitis), been hospitalized, received IV antibiotics for an infection within 12 weeks of Visit 2, or had a serious bone or joint infection within 24 weeks prior to baseline, or have ever had an infection of an artificial joint, or are immunocompromised to an extent such that participation in the study would pose an unacceptable risk to the patient. | Monitor | Monitor's list | Yes |
| [37] have or had an opportunistic infection characteristic of an immunocompromised host and/or that occurs with increased incidence in an immunocompromised host (including but not limited to <i>Pneumocystis jirovecii</i> pneumonia, histoplasmosis, coccidioidomycosis, or cryptococcosis) or have a known immunodeficiency | Monitor | Monitor's list | Yes |
| [38] have or had a herpes zoster or any other clinically apparent varicella-zoster virus infection within 12 weeks of baseline (Week 0, Visit 2) | Monitor | Monitor's list | Yes |
| [39] Evidence or suspicion of active or latent TB (refer to Protocol Section 10.3.2.2 for details on determining full TB exclusion criteria). | Monitor | Monitor's list | Yes |
| [40] within 4 weeks of baseline (Week 0, Visit 2), have any active or recent infection other than those mentioned in exclusion criteria 36-39 that, in the opinion of the investigator, would pose an unacceptable risk to the patient if participating in the study; these patients may be rescreened once ≥4 weeks after documented resolution of | Monitor | Monitor | Yes |

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| symptoms | | | |
| [41] Body temperature ≥38 degrees Celsius (100.5°F) at Visit 2 or at rescreen (1 time) ≥4 weeks after documented resolution of elevated temperature | Monitor and Stats | Monitor's list, or,<br>If a patient's temperature is ≥38 digress Celsius at Visit 2 | Yes |
| Important Protocol Deviation | Source to Identify Protocol | Statistical Programming Guidance for Clinical Study | Exclude |
| Category/Subcategory | Deviation | Report | from the PPS? |
| [42] Have uncontrolled arterial hypertension characterized by a systolic blood pressure (BP) >160 mm Hg or diastolic BP >100 mm Hg. Determined by 2 consecutive elevated readings | Monitor and Stats | Monitor's list, or, If a patients SBP > 160 or DBP > 100 mmHg at Visit 1 | Yes |
| [43] Are positive for human immunodeficiency virus (HIV) serology (positive for HIV antibody) | Monitor and Stats | Monitor's list, or,<br>If a patients laboratory tests at Visit 1 indicate they are positive<br>for HIV antibody | Yes |

| Important Protocol Deviation Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| [44] Have evidence of or test positive for hepatitis B by any of the following criteria: 1) positive for hepatitis B surface antigen (HBsAg+); 2) positive for anti-hepatitis B core antibody (HBcAb+) and negative for anti-hepatitis B surface antibody (HBsAb-); 3) positive for anti-hepatitis B core antibody (HBcAb+) and positive for anti-hepatitis B surface antibody (HBsAb+) with a concentration of HBsAb <200 mIU/mL; or 4) HBcAb+, HBsAb+ (regardless of HBsAb level), and positive for serum hepatitis B virus (HBV) DNA. (Note: Patients who are negative for hepatitis B surface antigen (HBsAg-), HBcAb+, HBsAb+ with a concentration of HBsAb ≥200 mIU/mL, and negative for serum HBV DNA may participate in the study. Patients who meet these criteria at screening will be identified by the central laboratory and monitored during the study as detailed in Section 10.3.3.3 of the RHBF protocol). | Monitor and Stats | Monitor's list, or, If a patients laboratory tests at Visit 1 indicate they are positive for hepatitis B | Yes |
| [45] Have evidence of or test positive for hepatitis C virus (HCV). A positive test for HCV is defined as: 1) positive for hepatitis C antibody (anti-HCV Ab), and 2) positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction). | Monitor and Stats | Monitor's list, or, If a patient's laboratory tests at Visit 1 indicate they are positive for hepatitis C virus | Yes |
| [46] Have clinical laboratory test results at screening that are outside the normal reference range for the population and are considered clinically significant, and/or have any of the following specific abnormalities: | Monitor and Stats | Monitor's list, or, If a patients laboratory tests at Visit 1 indicate any of the following: 1. Neutrophil count <1500 cells/µL 2. Lymphocyte count <800 cells/µL | Yes |

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| [46a] Neutrophil count <1500 cells/μL [46b]Lymphocyte count <800 cells/μL [46c] Platelet count <100,000 cells/μL [46d]Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times the upper limit of normal (ULN) [46e] Total white blood cell (WBC) count <3000 cells/μL [46f] Hemoglobin <8.5 g/dL (85.0 g/L) for male patients and <8.0 g/dL (80 g/L) for female patients [46g]Serum creatinine >2.0 mg/dL. | | <ol> <li>Platelet count &lt;100,000 cells/µL</li> <li>AST or ALT &gt;2.5 times the ULN</li> <li>Total WBC &lt;3000 cells/µL</li> <li>Hemoglobin &lt;8.5 g/dL for male patients and &lt;8 g/dL for female patients</li> <li>Serum creatinine &gt;2 mg/dL</li> </ol> | |
| [47] Have electrocardiogram (ECG) abnormalities that are considered clinically significant and would pose an unacceptable risk to the patient if participating in the study | Monitor | Monitor's list | Yes |
| [48] Have any other condition that precludes the patient from following and completing the protocol. | Monitor | Monitor's list | Yes |
| [49] have donated blood of more than 1 unit (approximately 500 mL) within the last 4 weeks or intend to donate blood during the course of the study | Monitor | Monitor's list | Yes |
| [50] Are women who are lactating or breastfeeding | Monitor | Monitor's list | Yes |
| [51] are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted. | Monitor | Monitor's list | Yes |
| [52] are employees of Lilly or its designee or are employees of third-party organizations (TPOs) | Monitor | Monitor's list | Yes |

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| involved in the study | | | |
| [53] are currently enrolled in a clinical trial involving an investigational product or nonapproved use of a drug or device (other than the investigational product used in this study) or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study | Monitor | Monitor's list | Yes |
| [54] have been discontinued from a clinical trial involving an investigational product or nonapproved use of a drug or device within the last 4 weeks or a period of at least 5 half-lives of the last administration of the drug, whichever is longer | Monitor | Monitor's list | Yes |
| Met study discontinuation criteria but continued | | No. 14 2 11 4 | 37 |
| [D1] Neutrophil (segmented) counts: $<500 \text{ cells/}\mu\text{L}$ ; or $\geq500 \text{ and} <1000 \text{ cells/}\mu\text{L}$ (from 2 test results; the second test must be performed within 1 week from knowledge of the initial result); or $\geq1000 \text{ and} <1500 \text{ cells/}\mu\text{L}$ (from 3 test results) and an infection that is not fully resolved | Monitor and Stats | Monitor's list, or, If a patient still receives study treatment after 10 days with confirmed segmented neutrophil counts <500 cells/ $\mu$ L; $\geq$ 500 and <1000 cells/ $\mu$ L (from a test and a re-test result; the re-test must be performed within 1 week from knowledge of the initial result); or $\geq$ 1000 and <1500 cells/ $\mu$ L (from a test and 2 re-test results) and an infection that is not fully resolved If there are missing re-test results, use the non-missing results | Yes |
| [D2] Total WBC count <2000 cells/μL | Monitor and Stats | Monitor's list, or, If a patient still receives study treatment after 10 days with confirmed total WBC count <2000 cells/ $\mu$ L (defined as a test and a retest within 10 days); If no retest, use the test results | Yes |
| [D3] Lymphocyte count <500 cells/μL | Monitor and Stats | Monitor's list, or, If a patient still receives study treatment after 10 days with confirmed lymphocyte count $<$ 500 cells/ $\mu$ L (defined as a test and a retest within 10 days ) | Yes |

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | |
|---|---|---|---|
| | | If no retest, use the test results | |
| [D4] Platelet count <50,000 cells/μL | Monitor and Stats | Monitor's list, or, If a patient still receives study treatment after 10 days with confirmed platelet count <50,000 cells/μL (defined as a test and a re-test within 10 days ) If no retest, use the test results | Yes |
| [D5] Patient has a clinically significant systemic<br>hypersensitivity reaction after subcutaneous (SC)<br>administration of investigational product | Monitor | Monitor's list | Yes |
| [D6] Patient becomes pregnant | Monitor | Monitor's list | Yes |
| [D7] The patient develops a malignancy. (No more than 2 nonmelanoma skin cancers over any 12-month period during the study.) | Monitor | Monitor's list | Yes |
| [D8] The result of the TB test is positive at Week 52 (Visit 16) or later AND the patient is diagnosed with active infection | Monitor | Monitor's list | Yes |
| [D9] Patient develops symptoms suggestive of a lupus-like syndrome or is positive for antibodies against double-stranded DNA | Monitor | Monitor's list | Yes |
| [D10] If the patient for any reason requires treatment with another therapeutic agent that has been demonstrated to be effective for the treatment of PsA or psoriasis before the post-treatment follow-up period. | Monitor | Monitor's list | Yes |
| [D11] Enrollment in any other clinical trial involving an investigational product or enrollment in any other type of medical research judged not to be scientifically or medically compatible with this study | Monitor | Monitor's list | Yes |
| [D12] The patient scores a 3 for Item 12 (Thoughts of Death or Suicide) on the QIDS-SR16 at any time in the study. | Monitor and Stats | Monitor's list, or, If patient still receives study treatment on the same day or after the date with a score of 3 for Item 12 on the QIDS-SR16 | Yes |

| Important Protocol Deviation<br>Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| [D13] Failure to demonstrate at least a 20% improvement from baseline in both TJC and SJC at Week 24 or at any subsequent visit through Week 104 except from the point of randomization until the visit after relapse for those patients who are randomized in Period 3 | Monitor and Stats | Monitor's list, or, If a patients has <20% improvement from baseline in both TJC and SJC at either Week 24 or any other subsequent visit through Week 104, with the exception of randomization through the following visit after relapse for those patients who are randomized. | Yes |
| [D14] Lilly or its designee stops the patient's participation in the study or Lilly stops the study for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and GCP | Monitor | Monitor's list | Yes |
| [D15] The patient becomes HBV DNA positive. | Monitor | Monitor's list | Yes |
| Missing Data/Assessments not Done | | | |
| MDA missing due to missing values of MDA components at baseline or any visit. | Stats | If missing any individual component of MDA at baseline or any visit from Weeks 24 through 104. | No |
| Missing ECG: missing baseline | Monitor | Monitor listing | No |
| Missing C-SSRS while on study medication | Monitor | If missing C-SSRS at any Visit From Week 2 through Week 104 after Amendment A implemented at site | No |
| Patient was inadvertently randomized. Due to a discrepancy in recorded ePRO data versus the IWRS data for meeting Coates Criteria for MDA. | Monitor | Monitor listing | Yes |
| Patient started on ixekizumab 80 mg Q2W after randomization to placebo and prior to experiencing a relapse (no longer meeting Coates criteria for MDA in Period 3). | Monitor and Stats | Monitor listing, or, programming for exposure to ixekizumab 80 mg Q2W after randomization and exposure to placebo in period 3 and prior to relapse. | Yes |
| Patient took incorrect medication | Monitor and Stats | Monitor's list, or, If patient randomized and exposure data shows the patient took incorrect study medication | No |
| Patient did not take any study medication | Monitor and Stats | Monitor's list, or, If patient randomized and exposure data shows the patient took no study medication | Yes |
| Patient non-compliant with study medication | Monitor and Stats | Monitor's list, or, | Yes |

| Important Protocol Deviation Category/Subcategory | Source to Identify Protocol<br>Deviation | Statistical Programming Guidance for Clinical Study<br>Report | Exclude from the PPS? |
|---|---|---|---|
| <b>regimen.</b> Patient missing 2 consecutive doses or take 2 doses of study medication on the same day (i.e. double-dosing) are considered to be non-compliant. | | Study drug exposure is reported as missing more than 20% of expected doses for a study period or is missing 2 consecutive doses. | |
| Patient took prohibited concomitant medication | Monitor and Stats | Monitor's list, or, If patient takes prohibited concomitant medication. (Note: Prohibited concomitant medication will be provided by medical in a separate file.) | Yes |
| Unblinding is considered unjustified if the unblinding occurred on a patient where the patient's wellbeing was not dependent upon knowing their treatment assignment. | Monitor | Monitor's list | Yes |

Abbreviations: ATC = anatomical therapeutic chemical; BCG = Bacille de Calmette et Guérin; bDMARD = biologic disease-modifying antirheumatic drug; bHCG = beta human chorionic gonadotropin; ; CASPAR = classification for psoriatic arthritis; cDMARD = conventional disease-modifying antirheumatic drug; DBP = diastolic blood pressure; ePRO = electronic patient reported outcomes; GCP = good clinical practice; IV = intravenous; IWRS = interactive webresponse system; MDA = minimal disease activity; MI = myocardial infarction; MTX = methotrexate; NSAID = nonsteroidal anti-inflammatory drug; NYHA = New York Heart Association; PPS = per protocol set; PsA = psoriatic arthritis; QIDS-SR16 = quick inventory of depressive symptomatology–self-report 16 items; SBP = systolic blood pressure; SJC = swollen joint count; TB = tuberculosis; TJC = tender joint count; WHO = World Health Organization.

The term "Monitor" indicates the protocol deviation will be identified by site monitors and entered into monitor's list using a spreadsheet. The spreadsheet will be exported as Study Data Tabulation Model (SDTM) DV domain.

The term "Stats" indicates the protocol deviation will be programmed based on data in clinical database by statistical programmers with the statistical programming guidance provided as the last column. The detailed programming specification will be documented in Analysis Data Model (ADaM) specification.

The terms "Monitor and Stats" indicates the protocol deviation will be a combination of monitor's list (SDTM.DV domain) and statistical programming from clinical database, the deviation will show if either source identifies.

# 6.18. Interim Analyses and Data Monitoring

The study will have approximately 2 interim and 1 final database locks. The first interim database lock may occur once all patients complete or discontinue in the open-label treatment period the visit of randomization or Week 64 for patients who do not meet the randomization criteria); only data from the open-label treatment period will be summarized. The second interim database lock may occur when all patients complete Week 104 or discontinue study treatment prior to the end of the randomized double-blind withdrawal period. The final database lock will occur when all patients complete or discontinue the study. The second interim lock and final database lock may be combined depending upon the timing of last patient visit. Additional analyses and snapshots of study data may be performed to fulfill the need for regulatory interaction or publication purposes

Information that may unblind the study during the analyses will not be reported to study sites or the blinded study team until the study has been unblinded. All investigators and patients will remain blinded to treatment assignments until the last patient completes the randomized double-blind withdrawal period and the final database lock occurs.

# 6.19. Planned Exploratory Analyses

# 6.19.1. Planned Exploratory Efficacy Analysis

Table RHBF.6.9 includes the description and derivation of the exploratory outcomes.

Table RHBF.6.10 provides the detailed analyses including analysis type, method and imputation, population, time point, and comparisons for exploratory analyses.

 Table RHBF.6.9.
 Description and Derivation of Additional Exploratory Outcomes

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| Physician's | Physician Global VAS: overall | Change from baseline in | Range: 0 to 100 mm | single measure, missing if |
| Global | assessment of the severity of the patient's | Physician Global VAS | 0 represents no disease activity | missing |
| Assessment of Disease | current PsA activity using a 100-mm horizontal VAS. The investigator making | Percent improvement in | 100 represents extremely active disease activity | missing if baseline or observed value are missing |
| Activity Visual | the assessment must be a rheumatologist | Physician Global VAS | disease activity | observed value are missing |
| Analog Scale (VAS) | or medically qualified physician. | | | |
| Leeds<br>Enthesitis | LEI: For patients with enthesitis, an assessment that consists of 18 entheseal | Change from baseline in LEI | Each site is assigned a score of 0 (absent) or 1 (present); the | if one or more sites are missing, then set to |
| Index (LEI) | points is performed by site personnel. | Percent Improvement in LEI | results from each site are then | missing |
| | The LEI has been developed specifically for use in PsA and measures enthesitis at | | added to produce a total score (range: 0 to 6). | missing if baseline or observed value are missing |
| | 6 sites (lateral epicondyle [left and right],<br>medial femoral condyle [left and right],<br>and Achilles tendon insertion [left and<br>right]) (Healy and Helliwell 2008). | Proportion of patients with resolution in enthesitis (LEI score = 0) | For patients with baseline enthesitis (LEI ≥1), number of patients LEI score of 0 | if one or more sites are<br>missing, then set to<br>missing |
| | right]) (Fleary and Flemwen 2000). | | | missing if baseline or observed value are missing |
| Leeds | LDI-B: measure of severity of dactylitis | Change from baseline in LDI-B | Once the presence of dactylitis | |
| Dactylitis | for patients with dactylitis. Each dactylic | | is established in each digit, the | |
| Index-Basic | digit is defined by a minimum increase of | Percent improvement in LDI-B | ratio of the circumference of the | |
| (LDI-B) | 10% in circumference over the | | affected digit to the | |
| | contralateral digit. If the same digits on both hands or feet are thought to be | | on the patient's other hand or | |
| | involved, the clinician will refer to a table | | foot is measured (Helliwell et | |
| | of normative values (provided to | | al. 2005). If the circumference | |
| | investigative sites) for a value that will be | | of the affected digit ratio is 10% | |
| | used to provide the comparison. | | greater than the contra digit, the | |
| | - | | calculated ratio is minus 1 and | |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if<br>with Missing<br>Components |
|---|---|---|---|---|
| | | Proportion of patients with resolution of dactylitis (LDI-B score =0) | then multiplied 100 and then multiplied by a tenderness score of 0 (not tender) or 1 (tender). Tenderness is assessed in the area between the joints. The results of each digit are then added to produce a total score (Healy and Helliwell 2007). For patients with baseline dactylitis (LDI-B score >0), number of patients with resolution of dactylitis (LDI-B score = 0) | NA |
| Spondyloarthri<br>tis Research<br>Consortium of<br>Canada<br>(SPARCC) | SPARCC: For patients with enthesitis, an assessment that consists of 18 entheseal points is performed by site personnel. From this assessment the SPARCC index evaluates tenderness in a total of 16 enthesitis sites: the greater trochanter (right and left), quadriceps tendon insertion into the patella (right and left), patellar ligament insertion into the patella and tibial tuberosity (right and left), Achilles tendon insertion (right and left), plantar fascia insertion (right and left), medial epicondyles (right and left), and the supraspinatus insertion (right and left) (Mease 2011). | Change from baseline in SPARCC Percent improvement in SPARCC Proportion of patients with resolution of enthesitis (SPARCC >0) | Tenderness at each site is quantified on a dichotomous basis: 0 = nontender and 1 = tender. The results from each site are then added to produce a total score (range, 0 to 16). | if one or more sites are missing, then set to missing. missing if baseline or observed value are missing |
| Disease<br>Activity Score | DAS28-CRP: is a measure of disease activity in 28 joints that consists of a | Change from baseline in DAS28-CRP | The following equation will be used to calculate the DAS28- | if one or more component are missing, then set to |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| (28 diathrodial joint count) based on C-reactive protein (DAS28-CRP) | composite numerical score using the following measures: TJC, SJC, C-reactive protein (mg/L), and patient's global assessment of disease activity recorded by patients in a 100-mm VAS. The 28 joints to be examined and assessed as tender or not tender and as swollen or not swollen are a subset of those assessed for the TJC and SJC and include 14 joints on each side of the patient's body: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees (Smolen et al. 1995). | Percent improvement in DAS-CRP | CRP (Vander Cruyssen et al. 2005) See Appendix 3 for further details on calculating joint counts. Sum of the following: 1. $0.56(\sqrt{TJC28})$ 2. $0.28(\sqrt{SJC28})$ 3. $0.36(\ln[CRP + 1])$ 4. $0.014(PatientGlo\ balVAS)$ 5. $0.96$ Higher DAS28-CRP scores indicate more severe symptoms and greater functional impairment. | missing if baseline or observed value are missing |
| Psoriatic<br>Arthritis<br>Disease<br>Activity Score<br>(PASDAS) | PASDAS is a weighted index comprising assessments of joints, function, acute phase response, quality of life, and patient and physician global assessment of disease by VAS (0 mm to 10 mm). The TJC is 68 joints, the SJC is 66 joints. Worse disease activity is represented by higher scores (Helliwell et al. 2013). | PASDAS | Sum the following:<br>1. $0.18(\sqrt{PhysicianGlobalVAS})$<br>2. $0.159(\sqrt{PatientGlobalVAS})$<br>3. $-0.253(\sqrt{PCS})$<br>4. $0.101*[\ln(SJC+1)]$<br>5. $0.048*[\ln(TJC+1)]$<br>6. $0.23*[\ln(LEI+1)]$<br>7. $0.377*[\ln(TDC+1)]$<br>8. $0.102*[\ln(CRP+1)]+2$<br>Then multiply by 1.5 | if one or more components are missing, then set to missing. |
| Composite Psoriatic Disease Activity Index | CPDAI is a validated instrument to assess composite psoriatic disease activity and response to therapy (Mumtaz et al. 2011). This instrument assesses individual | Change from baseline in CPDAI Percent improvement in CPDAI | Each domain is scored from 0–3. Individual domain scores are summed to give an overall composite score (range 0–12). | if one or more domains are missing, then set to missing. |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| (CPDAI) | domains: • peripheral arthritis as assessed by the number of tender and swollen joints and the HAQ-DI, • skin as assessed by the PASI and the DLQI, • enthesitis as assessed by the number of sites with enthesitis and the HAQ-DI, and • dactylitis as assessed by the number of digits affected and the HAQ-DI. A modified version that does not include the axial domain is being used in this study. Scores range from 0 to 12; a higher score indicates higher disease activity. | | The composite scores range from 0 to 12 for assessment excluding spinal disease, with a higher score indicating higher disease activity. See Appendix 10 for further details. | missing if baseline or observed value are missing |
| Psoriasis Area<br>and Severity<br>Index (PASI) | PASI improvement from baseline | PASI 75 Flag PASI 90 Flag PASI 100 Flag | Defined as at least a 75%, 90%, or 100% improvement from baseline in PASI score See Table RHBF.6.3 for details on the calculation of PASI | Single item, missing if missing |
| Psoriatic<br>Arthritis<br>Response<br>Criteria<br>(PsARC) | PsARC is a composite criteria reported in terms of the percentage of patients achieving response according to the following criteria: 1. Physician Global Assessment of Disease Activity, 2. Patient Global Assessment of Disease Activity, 3. TJC, and | PsARC responder Flag | Response is defined by improvement from baseline assessment in 2 of the 4 criteria, 1 in which must be a joint count; and there must not be worsening of any of the 4 criteria: 1. ≥30% reduction in TJC, 2. ≥30% reduction in SJC, | If one or more criteria are missing then missing |

| Measure | Description | Variable | Derivation / Comment | Imputation Approach if<br>with Missing<br>Components |
|---|---|---|---|---|
| Static | 4. SJC<br>sPGA (0,1) | sPGA (0,1) Flag | <ul> <li>3. ≥20 mm reduction in the physician's assessment (VAS), and</li> <li>4. ≥20 mm reduction in the patient's assessment (VAS) (Clegg et al. 1996)</li> <li>Defined as plaques that are</li> </ul> | Single item, missing if |
| Physician's<br>Global<br>Assessment<br>(sPGA) (0,1)<br>and (0) | sPGA (0) | PGA (0) Flag | either clear or minimal (0,1) Defined as plaques that are clear (0) | missing Single item, missing if missing |
| Disease<br>Activity index<br>for PSoriatic<br>Arthritis<br>(DAPSA) | Composite score that includes at least one variable from each factor to cover all important domains of the multifaceted systemic disease with a main focus on the musculoskeletal system and excludes the skin domain (Smolen et al. 2015). | Change from baseline in DAPSA score Percent improvement in DAPSA score | Sum of the following: 1. SJC 2. TJC 3. patient pain VAS score 4. patient global VAS score 5. CRP (mg/L) | If any item is missing, then missing |
| | | DAPSA Low Disease Activity (LDA) DAPSA Remission | 4 < DAPSA ≤14 DAPSA ≤4 | If DAPSA is missing, missing If DAPSA is missing, missing |
| | | DAPSA ≤14 | DAPSA ≤14 | If DAPSA is missing, missing |

Abbreviations: NA = not applicable; PsA = psoriatic arthritis; SJC = swollen joint count; TJC = tender joint count.

 Table RHBF.6.10.
 Description of Planned Exploratory Efficacy Analyses

| Measure | Variable | Analysis Method<br>(Section 6.1) | Population<br>(Section 6.6.1) | Comparison/Time Point |
|---|---|---|---|---|
| Coates criteria for<br>minimal disease<br>activity (MDA) | Time-to achieve<br>sustained Coates Criteria<br>for MDA (MDA for 12<br>consecutive months) | Descriptive Statistics for ixekizumab 80 mg Q2W (including Kaplan Meier estimates of the survival curve) | Ixekizumab-treated patients: nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and 3 combined |
| Disease Activity<br>Score (28 | Time-to achieve DAS28-CRP low disease activity | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| arthrodial joint<br>count) based on<br>CRP (DAS28- | (score ≤2.8)<br>(Helliwell et al. 2014) | (including Kaplan Meier estimates of the survival curve) | Ixekizumab-treated patients: nonrandomized population and randomized withdrawal ITT population | Assessed during Periods 2 and 3 combined |
| CRP) | Change from baseline in DAS28-CRP | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | Percent improvement in DAS28-CRP | | Ixekizumab-treated patients:<br>nonrandomized population and<br>randomized withdrawal ITT population | Assessed during Periods 2 and 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3, patients with 40 Weeks of Randomized Treatment |
| Psoriatic Arthritis Disease Activity | Time-to achieve<br>PASDAS low disease | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| Score (PASDAS) | activity (score ≤3.2)<br>(Helliwell et al. 2014) | (including Kaplan Meier estimates of the survival curve) | Ixekizumab-treated patients: nonrandomized population and randomized withdrawal ITT population | Assessed during Periods 2 and 3 combined |
| | Change from baseline in PASDAS | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |

| | | Analysis Method | Population | |
|---|---|---|---|---|
| Measure | Variable | (Section 6.1) | (Section 6.6.1) | Comparison/Time Point |
| | Percent improvement in PASDAS | | Ixekizumab-treated patients:<br>nonrandomized population and<br>randomized withdrawal ITT population | Assessed during Periods 2 and 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 Weeks of Randomized<br>Treatment |
| Composite Psoriatic Disease Active Index | Time-to achieve<br>modified CPDAI low<br>disease activity (score | Descriptive Statistics for ixekizumab 80 mg Q2W (including Kaplan Meier | Initial open-label treatment period population | Assessed during Period 2 |
| (CPDAI) | ≤3) e | estimates of the survival curve) | Ixekizumab-treated patients:<br>nonrandomized population and<br>randomized withdrawal ITT population | Assessed during Periods 2 and 3 combined |
| | Change from baseline in CPDAI domain scores | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | Change from baseline in CPDAI composite scores | | Ixekizumab-treated patients:<br>nonrandomized population and<br>randomized withdrawal ITT population | Assessed during Periods 2 and 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 Weeks of Randomized<br>Treatment |
| Psoriatic Arthritis<br>Response Criteria | PsARC responder | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| (PsARC) | | | Ixekizumab-treated patients: nonrandomized population and randomized withdrawal ITT population | Assessed during Periods 2 and 3 combined |
| | | Logistic regression analysis with NRI; | Randomized withdrawal ITT population | Assess during Period 3 through 40 Weeks of Randomized |
| | | Fisher's exact test with NRI | | Treatment |
| | | Analysis Method | Population | |
|---|---|---|---|---|
| Measure | Variable | (Section 6.1) | (Section 6.6.1) | Comparison/Time Point |
| Psoriasis Area and<br>Severity Index<br>(PASI) 75, 90, and | Proportion of patients with PASI 75 | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment population with baseline psoriatic lesions involving BSA ≥3% | Assessed during Period 2 |
| 100 | Proportion of patients<br>with PASI 90<br>Proportion of patients<br>with PASI 100 | | Ixekizumab-treated patients with baseline psoriatic lesions involving BSA ≥3%: nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | Logistic regression analysis with NRI; Fisher's exact test with NRI | Randomized withdrawal ITT population with baseline psoriatic lesions involving BSA ≥3% | Assess during Period 3 through<br>40 Weeks of Randomized<br>Treatment |
| | Change from baseline in PASI Total Score | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment population with baseline psoriatic lesions involving BSA ≥3% | Assessed during Period 2 |
| | Percent Improvement in Total Score | | Ixekizumab-treated patients with baseline psoriatic lesions involving BSA ≥3%: nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population with baseline psoriatic lesions involving BSA ≥3% | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| Static Physician's<br>Global Assessment | Proportion of patients with sPGA (0,1) | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment population with sPGA ≥3 at baseline | Assessed during Period 2 |
| sPGA of Psoriasis (0,1) and (0) | Proportion of patients with sPGA(0) | | Ixekizumab-treated patients with sPGA ≥3 at baseline: nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |

| Measure | Variable | Analysis Method<br>(Section 6.1) | Population<br>(Section 6.6.1) | Comparison/Time Point |
|---|---|---|---|---|
| | | Logistic regression analysis with NRI;<br>Fisher's exact test with NRI | Randomized withdrawal ITT population with sPGA $\geq$ 3 at baseline | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| Body surface area (BSA) | Change from baseline in percent involvement of BSA | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment population with baseline Psoriatic Lesions Involving ≥3% BSA | Assessed during Period 2 |
| | | | Ixekizumab-treated patients with baseline Psoriatic Lesions Involving ≥3% BSA: nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population with baseline Psoriatic Lesions Involving ≥3% BSA | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| Patient's Assessment of | Change in baseline in<br>Patient Pain VAS | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| Pain Visual<br>Analog Scale<br>(VAS) | Percent improvement in Patient Pain VAS | | Ixekizumab-treated patients:<br>nonrandomized population and<br>randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| Patient's Global<br>Assessment of | Change in baseline in patient global VAS | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| Disease Activity<br>VAS | Percent improvement in patient global VAS | | Ixekizumab-treated patients:<br>nonrandomized population and<br>randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |

| Measure | Variable | Analysis Method<br>(Section 6.1) | Population (Section 6.6.1) | Comparison/Time Point |
|---|---|---|---|---|
| Physician's Global<br>Assessment of | Change in baseline in physician global VAS | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| Disease Activity<br>VAS | Percent improvement in physician global VAS | | Ixekizumab-treated patients:<br>nonrandomized population and<br>randomized withdrawal ITT population | Assessed during Period 2 and<br>Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| Spondyloarthritis<br>Research<br>Consortium of | Change from baseline in SPARCC | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population with baseline enthesitis (SPARCC >0) | Assessed during Period 2 |
| Canada (SPARCC) Percent improvement in SPARCC | - | | Ixekizumab-treated patients with baseline enthesitis (SPARCC >0): nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population with Baseline Enthesitis (SPARCC >0) | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |

| Measure | Variable | Analysis Method<br>(Section 6.1) | Population (Section 6.6.1) | Comparison/Time Point |
|---|---|---|---|---|
| | Proportion of patients<br>with resolution in<br>enthesitis (SPARCC =0) | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population with Baseline Enthesitis (SPARCC >0) | Assessed during Period 2 |
| | | Logistic regression analysis with NRI;<br>Fisher's exact test with NRI | Randomized withdrawal ITT population with Baseline Enthesitis (SPARCC >0) | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| Leeds Dactylitis<br>Index - Basic<br>(LDI-B) | Change from baseline in LDI-B | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population with baseline dactylitis (LDI-B Score >0) | Assessed during Period 2 |
| | Percent improvement in LDI-B | | Ixekizumab-treated patients with baseline dactylitis (LDI-B Score >0): nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population with baseline dactylitis (LDI-B Score >0) | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| | Proportion of patients with improvement in dactylitis ( ≥1 digit | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population with baseline dactylitis (LDI-B Score >0) | Assessed during Period 2 |
| | Proportion of patients with resolution of | | Ixekizumab-treated patients with baseline dactylitis (LDI-B Score >0): nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | dactylitis (LDI-B = 0) | Logistic regression analysis with NRI;<br>Fisher's exact test with NRI | Randomized withdrawal ITT population with baseline dactylitis (LDI-B Score >0) | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| Leeds Enthesitis<br>Index (LEI) | Change from baseline in LEI | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population with baseline enthesitis (LEI Score >0) | Assessed during Period 2 |

| | | Analysis Method | Population | |
|---|---|---|---|---|
| Measure | Variable | (Section 6.1) | (Section 6.6.1) | Comparison/Time Point |
| | Percent improvement in LEI | | Ixekizumab-treated patients with baseline enthesitis (LEI Score >0): nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population with baseline enthesitis (LEI Score >0) | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| | Proportion of patients with resolution in enthesitis (LEI =0) | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population with baseline enthesitis (LEI Score >0) | Assessed during Period 2 |
| | | | Ixekizumab-treated patients with baseline enthesitis (LEI Score >0: nonrandomized population and randomized withdrawal ITT population) | Assessed during Period 2 and Period 3 combined |
| | | Logistic regression analysis with NRI;<br>Fisher's exact test with NRI | Randomized withdrawal ITT population with baseline enthesitis (LEI Score >0) | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| Enthesitis, 18 entheseal points (as measured by a | Change from baseline in Enthesitis, 18 entheseal points | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population with baseline enthesitis (18 entheseal point score >0) | Assessed during Period 2 |
| combination of the<br>LEI and the<br>SPARCC) | Percent improvement in Enthesitis, 18 entheseal points | | Ixekizumab-treated patients with baseline enthesitis (18 entheseal point score >0): nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population with baseline enthesitis (18 entheseal points score >0) | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| | Proportion of patients with resolution in enthesitis (18 entheseal | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population with baseline enthesitis (18 entheseal points score >0) | Assessed during Period 2 |

| | | Analysis Method | Population | |
|---|---|---|---|---|
| Measure | Variable | (Section 6.1) | (Section 6.6.1) | Comparison/Time Point |
| | points score =0) | | Ixekizumab-treated patients with baseline enthesitis (18 entheseal points score >0: nonrandomized population and randomized withdrawal ITT population) | Assessed during Period 2 and Period 3 combined |
| | | Logistic regression analysis with NRI; Fisher's exact test with NRI | Randomized withdrawal ITT population with baseline enthesitis (18 entheseal points score >0) | Assess during Period 3 through<br>40 Weeks of Randomized<br>Treatment |
| Swollen joint count (SJC) | Change from baseline in SJC | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | Percent improvement in SJC | | Ixekizumab-treated patients:<br>nonrandomized population and<br>randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| Tender joint count (TJC) | Change from baseline in TJC | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | Percent improvement in TJC | | Ixekizumab-treated patients:<br>nonrandomized population and<br>randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| Disease Activity index for PSoriatic | Change from baseline in DAPSA score | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| Arthritis (DAPSA) | Percent improvement in DAPSA score | | Ixekizumab-treated patients:<br>nonrandomized population and<br>randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |

| | | Analysis Method | Population | |
|---|---|---|---|---|
| Measure | Variable | (Section 6.1) | (Section 6.6.1) | Comparison/Time Point |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 weeks of Randomized<br>Treatment |
| | Proportion of patients<br>with DAPSA LDA<br>(DAPSA >4 and DAPSA | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | (DAPSA ≥4 and DAPSA ≤14) | | Ixekizumab-treated patients (nonrandomized population and randomized withdrawal ITT population) | Assessed during Period 2 and Period 3 combined |
| | | Logistic regression analysis with NRI;<br>Fisher's exact test with NRI | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 Weeks of Randomized<br>Treatment |
| | Proportion of patients with DAPSA remission | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | (DAPSA ≤4) | | Ixekizumab-treated patients (nonrandomized population and randomized withdrawal ITT population) | Assessed during Period 2 and Period 3 combined |
| | | Logistic regression analysis with NRI; Fisher's exact test with NRI | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 Weeks of Randomized<br>Treatment |
| | Proportion of patients with DAPSA ≤14 | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | | | Ixekizumab-treated patients (nonrandomized population and randomized withdrawal ITT population) | Assessed during Period 2 and Period 3 combined |
| | | Logistic regression analysis with NRI; Fisher's exact test with NRI | Randomized withdrawal ITT population | Assess during Period 3 through<br>40 Weeks of Randomized<br>Treatment |

Abbreviations: ANCOVA = analysis of covariance; ITT = intent-to-treat; mBOCF = modified baseline observation carried forward; MMRM = mixed-effects model of repeated measures; NRI = nonresponder imputation; Q2W = every 2 weeks.

### 6.19.2. Planned Exploratory Health Outcomes/Quality-of-Life Analyses

The health outcomes and quality of life (QOL) measures are Itch NRS, Fatigue Severity NRS, DLQI, SF-36 Mental and Physical Component Summary Scores, EQ-5D-5L, Work Productivity and Activity Impairment Questionnaire-Specific Health Problem, and the QIDS-SR16. There will be no adjustment for multiple comparisons.

Table RHBF.6.11 includes the description and derivation of the health outcomes and QOL measures.

Table RHBF.6.12 provides the detailed analyses including analysis type, method and imputation, population, time point, and comparisons for health outcomes and QOL analyses.

 Table RHBF.6.11.
 Description and Derivation of Health Outcomes and Quality-of-Life Measures

| Measure | Description | Variable | Derivation / Comment | Missing Items |
|---|---|---|---|---|
| Itch Numeric | Itch NRS: is a single-item, patient- | Itch NRS score | Range from 0 to 10. | Single item, missing if |
| Rating Scale | reported outcome (PRO) measure | | | missing |
| (NRS) | designed to capture information on the | Itch NRS change from baseline | Calculated as: | 1.Missing if baseline or |
| | overall severity of a patient's itching | | 1. observed Itch NRS – baseline Itch | observed value is |
| | due to their psoriatic skin condition by | | NRS | missing |
| | having the patient selecting the integer | | 2. mBOCF Itch NRS | 2.Missing if baseline is |
| | that best describes the worst level of | | | missing |
| | itching in the past 24 hours on an 11- | Itch NRS ≥3 improvement | Reduced/decreased of ≥3 point from | Missing if baseline or |
| | point NRS anchored at 0 representing | from baseline | baseline | observed value is missing |
| | "no itching" and 10 representing | Itch NRS =0 | Defined as a post-baseline Itch NRS | Missing if Itch NRS score |
| | "worst itch imaginable." | | score of 0 | is missing |
| Fatigue | Fatigue Severity NRS: is a patient- | Fatigue Severity NRS | Range from 0 to 10. | Single item, missing if |
| Severity | administered single-item 11-point | | | missing |
| Numeric | horizontal scale anchored at 0 and 10, | Fatigue Severity NRS change | Calculated as: | 1.Missing if baseline or |
| Rating Scale | on which 0 represents "no fatigue" and | from baseline | 1. observed Fatigue Severity NRS – | observed value is |
| | 10 represents "as bad as you can | | baseline Fatigue Severity NRS | missing |
| | imagine." Patients rate their fatigue | | 2. mBOCF Fatigue Severity | 2.Missing if baseline is |
| | (feeling tired or worn out) by selecting | | | missing |
| | the single number that describes their | Fatigue Severity $NRS = 0$ | Defined as a post-baseline Fatigue | Missing if Fatigue |
| | worst level of fatigue during the past | | Severity NRS score of 0 | Severity NRS score is |
| | 24 hours. | | | missing |
| | | Improvement in 2 points and 3 | Defined as a change from baseline in | Missing if Fatigue |
| | | points in Fatigue Severity NRS | Fatigue Severity NRS score of ≥2; | Severity NRS score is |
| | | | and | missing |
| | | | Defined as a change from baseline in | |
| | | | Fatigue Severity NRS score of ≥3 | |

| Measure | Description | Variable | Derivation / Comment | Missing Items |
|---|---|---|---|---|
| Dermatology | DLQI: is a validated, dermatology- | DLQI symptoms and feelings | Sum of responses of questions #1 | If one question in a |
| Life Quality | specific, patient-reported measure that | domain | and #2: | domain is missing, that |
| Index (DLQI) | evaluates patient's health-related | | #1. How itchy, sore, painful or | domain is missing. |
| | quality of life. This questionnaire has | | stinging has your skin been? | |
| | 10 items that are grouped in 6 domains, | | #2. How embarrassed or self- | |
| | including symptoms and feelings, daily | | conscious have you been because of | |
| | activities, leisure, work and school, | | your skin? | |
| | personal relationships, and treatment. | DLQI daily activities domain | Sum of responses of questions #3 | If one question in a |
| | The recall period of this scale is over | | and #4: | domain is missing, that |
| | the "last week". Response categories | | #3. How much has your skin | domain is missing. |
| | and corresponding scores are: | | interfered with you going shopping | |
| | Very much = 3 | | or looking after your home or | |
| | A lot = 2 | | garden? | |
| | A little = 1 | | #4. How much has your skin | |
| | Not at all $= 0$ | | influenced the clothes you wear? | |
| | Not relevant $= 0$ | DLQI leisure domain | Sum of responses of questions #5 | If one question in a |
| | | | and #6: | domain is missing, that |
| | | | #5. How much has your skin | domain is missing. |
| | | | affected any social or leisure | |
| | | | activities? | |
| | | | #6. How much has your skin make it | |
| | | | difficult for you to do any sport? | |
| | | DLQI work and school domain | Sum of responses of questions | If the answer to question |
| | | | question #7A and #7B: | #7A is missing, this |
| | | | #7A. Has your skin prevented you | domain is missing. If |
| | | | from working or studying? | #7A is No, and #7B is |
| | | | #7B. If No: how much has your skin | missing, this domain is |
| | | | been a problem at work or studying? | missing. |

| Measure | Description | Variable | Derivation / Comment | Missing Items |
|---|---|---|---|---|
| | | DLQI personal relationships domain | Sum of responses of questions #8 and #9: #8. How much has your skin created problems with your partner or any of your close friends or relatives? #9. How much has your skin caused any sexual difficulties? | If one question in a domain is missing, that domain is missing. |
| | | DLQI treatment | Response of question #10:<br>#10. How much of a problem has<br>the treatment for your skin been, for<br>example by making your home<br>messy, or by taking up time? | If one question in a domain is missing, that domain is missing. |
| | | DLQI total score | A DLQI total score is calculated by summing all 10 question responses, and has a range of 0 to 30 (less to more impairment) (Finlay and Khan 1994; Basra et al. 2008). | If two or more questions are missing, the total score is missing. (Note: #7B could be a valid missing while #7A is not "No." That is, #7 should be considered as one question.) |
| | | DLQI (0,1) | A DLQI (0,1) response is defined as a post-baseline DLQI total score of 0 or 1. A DLQI total score of 0 to 1 is considered as having no effect on a patient's HRQoL (Khilji et al. 2002; Hongbo et al. 2005). | Missing if DLQI total score is missing |
| | | DLQI total score ≥5 improvement from baseline | Reduction/decrease of ≥5 points from baseline. A 5-point change from baseline is considered as the minimal clinically important difference threshold. | Missing if baseline or observed value is missing |
| | | DLQI total score and domain scores change from baseline | Calculated as: observed DLQI (total score or domain scores) – baseline DLQI (total score or domain scores) | Missing if baseline or observed value is missing |

| Measure | Description | Variable | Derivation / Comment | Missing Items |
|---|---|---|---|---|
| Medical | SF-36: is a 36-item patient- | 8 associated domain scores: | Per copyright owner, the | Missing data handling |
| Outcomes | administered measure designed to be a | <ul> <li>Physical Functioning,</li> </ul> | QualityMetric Health Outcomes <sup>TM</sup> | offered by SF-36 software |
| Study 36-item | short, multipurpose assessment of | Role Physical, | Scoring Software 4.5 will be used to | will not be used. |
| Short-Form | health in the areas of physical | Bodily Pain, | derive SF-36 domain and component | |
| Health | functioning, role-physical, role- | General Health, | scores. After data quality-controls, | |
| Survey (SF- | emotional, bodily pain, vitality, social | • Vitality, | the SF-36 software will re-calibrate | |
| 36) | functioning, mental health, and general | <ul> <li>Social Functioning,</li> </ul> | the item-level responses for | |
| | health. The 2 overarching domains of | Role Emotional, and Mental | calculation of the domain and | |
| | mental well-being and physical well- | Health | component scores. These raw scores | |
| | being are captured by the Mental | 2 component Scores: | will be transformed into the domain | |
| | Component Summary (MCS) and | MCS Score | scores (t-scores) using the 1-week | |
| | Physical Component Summary (PCS) | PCS Score | recall period. The procedure to | |
| | scores. The summary scores range | | derive the SF-36 scores is described | |
| | from 0 to 100; higher scores indicate | | in Appendix 6. It entails exporting | |
| | better levels of function and/or better | | the patient data in a CSV or tab- | |
| | health. Items are answered on Likert | | delimited file for import, generation | |
| | scales of varying lengths. The SF-36 | | of the SF-36 scores and reports, and | |
| | version 2 (acute version) health survey | | export of the calculated scores in a | |
| | will be used, which has a 1-week recall | | CSV or tab-delimited file for | |
| | period (Brazier et al. 1992; Ware and | | integration into SDTM/ADaM | |
| | Sherbourne 1992). | | datasets. The summary scores range | |
| | | | from 0 to 100. | |
| Work | Work Productivity and Activity | percentage of absenteeism | Percent work time missed due to | if Q2 or Q4 is missing, |
| Productivity | Impairment-Specific Health Problem: | | problem: $(Q2/(Q2 + Q4))*100$ | then missing |
| and Activity | consists of 6 questions to determine | | | |
| Impairment- | employment status, hours missed from | percentage of presenteeism | Percent impairment while working | if Q5 is missing, then |
| Specific | work because of PsA, hours missed | (reduced productivity while at | due to problem: (Q5/10)*100 | missing |
| Health | from work for other reasons, hours | work) | | _ |
| Problem | actually worked, the degree to which | overall work impairment score | Percent overall work impairment due | if Q2, Q4, or Q5 is |
| | PsA affected work productivity while | that combines absenteeism and | to problem: (Q2/(Q2+ Q4) + [(1- | missing, then missing |
| | at work, and the degree to which PsA | presenteeism | Q2/(Q2+Q4))*(Q5/10)])*100 | |
| | affected activities outside of work. | | | |

| Measure | Description | Variable | Derivation / Comment | Missing Items |
|---|---|---|---|---|
| | Four scores are derived: percentage of | percentage of impairment in | Percent activity impairment due to | if Q6 is missing, then |
| | absenteeism, percentage of | activities performed outside of | problem: (Q6/10)*100 | missing |
| | presenteeism (reduced productivity | work | | |
| | while at work), an overall work | | | |
| | impairment score that combines | | | |
| | absenteeism and presenteeism, and | | | |
| | percentage of impairment in activities | | | |
| | performed outside of work. Greater | | | |
| | scores indicate greater impairment | | | |
| | (Reilly et al. 1993; Reilly Associates | | | |
| | Health Outcomes Research [WWW]). | | | |
| European | EQ-5D-5L is a standardized measure of | EQ-5D mobility, | Five health profile dimensions, each | Each dimension is a |
| Quality of | health status used to provide a simple, | EQ-5D self-care, | dimension has 5 levels: | single item, missing if |
| Life – 5 | generic measure of health for clinical | EQ-5D usual activities, EQ-5D | 1 = no problems | missing. (Note: Score of |
| Dimensions 5 | and economic appraisal. The EQ-5D- | pain/ discomfort, | 2 = slight problems | 9 is missing.) |
| Level (EQ- | 5L consists of 2 components: a | EQ-5D anxiety/ depression | 3 = moderate problems | |
| 5D-5L) | descriptive system of the respondent's | | 4 = severe problems | |
| | health and a rating of his/her current | | 5 = extreme problems | |
| | health state using a 0- to 100-mm VAS. | | It should be noted that the numerals | |
| | The descriptive system comprises the | | 1 to 5 have no arithmetic properties | |
| | following 5 dimensions: | | and should not be used as a primary | |
| | item 1: mobility | | score. | |
| | item 2: self-care | EQ-5D-5L UK Population- | Uses the concatenation of the value | If any of the items is |
| | item 3: usual activities | based index score | of each EQ-5D-5L dimension score | missing or equal to 9, the |
| | item 4: pain/discomfort | | in the order: item1; item2; item3; | index score is missing |
| | item 5: anxiety/depression | | item4; item5. Derive EQ-5D-5L UK | |
| | The respondent is asked to indicate | | Population-based index score | |
| | his/her health state by ticking (or | | according to the link by using the | |
| | placing a cross) in the box associated | | UK algorithm (Szende et al. 2007) to | |
| | with the most appropriate statement in | | produce a patient-level index score | |
| | each of the 5 dimensions. | | between -0.59 and 1.0 (continuous | |
| | | | variable): | |
| | | | http://www.euroqol.org/fileadmin/us | |
| | | | er_upload/Documenten/Excel/Cross | |

| Measure | Description | Variable | Derivation / Comment | Missing Items |
|---|---|---|---|---|
| | | | walk_5L/EQ-5D-<br>5L Crosswalk Value Sets.xls | |
| | The EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, may be converted into a single summary index by applying a formula that essentially attaches values (also called weights) to each of the levels in each dimension (EuroQol Group 2013 [WWW]). The VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labeled 100 = "best imaginable health state" and 0 = "worst imaginable health state." This information can be used as a quantitative measure of health outcome. | EQ-5D VAS | Range from 0 = "worst imaginable health state" to 100 = "best imaginable health state". (Note: Higher value indicates better health state.) | Single item, missing if missing |
| Quick<br>Inventory of<br>Depressive<br>Symptoma-<br>tology-Self<br>Report (16 | QIDS-SR16 is a self-administered 16-<br>item instrument intended to assess the<br>existence and severity of symptoms of<br>depression as listed in the American<br>Psychiatric Association's Diagnostic<br>and Statistical Manual of Mental | Sleep disturbance (initial, middle, and late insomnia or hypersomnia) Change from baseline in sleep disturbance | the highest score recorded for the 4 sleep items: #1 (falling asleep), #2 (sleep during the night), #3 (waking up too early) and #4 (sleeping too much). | Domain is missing if all items are missing. |

| Measure | Description | Variable | Derivation / Comment | Missing Items |
|---|---|---|---|---|
| | | Sad mood | Score recorded for item #5 | Domain is missing if the item is missing. |
| | | Change from baseline in sad mood | | _ |
| | | Decrease/increase in appetite/weight | the highest score recorded for the appetite/weight items (items #6 to #9) | Domain is missing if all items are missing or not applicable. |
| | | Change from baseline in decrease/increase in appetite/weight | | |
| | | Concentration Change from baseline in concentration | Score recorded for item #10 (concentration/ decision making) | Domain is missing if the item is missing. |
| | | Self-criticism Change from baseline in self-criticism | Score recorded for item #11 (view of myself) | Domain is missing if the item is missing. |
| | | Suicidal ideation Change from baseline in | Score recorded for item #12 (thoughts of death or suicide) | Domain is missing if the item is missing |
| | | Suicidal ideation Interest Change from baseline in interest | Score recorded for item #13 (general interest) | Domain is missing if the item is missing. |
| | | Energy/fatigue Change from baseline in energy/fatigue | Score recorded for item #14 (energy level) | Domain is missing if the item is missing. |
| | | Psychomotor agitation/ retardation Change from baseline in | The highest score recorded for the two psychomotor items: #15 (feeling slowed down) and #16 (feeling restless). | Domain is missing if all items are missing. |

| Measure | Description | Variable | Derivation / Comment | Missing Items |
|---|---|---|---|---|
| | | psychomotor agitation/ | | |
| | | retardation | | |
| | | QIDS-SR16 total score | QIDS-SR16 total score is the sum of | The total score will be |
| | | | the domain scores. The range for | missing if any domain |
| | | Change from baseline in QIDS- | total score is 0 to 27. | score is missing. |
| | | SR16 total score | | |
| | | Proportion of patients with at | QIDS-SR16 total score at each post- | The total score will be |
| | | least a 50% decrease in QIDS- | baseline visit is at least a 50% | missing if any domain |
| | | SR16 total score | reduction of the patient's baseline | score is missing |
| | | | QIDS-SR16 total score | |

Abbreviations: ADaM = Analysis Data Model; mBOCF = modified baseline observation carried forward; PsA = psoriatic arthritis; SDTM = Study Data Tabulation Model; UK = United Kingdom.

Table RHBF.6.12. Description of Planned Exploratory Health Outcomes and Quality-of-Life Analyses

| Measure | Variable | Analysis Method (Section 6.1) | Population (Section 6.6.1) | Comparison/Time Point |
|---|---|---|---|---|
| Itch Numeric | Itch NRS ≥3 improvement | Descriptive Statistics for | Initial open-label treatment period | Assessed during Period 2 |
| Rating Scale | from baseline | ixekizumab 80 mg Q2W | population with baseline psoriatic lesions | |
| (NRS) | | | involving ≥3% BSA and baseline Itch NRS | |
| | | | score ≥3 | |
| | | | Ixekizumab-treated patients with baseline | Assessed during Period 2 and |
| | | | psoriatic lesions involving ≥3% BSA and | Period 3 combined |
| | | | baseline Itch NRS score ≥3: nonrandomized | |
| | | | and Randomized withdrawal ITT population | |
| | | Logistic regression analysis with | Randomized withdrawal ITT population | Assessed during Period 3 |
| | | NRI; Fisher's exact test with | with baseline psoriatic lesions involving | through 40 weeks of |
| | | NRI | ≥3% BSA and baseline Itch NRS score ≥3 | Randomized Treatment |
| | Itch NRS =0 | Descriptive Statistics for | Initial open-label treatment period | Assessed during Period 2 |
| | | ixekizumab 80 mg Q2W | population with baseline psoriatic lesions | |
| | | | involving ≥3% BSA and baseline Itch NRS | |
| | | | score >0 | |
| | | | Ixekizumab-treated patients with baseline | Assessed during Period 2 and |
| | | | psoriatic lesions involving ≥3% BSA and | Period 3 combined |
| | | | baseline Itch NRS score >0: nonrandomized | |
| | | | and Randomized withdrawal ITT population | |
| | | Logistic regression analysis with | Randomized withdrawal ITT population | Assessed during Period 3 |
| | | NRI; Fisher's exact test with | with baseline psoriatic lesions involving | through 40 weeks of |
| | | NRI | ≥3% BSA and baseline Itch NRS score >0 | Randomized Treatment |
| | Itch NRS change from | Descriptive Statistics for | Initial open-label treatment period | Assessed during Period 2 |
| | baseline | ixekizumab 80 mg Q2W | population with baseline psoriatic lesions involving BSA $\geq$ 3% | |
| | | | Ixekizumab-treated patients with baseline | Assessed during Period 2 and |
| | | | psoriatic lesions involving BSA≥3%: | Period 3 combined |
| | | | nonrandomized population and Randomized | |
| | | | withdrawal ITT population | |
| | | MMRM; ANCOVA with | Randomized withdrawal ITT population | Assessed during Period 3 |
| | | mBOCF | with baseline psoriatic lesions involving | through 40 weeks of |
| | | | BSA ≥3% | Randomized Treatment |

| Measure | Variable | Analysis Method (Section 6.1) | Population (Section 6.6.1) | Comparison/Time Point |
|---|---|---|---|---|
| Fatigue | Fatigue Severity NRS =0 | Descriptive Statistics for | Initial open-label treatment period | Assessed during Period 2 |
| Severity | | ixekizumab 80 mg Q2W | population | |
| NRS | | | Ixekizumab-treated patients: | Assessed during Period 2 and |
| | | | nonrandomized population and Randomized | Periods 3 combined |
| | | | withdrawal ITT population | |
| | | Logistic regression analysis with | Randomized withdrawal ITT population | Assessed during Period 3 |
| | | NRI; Fisher's exact test with | | through 40 weeks of |
| | | NRI | | Randomized Treatment |
| | Fatigue Severity NRS change | Descriptive Statistics for | Initial open-label treatment period | Assessed during Period 2 |
| | from baseline | ixekizumab 80 mg Q2W | population | |
| | | | Ixekizumab-treated patients: | Assessed during Period 2 and |
| | | | nonrandomized population and Randomized | Period 3 combined |
| | | | withdrawal ITT population | |
| | | MMRM; | Randomized withdrawal ITT population | Assessed during Period 3 |
| | | | | through 40 weeks of |
| | | ANCOVA with mBOCF | | Randomized Treatment |
| Dermatology | DLQI (0,1), | Descriptive Statistics for | Initial open-label treatment period | Assessed during Period 2 |
| Life Quality | | ixekizumab 80 mg Q2W | population with baseline psoriatic lesions | |
| Index | | | involving BSA≥3% | |
| (DLQI) | | | Ixekizumab-treated patients with baseline | Assessed during Period 2 and |
| | | | psoriatic lesions involving BSA\ge 3\%: | Period 3 combined |
| | | | nonrandomized population and | |
| | | | Randomized withdrawal ITT population | |
| | | Logistic regression analysis with | Randomized withdrawal ITT population | Assessed during Period 3 |
| | | NRI; Fisher's exact test with | with baseline psoriatic lesions involving | through 40 weeks of |
| | | NRI | BSA≥3% | Randomized Treatment |
| | DLQI total score and domain | Descriptive Statistics for | Initial open-label treatment period | Assessed during Period 2 |
| | scores change from baseline | ixekizumab 80 mg Q2W | population with baseline psoriatic lesions | |
| | | | involving BSA ≥3% | |
| | | | Ixekizumab-treated patients with baseline | Assessed during Period 2 and |
| | | | psoriatic lesions involving BSA ≥3%: | Period 3 combined |
| | | | nonrandomized population and Randomized | |
| | | | withdrawal ITT population | |

| Measure | Variable | Analysis Method (Section 6.1) | Population (Section 6.6.1) | Comparison/Time Point |
|---|---|---|---|---|
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population with baseline psoriatic lesions involving BSA ≥3% | Assessed during Period 3<br>through 40 weeks of<br>Randomized Treatment |
| 36 item<br>Short Form | 8 associated domain scores: • Physical Functioning | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| Health<br>Survey | , and the second | | Ixekizumab-treated patients:<br>nonrandomized population and Randomized<br>withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | <ul><li> Vitality</li><li> Social Functioning</li><li> Role Emotional</li><li> Mental Health</li></ul> | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assessed during Period 3<br>through 40 weeks of<br>Randomized Treatment |
| | MCS Score | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | | | Ixekizumab-treated patients:<br>nonrandomized population and Randomized<br>withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assessed during Period 3<br>through 40 weeks of<br>Randomized Treatment |
| | PCS Score | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | | | Ixekizumab-treated patients:<br>nonrandomized population and Randomized<br>withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assessed during Period 3<br>through 40 weeks of<br>Randomized Treatment |
| Work<br>Productivity | Change from baseline in the following: | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| and Activity Impairment Specific | <ul> <li>percentage of absenteeism</li> <li>percentage of presenteeism (reduced</li> </ul> | | Ixekizumab-treated patients: nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |

| Measure | Variable | Analysis Method (Section 6.1) | Population (Section 6.6.1) | Comparison/Time Point |
|---|---|---|---|---|
| Health<br>Problem | productivity while at work) • overall work impairment score that combines absenteeism and presenteeism • percentage of impairment in activities performed outside of work | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assessed during Period 3<br>through 40 weeks of<br>Randomized Treatment |
| European Quality of Life – 5 dimensions 5 level (EQ- 5D) | EQ-5D mobility, EQ-5D self-care, EQ-5D usual activities, EQ-5D pain/discomfort, EQ-5D anxiety/depression | For each EQ-5D dimension, the proportion of patients with "no problems" will be summarized using descriptive statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population Ixekizumab-treated patients: nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 Assessed during Period 2 and Period 3 combined |
| 30) | | For each EQ-5D dimension, the proportion of patients with "no problems" will be analyzed by: Logistic regression analysis with NRI; Fisher's exact test with NRI | Randomized withdrawal ITT population | Assessed during Period 3<br>through 40 weeks of<br>Randomized Treatment |
| | EQ-5D-5L UK Population-<br>based index score, | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | EQ-5D VAS | | Ixekizumab-treated patients:<br>nonrandomized population and randomized<br>withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assessed during Period 3<br>through 40 weeks of<br>Randomized Treatment |
| Quick<br>Inventory of | Observed and change from baseline in the following | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| Depressive<br>Symptoma-<br>tology-Self | QIDS-SR16 domains: (1) sad mood (2) concentration | | Ixekizumab-treated patients: nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |

| Measure | Variable | Analysis Method (Section 6.1) | Population (Section 6.6.1) | Comparison/Time Point |
|---|---|---|---|---|
| Report 16 Items (QIDS- | (3) self-criticism (4) suicidal ideation (5) interest | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population | Assessed during Period 3<br>through 40 weeks of<br>Randomized Treatment |
| SR16) | (6) energy/fatigue<br>(7) sleep disturbance (initial, middle, and late insomnia or | Descriptive Statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population with baseline QIDS-SR16 total score of ≥11 | Assessed during Period 2 |
| | hypersomnia (8) decrease/increase in appetite/weight (9) psychomotor | | Ixekizumab-treated patients with baseline QIDS-SR16 total score of ≥11: nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | agitation/retardation Observed and change from baseline in QIDS-SR16 total score | MMRM;<br>ANCOVA with mBOCF | Randomized withdrawal ITT population with baseline QIDS-SR16 total score of ≥11 | Assessed during Period 3<br>through 40 weeks of<br>Randomized Treatment |
| | QIDS-SR16 total score categories: None (no depression): 0-5 Mild: 6-10 Moderate: 11 – 15 Severe: 16 – 20 Very severe: 21 – 27. | Descriptive Statistics for ixekizumab 80 mg Q2W Shift table from maximum baseline for ixekizumab 80 mg Q2W Descriptive statistics on the category based on the maximum post-baseline: for ixekizumab 80 mg Q2W • Improved; maximum post-baseline category < | Initial open-label treatment period population | All post-baseline visits in Period 2 |
| | | maximum baseline category o Worsened; maximum post-<br>baseline category > maximum baseline category | Ixekizumab-treated patients:<br>nonrandomized population and randomized<br>withdrawal ITT population | All post-baseline visits in<br>Period 2 and Period 3<br>combined |
| | | <ul> <li>Same; maximum post-<br/>baseline category =<br/>maximum baseline<br/>category.</li> </ul> | Randomized withdrawal ITT population | Assessed during Period 3<br>through 40 weeks of<br>Randomized Treatment |

| Measure | Variable | Analysis Method (Section 6.1) | Population (Section 6.6.1) | Comparison/Time Point |
|---|---|---|---|---|
| | Proportion of patients with at least a 50% decrease in | Descriptive statistics for ixekizumab 80 mg Q2W | Initial open-label treatment period population | Assessed during Period 2 |
| | QIDS-SR16 total score | | Ixekizumab-treated patients: nonrandomized population and randomized withdrawal ITT population | Assessed during Period 2 and Period 3 combined |
| | | Logistic regression analysis with NRI; Fisher's exact test with NRI | Randomized withdrawal ITT population | Assessed during Period 3<br>through 40 Weeks of<br>Randomized Treatment |

Abbreviations: ANCOVA = analysis of covariance; ITT = intent-to-treat; mBOCF = modified baseline carried forward; MCS = Mental Component Summary; MMRM = mixed-effects model of repeated measures; NRI = nonresponder imputation; PCS = Physical Component Summary; Q2W = every 2 weeks; UK = United Kingdom; VAS = visual analog scale.

### 6.20. Annual Report Analyses

Annual report analyses will be documented in a separate document.

### **6.21. Clinical Trial Registry Analyses**

Additional analyses will be performed for the purpose of fulfilling the Clinical Trial Registry (CTR) requirements.

Analyses provided for the CTR requirements include summary of AEs, provided as a dataset which will be converted to an XML file. Both Serious Adverse Events and 'Other' Adverse Events are summarized: by treatment group and MedDRA PT.

- An AE is considered 'Serious' whether or not it is a TEAE.
- An AE is considered in the 'Other' category if it is both a TEAE and is not serious. For each Serious AE and 'Other' AE, for each term and treatment group, the following are provided:
  - o the number of participants at risk of an event
  - o the number of participants who experienced each event term
  - o the number of events experienced.
- Consistent with www.ClinicalTrials.gov requirements, 'Other' AEs that occur in fewer than 5% of patients/subjects in every treatment group may not be included if a 5% threshold is chosen (5% is the minimum threshold).
- Adverse event reporting is consistent with other document disclosures for example, the clinical study report (CSR), manuscripts, and so forth.

## 7. Unblinding Plan

Refer to the I1F-MC-RHBF Blinding and Unblinding plan.

#### 8. References

- [APA] American Psychiatry Association. Diagnostic and Statistical Manual of Mental Disorders. 4th ed. Washington DC: American Psychiatric Association; 1994.
- Basra MKA, Fenech R, Gatt RM, Salek MS, Finlay AY. The Dermatology Life Quality Index 1994-2007: a comprehensive review of validation data and clinical results. *Br J Dermatol*. 2008;159(5):997-1035.
- Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. *BMJ*. 1992;305(6846):160-164.
- Clegg DO, Reda DJ, Mejias E, Cannon GW, Weisman MH, Taylor T, Budiman-Mak E, Blackburn WD, Vassey FB, Mahowald ML, Cush JJ, Schumacher HR Jr, Silverman SL, Alepa FP, Luggen ME, Cohen MR, Makkena R, Haakenson CM, Ward RH, Manaster BJ, Anderson RJ, Ward JR, Henderson WG. Comparison of sulfasalazine and placebo in the treatment of psoriatic arthritis. A Department of Veterans Affairs Cooperative Study. *Arthritis Rheum*. 1996;39(12):2013-2020.
- Coates LC, Fransen J, Helliwell PS. Defining minimal disease activity in psoriatic arthritis: a proposed objective target for treatment. *Ann Rheum Dis.* 2010;69(1):48–53.
- Coates LC, Helliwell PS. Validation of minimal disease activity criteria for psoriatic arthritis using interventional trial data. *Arthritis Care Res.* 2010;62(7):965–969.
- Columbia University Medical Center. Columbia–Suicide Severity Rating Scale (C-SSRS) web site. Available at: http://www.cssrs.columbia.edu. Accessed April 21, 2011.
- [EMA] European Medicines Agency. Committee for Medicinal Products for Human Use (CHMP). Guideline on clinical investigation of medicinal products indicated for the treatment of psoriasis. November 2004. Available at: http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2009/09/WC50 0003329.pdf. Accessed March 17, 2015.
- EuroQol Group. EQ-5D-5L User Guide. Basic information on how to use the EQ-5D-5L instrument. Version 2.0. October 2013. Available at: http://www.euroqol.org/fileadmin/user\_upload/Documenten/PDF/Folders\_Flyers/EQ-5D-5L\_UserGuide\_2015.pdf. Accessed July 28, 2015.
- Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)—a simple practical measure for routine clinical use. *Clin Exp Dermatol*. 1994;19(3):210-216.
- Fredriksson T, Pettersson U. Severe psoriasis—oral therapy with a new retinoid. *Dermatologica*. 1978;157(4):238-244.
- Fries JF, Spitz P, Kraines RG, Holman HR. Measurement of patient outcome in arthritis. *Arthritis Rheum.* 1980;23(2):137-145.
- Fries JF, Spitz PW, Young DY. The dimensions of health outcomes: the health assessment questionnaire, disability and pain scales. *J Rheumatol*. 1982;9(5):789-793.

- Healy PJ, Helliwell PS. Measuring dactylitis in clinical trials: which is the best instrument to use? *J Rheumatol*. 2007;34:1302-1306.
- Healy PJ, Helliwell PS. Measuring clinical enthesitis in psoriatic arthritis: assessment of existing measures and development of an instrument specific to psoriatic arthritis. *Arthritis Rheum*. 2008;59(5):686-691.
- Helliwell PS, Firth J, Ibrahim GH, Melsom RD, Shah I, Turner DE. Development of an assessment tool for dactylitis in patients with psoriatic arthritis. *J Rheumatol*. 2005;32:1745-1750.
- Helliwell PS, FitzGerald O, Fransen J, Gladman DD, Kreuger GG, Callis-Duffin K, McHugh N, Mease PJ, Strand V, Waxman R, Azevedo VF, Beltran Ostos A, Carneiro S, Cauli A, Espinoza LR, Flynn JA, Hassan N, Healy P, Kerzberg EM, Lee YJ, Lubrano E, Marchesoni A, Marzo-Ortega H, Porru G, Moreta EG, Nash P, Raffayova H, Ranza R, Raychaudhuri SP, Roussou E, Scarpa R, Song YW, Soriano ER, Tak PP, Ujfalussy I, de Vlam K, Walsh JA. The development of candidate composite disease activity and responder indices for psoriatic arthritis (GRACE project). *Ann Rheum Dis.* 2013;72(6):986-991.
- Helliwell PS, FitzGerald O, Fransen J. Composite disease activity and responder indices for psoriatic arthritis: a report from the GRAPPA 2013 meeting on development of cutoffs for both disease activity states and response. *J Rheumatol*. 2014;41(6):1212-1217.
- Hongbo Y, Thomas CL, Harrison MA, Salek MS, Finlay AY. Translating the science of quality of life into practice: What do dermatology life quality index scores mean? *J Invest Dermatol*. 2005;125(4):659-664.
- Khilji FA, Gonzalez M, Finlay AY. Clinical meaning of change in Dermatology Life Quality Index scores. *Br J Dermatol*. 2002;147(suppl 62):50.
- Mease PJ. Measures of psoriatic arthritis: Tender and Swollen Joint Assessment, Psoriasis Area and Severity Index (PASI), Nail Psoriasis Severity Index (NAPSI), Modified Nail Psoriasis Severity Index (mNAPSI), Mander/Newcastle Enthesitis Index (MEI), Leeds Enthesitis Index (LEI), Spondyloarthritis Research Consortium of Canada (SPARCC), Maastricht Ankylosing Spondylitis Enthesis Score (MASES), Leeds Dactylitis Index (LDI), Patient Global for Psoriatic Arthritis, Dermatology Life Quality Index (DLQI), Psoriatic Arthritis Quality of Life (PsAQOL), Functional Assessment of Chronic Illness Therapy—Fatigue (FACIT-F), Psoriatic Arthritis Response Criteria (PsARC), Psoriatic Arthritis Joint Activity Index (PsAJAI), Disease Activity in Psoriatic Arthritis (DAPSA), and Composite Psoriatic Disease Activity Index (CPDAI). *Arthritis Care Res.* 2011;63(S11):S64–S85.
- Mease PJ, Heckaman M, Kary S, Kupper H. Application and modifications of minimal disease activity measures for patients with psoriatic arthritis treated with adalimumab: subanalyses of ADEPT. *J Rheumatol.* 2013;40(5):647-52.
- Mumtaz A, Gallagher P, Kirby B, Waxman R, Coates LC, Veale JD, Helliwell P, FitzGerald O. Development of a preliminary composite disease activity index in psoriatic arthritis. *Ann Rheum Dis.* 2011;70(2):272-277.
- [NPF] National Psoriasis Foundation. The Psoriasis and Psoriatic Arthritis Pocket Guide. Portland, OR. 2009.

- Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. *Am J Pyschiatry*. 2007;164(7):1035-1043.
- Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. *Pharmacoeconomics*. 1993;4(5):353-365.
- Reilly Associates. Work Productivity and Activity Impairment Questionnaire: Specific Health Problem V2.0 (WPAI:SHP). Available at: http://www.reillyassociates.net/WPAI\_SHP.html. Accessed 8 July 2014.
- Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item quick inventory of depressive symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. *Biol Psychiatry*. 2003;54(50):573-583. Erratum in *Biol Psychiatry*. 2003;54(5);585.
- Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: Summary report-Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. *J Allergy Clin Immunol*. 2006;117(2):391–397.
- Saris-Baglama RN, Dewey CJ, Chisholm GB, Plumb E, King J, Rasicot P, Kosinski M, Bjorner JB, Ware JE. QualityMetric Health Outcomes<sup>TM</sup> Scoring Software 4.5 User's Guide. Lincoln, RI: QualityMetric Incorporated; 2004.
- Smolen JS, Breedveld FC, Eberl G, Jones I, Leeming M, Wylie GL, Kirkpatrick J. Validity and reliability of the twenty-eight-joint count for the assessment of rheumatoid arthritis activity. *Arthritis Rheum.* 1995;38(1):38-43.
- Smolen JS, Schoels M, Aletaha D. Disease Activity and response assessment in psoriatic arthritis using the Disease Activity Index for Psoriatic Arthritis (DAPSA). A brief review. *Clin Exp Rheumatol*. 2015;33(93):S48-S50.
- Szende A, Oppe M, Devlin N, eds. EQ-5D Value Sets: Inventory, Comparative Review and User Guide. Dordrecht, Netherlands: Springer; 2007.
- Trivedi MH, Rush AJ, Ibrahim HM, Carmody TJ, Biggs MM, Suppes T, Crismon ML, Shores-Wilson K, Toprac MG, Dennehy EB, Witte B, Kashner TM. The Inventory of Depressive Symptomatology, Clinician Rating (IDS-C) and Self-Report (IDS-SR), and the Quick Inventory of Depressive Symptomatology, Clinician Rating (QIDS-C) and Self-Report (QIDS-SR) in public sector patients with mood disorders: a psychometric evaluation. *Psychol Med.* 2004;34(1):73-82.
- University of Pittsburgh Epidemiology Data Center. Inventory of Depressive Symptomatology (IDS) and Quick Inventory of Depressive Symptomatology (QIDS). Available at: http://www.ids-qids.org. Accessed July 08, 2014.

Vander Cruyssen B, Van Looy S, Wyns B, Westhovens R, Durez P, Van den Bosch F, Veys EM, Mielants H, De Clerck L, Peretz A, Malaise M, Verbruggen L, Vastesaeger N, Geldhof A, Boullart L, De Keyser F. DAS28 best reflects the physician's clinical judgment of response to infliximab therapy in rheumatoid arthritis patients: validation of the DAS28 score in patients under infliximab treatment. *Arthritis Res Ther.* 2005;7(5):R1063-R1071.

Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36), I: Conceptual framework and item selection. *Med Care*. 1992;30(6):473-483.

## 9. Appendices

# Appendix 1. Algorithm for Calculating Classification for Psoriatic Arthritis (CASPAR) Total Score

The classification for psoriatic arthritis (CASPAR) total score is defined as the summation of the following 5 categories in patients with inflammatory articular disease (joint, spine, or entheseal):

- Either:
  - o Evidence of current psoriasis (2 points) or
  - o a personal history of psoriasis or a family history of psoriasis (1 point)
- Typical psoriatic nail dystrophy including onycholysis, pitting, and hyperkeratosis observed on current physical examination (1 point)
- A negative test result for the presence of rheumatoid factor by any method except latex (1 point)
- Either current dactylitis, defined as swelling of an entire digit, or a history of dactylitis recorded by a rheumatologist (1 point)
- Radiographic evidence of juxta-articular new bone formation appearing as illdefined ossification near joint margins (but excluding osteophyte formation) on plain radiographs of the hand or foot (1 point)

If any of the above individual categories have a missing score, then the CASPAR total score will be the sum of the non-missing categories. If all of the above categories are missing then the CASPAR total score will equal 0.

#### Note the following:

- Current psoriasis is defined as psoriatic skin or scalp disease present today as judged by a rheumatologist or dermatologist.†
- A personal history of psoriasis is defined as a history of psoriasis that may be
  obtained from a patient, family physician, dermatologist, rheumatologist, or
  other qualified health care provider.
- A family history of psoriasis is defined as a history of psoriasis in a first- or second-degree relative according to patient report.

Taylor, W, Gladman, D, Helliwell, P, Marchesoni, A, Mease, P, Mielants, H, CASPAR Study Group. Classification criteria for psoriatic arthritis: development of new criteria from a large international study. *Arthritis Rheum.* 2006;54(8):2665–2673.

# Appendix 2. Algorithm for Calculating Coates Criteria for Minimal Disease Activity (MDA)

Coates criteria for MDA defines a state of disease activity and not a change in disease and includes all attributes of PsA. Coates criteria for MDA uses a composite of 7 key outcome measures. A patient is considered as achieving MDA if they fulfill 5 of the following 7 outcome criterion (Coates et al. 2010; Coates and Helliwell 2010):

- TJC ≤ 1;
- SJC ≤ 1;
- PASI total score  $\leq 1$  or BSA  $\leq 3$ ;
- Patient pain VAS score of  $\leq 15$ ;
- Patient global VAS score of  $\leq 20$ ;
- HAQ-DI score  $\leq 0.5$ ;
- Tender entheseal points (of 18 entheseal points)  $\leq 1$ .

The modified Coates criteria for MDA is calculated in the same manner as the Coates criteria for MDA substituting sPGA for PASI. Therefore, a patient is considered as achieving modified MDA if they fulfill 5 of the following 7 outcome criterion (Mease et al. 2013):

- TJC  $\leq 1$ ;
- SJC ≤ 1;
- sPGA (0,1) or BSA  $\leq 3$ ;
- Patient pain VAS score of  $\leq 15$ ;
- Patient global VAS score of  $\leq 20$ ;
- HAQ-DI score  $\leq 0.5$ ;
- Tender entheseal points (of 18 entheseal points)  $\leq 1$ .

Note the 18 tender entheseal points are measured from combining the unique entheseal sites from the LEI and the SPARCC. The LEI consists of 6 entheseal sites and the SPARCC consists of 16 entheseal sites.

### **Appendix 3.** Algorithm for Calculating Joint Counts

Joints are evaluated and recorded as either non-evaluable, or if evaluable, then if tenderness is present or absent, and if swelling is present or absent. In total, 68 joints are assessed for tenderness and 66 are assessed for swelling. Hips are not assessed for swelling.

The number of tender/swollen joints will be calculated by summing all joints checked to have tenderness/swelling present. If at least half but not all of the joints are evaluable, then the observed prorated joint count will be calculated instead. The prorated scores for TJC will be adjusted based upon the number of evaluable joints: the counted score will be multiplied by 68 then divided by the number of joints evaluated (excluding non-evaluable joints and any joints with a missing response). For example: if only 60 of the 68 joints are assessed to be evaluable at a visit, and 32 of those 60 are tender, the prorated joint count is  $(32/60) \times 68 = 36.27$  (not 32). The prorated joint count will be rounded up to the next integer and be used in calculating the percent change from baseline in TJC. The same algorithm will be applied to the calculation of percent change from baseline in SJC with the exception that the counted score will be multiplied by 66 then divided by the number of joints evaluated. If less than half of the joints are evaluable, the number of tender/swollen joints is missing.

This same algorithm will be used for the calculation of TJC and SJC based on 28 joints, which is part of the 28 diarthrodial joint count, based on C-reactive protein (DAS28-CRP) score.

# Appendix 4. Algorithm for Calculating the Health Assessment Questionnaire—Disability Index (HAQ-DI)

The Health Assessment Questionnaire—Disability Index (HAQ-DI) is a patient-reported questionnaire to measure disease-associated disability (assessment of physical function). It consists of 24 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities (Fries et al. 1980, 1982).

- Dressing and grooming (C1. Dress yourself, including tying shoelaces and doing buttons, C2. Shampooing your Hair)
  - Includes 2 component questions, 1 device checkbox (devices used for dressing), 1 help checkbox
- Arising (C1. Stand up from straight chair, C2. Get in and out of bed)
  - o Includes 2 component questions, 1 device checkbox (built-up or special chair), 1 help checkbox
- Eating (C1. Cut your meat, C2. Lift a cup or glass to your mouth, C3. Open a new carton of milk)
  - Includes 3 component questions, 1 device checkbox (build-up or special utensils),
     1 help checkbox)
- Walking (C1. Walk outdoors on flat ground, C2. Climb up 5 steps)
  - o Includes 2 component questions, 4 device checkboxes (cane, walker, crutches, wheelchair), 1 help checkbox
- Hygiene (C1. Wash and dry your body, C2. Take a tub bath, C3. Gen on and off the toilet)
  - o Includes 3 component questions, 4 device checkboxes (raised toilet seat, bathtub seat, bathtub bar, long-handled appliances in bathroom), 1 help checkbox.
- Reach (C1. Reach and get down a 5 pound object (such as a bag of sugar) from just above your head, C2. Bend down to pick up clothing from the floor)
  - Includes 2 component questions, 1 device checkbox (long-handled appliances for reach), 1 help checkbox
- Grip (C1. Open car doors, C2. Open jars which have been previously opened, C3. Turn faucets on and off)
  - o Includes 3 component questions, 1 device checkbox (jar opener), 1 help checkbox
- Activities (C1. Run errands and shop, C2. Get in and out of a car, C3. Do chores such as vacuuming or yard work)
  - o Includes 3 component questions, 1 help checkbox

In order to compute the HAQ-DI (Standard Disability Index) score, the following scores are assigned to the responses:

- Without any difficulty = 0
- With some difficulty = 1

- With much difficulty = 2
- Unable to do = 3.

The disability section of the questionnaire scores the patient's self-perception on the degree of difficulty (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do) when dressing and grooming, arising, eating, walking, hygiene, reach, grip, and performing other daily activities. The reported use of special aids or devices and/or the need for assistance of another person to perform these activities is also assessed. The scores for each of the functional domains will be averaged to calculate the functional disability index.

#### **Calculating the HAQ-DI:**

The patient must have a score for at least 6 of the 8 categories. If there are <6 categories completed, a HAQ-DI cannot be computed.

- A category score is determined from the highest score of the subcategories, or components, in that category. (For example, in the category ARISING there are 3 subcategory items. If a patient responds with a 1, 2, and 0, respectively; the category score is 2.)
- Adjust for use of aids/devices and/or help from another person when indicated:
  - When there are no aids or devices or help indicated for a category, the category's score is not modified.
    - When aids or devices or help ARE indicated by the patient, adjust the score for a category by increasing a 0 or a 1 to a 2. If a patient's highest score for that sub-category is a 2 it remains a 2, and if a 3, it remains a 3.
  - o Sum the 8 category scores
  - o Divide the sum by the number of categories answered (range 6-8).

The scale is not truly continuous but has 25 possible values (that is, 0, 0.125, 0.250, 0.375 ... 3). The mapping of the aids or devices to the categories is the following:

| HAQ-DI Category | Companion aids or devices item |
|---|---|
| Dressing and Grooming | Devices used for dressing (button hook, zipper pull, long handled shoe horn, etc.) |
| Arising | Built up or special chair |
| Eating | Built up or special utensils |
| Walking | Cane, walker, crutches, wheelchair |
| Hygiene | Long handled appliances in bathroom; bathtub seat; raised toilet seat; bathtub bar |
| Reach | Long handled appliances for reach |
| Grip | Jar opener (for jars previously opened) |

Abbreviations: HAQ-DI = Health Assessment Questionnaire–disability index.

# Appendix 5. Algorithm for Determining American College of Rheumatology (ACR) Response

Details presented in this appendix will use "x" as a generic symbol, and the appropriate number (either 20, 50, or 70) is to be filled in when implementing in dataset programming code.

American College of Rheumatology (ACRx) response is defined as  $\ge x\%$  improvement from baseline in tender joint count (68 counts) and  $\ge x\%$  improvement in swollen joint count (66 counts), and  $\ge x\%$  improvement in at least 3 of the following 5 items:

- Patient's global assessment of arthritis pain
- Patient's global assessment of disease activity
- Physician's global assessment of disease activity
- Health Assessment Questionnaire–Disability Index (HAQ-DI)
- C-reactive protein (CRP)

The following abbreviations will be used throughout this appendix to refer to the items needed in the algorithm definitions:

| Parameter | Abbreviation for the Parameter |
|---|---|
| % improvement in tender joint count | TJC68 |
| % improvement in swollen joint count | SJC66 |
| % improvement in patient's assessment pain | PATPAIN |
| % improvement in patient's global assessment of disease activity | PATGA |
| % improvement in physician's global assessment of disease activity | PHYGA |
| % improvement in HAQ-DI | HAQ |
| % improvement in CRP | CRP |

For all 7 parameters mentioned above, % improvement at a visit is calculated as:

(baseline value – value at visit) \* 100 / baseline value.

#### To calculate the *observed* ACRx response at a visit:

- Step1: If the patient discontinued from the study prior to reaching the visit, then STOP assign ACRx response as blank (that is, missing). Otherwise, calculate the % improvement at the visit for all 7 parameters as described above.
- Step2:
  - If 68 total joint count score (TJC68) AND 66 swollen joint count score (SJC66) are BOTH  $\ge x\%$ , then proceed to Step 3.
  - O If both are non-missing but one or both is <x%, then STOP assign the patient as a nonresponder for ACRx.
  - o If either or both are missing, proceed as follows:

- a. If both are missing, then STOP assign ACRx response as blank (that is, missing).
- b. If one of TJC68 or SJC66 is missing and the non-missing value is < x%, then STOP assign the patient as a nonresponder for ACRx.
- c. If one of TJC68 or SJC66 is missing and the non-missing value is  $\ge x\%$ , then STOP assign ACRx response as blank (that is, missing).
- Step3: Consider the following 5 variables: patient's assessment pain (PATPAIN), patient's global assessment of disease activity (PATGA), physician's global assessment of disease activity (PHYGA), HAQ, and CRP.
  - o If 3 or more items are missing, then STOP assign ACRx response as blank (that is, missing).
  - o If 3 or more items are non-missing, then proceed with the following order:
    - d. If at least 3 items are  $\ge x\%$ , then STOP assign the patient as a responder for ACRx.
    - e. If at least 3 items are < x%, then STOP assign the patient as a nonresponder for ACRx.
    - f. If  $\leq$ 3 items are  $\geq$ x%, then STOP assign ACRx response as blank (that is, missing).

To calculate the ACRx response at post-baseline visits up to Week 104 using NRI:

- Step 1: Calculate the % improvement at the visit for all 7 parameters as described above.
- Step 2: If all 7 parameters are missing at the visit, or if the patient discontinued from the study prior to reaching the visit, then STOP assign the patient as a nonresponder for ACRx.
- Step 3: If at least 1 of the 7 parameters is non-missing at the visit and the patient is still enrolled in the study, then use LOCF to fill in any missing values.
- Step 4: If TJC68 AND SJC66 are BOTH  $\ge x\%$ , then proceed to Step 5. If both are non-missing but one or both is  $\le x\%$ , then STOP assign the patient as a nonresponder for ACRx. If either or both are missing, then STOP assign the patient as a nonresponder for ACRx.
- Step 5: Consider the following 5 variables: PATPAIN, PATGA, PHYGA, HAQ, CRP.
  - o If 3 or more of the 5 items are non-missing, then:
    - If 3 or more of the 5 items are  $\ge x\%$ , then STOP assign the patient as a responder for ACRx.
    - If <3 of those 5 items are  $\ge x\%$ , then STOP assign the patient as a nonresponder for ACRx.
  - o If  $\geq$ 3 of the 5 items are missing, then STOP assign the patient as a nonresponder for ACRx.
### Appendix 6. Derivation of SF-36v2® Health Survey, Acute Version Scores

The SF-36v2® Health Survey Scoring Software (QualityMetric Health Outcomes™ Scoring Software 4.5) will be used to calculate the SF-36v2® 8-domain and 2-component summary scores (Saris-Baglama et al. 2004). The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) is a 36-item, patient-completed measure designed to be a short, multipurpose assessment of health in the areas of physical functioning, role-physical, role-emotional, bodily pain, vitality, social functioning, mental health, and general health. The 2 overarching dimensions of mental well-being and physical well-being are captured by the Physical Component Summary (PCS) and Mental Component Summary (MCS) scores, respectively. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. Items are answered on Likert scales of varying lengths. In this study, the SF-36 acute version will be used, which has a 1-week recall.

The Scoring Software performs a 4-step process to calculate raw domain scores and t-scores consisting of

- 1. Data Cleaning and Item recording: First, data are checked for out of range values, converting invalid items to missing values. Next, items (BP01, BP02, GH01, GH03, GH05, VT01, VT02, SF01, MH03, MH05) are reverse scored, so that higher scores denote better health for all SF-36 items.
- 2. Although current research indicates a linear relationship between the SF-36 items and the underlying health concept, empirical research suggests that items GH01 and BP01 require recalibration to satisfy important scaling assumptions. Item GH01 will be rescored according to the following table:

| Response to GH01 | Recommended Value / Recalibrated Value |
|------------------|----------------------------------------|
| Excellent | 5.0 |
| Very Good | 4.4 |
| Good | 3.4 |
| Fair | 2.0 |
| Poor | 1.0 |

The BP01 will be rescored with

| Response Choices | Final Item Value |
|------------------|------------------|
| None | 6.0 |
| Very mild | 5.4 |
| Mild | 4.2 |
| Moderate | 3.1 |
| Severe | 2.2 |
| Very severe | 1.0 |

#### Item 08 (BP02) will be rescored if BP01 and BP02 were answered

| Response Choices | If BP02 Pre-coded<br>Item Value | and BP01 Pre-coded<br>Item Value | Then Final Item 08<br>(BP02) Value |
|---|---|---|---|
| Not at all | 1 | 1 | 6 |
| Not at all | 1 | 2-6 | 5 |
| A little bit | 2 | 1-6 | 4 |
| Moderately | 3 | 1-6 | 3 |
| Quite a bit | 4 | 1-6 | 2 |
| Extremely | 5 | 1-6 | 1 |

#### Scoring of BP02 if BP01 is not answered:

| Response Choices | Final Item Value |
|------------------|------------------|
| Not at all | 6.0 |
| A little bit | 4.75 |
| Moderately | 3.5 |
| Quite a bit | 2.25 |
| Extremely | 1.0 |

- 3. After this rescoring, the raw domain scores will be calculated for the scale. Domain scores are the simple algebraic sum of the final values for all items in that scale.
- 4. All raw domain scores will be transformed to a 0-100 scale, with 0 being the lowest and 100 the highest possible score.
- 5. Finally, the 0-100 scores will be transformed to t-score based scores. First, a z-score transformation using the mean for the respective recall period, here 1 week recall, of the 1998 general U.S. population will be used. Then the distribution of z-score is linearly transformed to have a mean of 50 and a SD of 10 by multiplying each z-score with 10 and adding 50.

The calculation of component scores is a 3-step process using the domain scores, calculated as described above:

- 1. The standardized scores from Step 5, depending on the chosen recall period, are calculated.
- 2. These standardized Physical and Mental component scores are calculated as the weighted sums by the factor score coefficients, derived from the 1990 general US population, with the domain scores. If any domain score is missing then the aggregate Physical or Mental score will not be calculated.
- 3. The PCS and MCS are linearly transformed by multiplying by 10 and adding 50 to obtain the aggregate t-score based scoring.

To run the scoring algorithm, the SF-36 items recorded in the study database will be exported into a comma- or tab-separated values file (\*.csv, \*.tab). This file will then be loaded into the Scoring Software to perform the calculations described above. The resulting raw domain scores and t-scores (domain scores) will then be exported into a comma- or tab-separated values file and imported into SAS for storage in the Study Data Tabulation Mode/Analysis Data Model (SDTM/ADaM) datasets.

The comma- or tab-separated values file, each row will be one patient record and the first row will comprise the header columns, will have the following column specification: (to comply with the Scoring Software requirements)

| eCRF<br>Row<br># | Column label<br>for export to<br>comma- or<br>tab-separated | Annotated SF-36 eCRF<br>Variable<br>[Format:<br>SF36V2RXX SF36V2F1] | Item Number,<br>Score range | eCRF question / Specification |
|---|---|---|---|---|
| | values file [*.csv, *.tab] | , | | |
| 1 | GH01 | [SF36V2R01_SF36V2F1] | Item # 1,<br>Range 1-5 | In general, would you say your health is: |
| 2 | HT | [SF36V2R02_SF36V2F1] | Item # 2,<br>Range 1-5 | Compared to one week ago, how would you rate your health in general now? |
| 3 | PF01 | [SF36V2R03_SF36V2F1] | Item # 3a,<br>Range 1-3 | Vigorous activities, such as running, lifting heavy objects, participating in strenuous sports |
| 4 | PF02 | [SF36V2R04_SF36V2F1] | Item # 3b,<br>Range 1-3 | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf |
| 5 | PF03 | [SF36V2R05_SF36V2F1] | Item # 3c,<br>Range 1-3 | Lifting or carrying groceries |
| 6 | PF04 | [SF36V2R06_SF36V2F1] | Item # 3d,<br>Range 1-3 | Climbing several flights of stairs |
| 7 | PF05 | [SF36V2R07_SF36V2F1] | Item # 3e,<br>Range 1-3 | Climbing one flight of stairs |
| 8 | PF06 | [SF36V2R08_SF36V2F1] | Item # 3f,<br>Range 1-3 | Bending, kneeling, or stooping |
| 9 | PF07 | [SF36V2R09_SF36V2F1] | Item # 3g,<br>Range 1-3 | Walking more than a mile |
| 10 | PF08 | [SF36V2R10_SF36V2F1] | Item # 3h, | Walking several hundred yards |

| eCRF | Column label | Annotated SF-36 eCRF | Item Number, | eCRF question / Specification |
|---|---|---|---|---|
| Row | for export to | Variable | Score range | |
| # | comma- or | [Format: | | |
| | tab-separated | SF36V2RXX_SF36V2F1] | | |
| | values file | | | |
| | [*.csv, *.tab] | | | |
| | | | Range 1-3 | |
| 11 | PF09 | [SF36V2R11_SF36V2F1] | Item # 3i, | Walking one hundred yards |
| | | | Range 1-3 | |
| 12 | PF10 | [SF36V2R12_SF36V2F1] | Item # 3j, | Bathing or dressing yourself |
| 12 | DD01 | ICEA (MARIA CEA (MAELL | Range 1-3 | |
| 13 | RP01 | [SF36V2R13_SF36V2F1] | Item # 4a, | Cut down the amount of time you spent |
| 1.4 | DD02 | ICEA (MARIA CEA (MAEI) | Range 1-5 | on work or other activities |
| 14 | RP02 | [SF36V2R14_SF36V2F1] | Item # 4b, | Accomplished less than you would like |
| 1.5 | DD02 | ICEA (MARAIS CEA (MARAI) | Range 1-5 | W. 1: 1: 1 1: 1 0 1 4 |
| 15 | RP03 | [SF36V2R15_SF36V2F1] | Item # 4c, | Were limited in the kind of work or other |
| 1.6 | DD04 | ICE2(MARIA CE2(MAEI) | Range 1-5 | activities |
| 16 | RP04 | [SF36V2R16_SF36V2F1] | Item # 4d, | Had difficulty performing the work or |
| | | | Range 1-5 | other activities (for example, it took extra |
| 17 | RE01 | [CE24V2D17 CE24V2E1] | Item # 5a, | effort) Cut down the amount of time you spent |
| 1 / | KEUI | [SF36V2R17_SF36V2F1] | Range 1-5 | on work or other activities |
| 18 | RE02 | [SF36V2R18_SF36V2F1] | Item # 5b, | Accomplished less than you would like |
| 10 | KEU2 | [5F30V2K16_5F30V2F1] | Range 1-5 | Accomplished less than you would like |
| 19 | RE03 | [SF36V2R19_SF36V2F1] | Item # 5c, | Did work or other activities less carefully |
| 19 | KE03 | [51:50 \ 2 \ K1 \ 2 \ 51:50 \ \ 2 \ F1 ] | Range 1-5 | than usual |
| 20 | SF01 | [SF36V2R20_SF36V2F1] | Item # 6, | During the past week, to what extent has |
| 20 | 51 01 | [51 50 12120_51 50 121 1] | Range 1-5 | your physical health or emotional |
| | | | Trainge 1 3 | problems interfered with your normal |
| | | | | social activities with family, friends, |
| | | | | neighbors, or groups? |
| 21 | BP01 | [SF36V2R21_SF36V2F1] | Item # 7, | How much bodily pain have you had |
| | | , | Range 1-6 | during the past week? |
| 22 | BP02 | [SF36V2R22_SF36V2F1] | Item # 8, | During the past week, how much did pain |
| | | | Range 1-5 | interfere with your normal work |
| | | | | (including both work outside the home |
| | | | | and housework)? |
| 23 | VT01 | [SF36V2R23_SF36V2F1] | Item # 9a, | Did you feel full of life? |
| | | | Range 1-5 | |
| 24 | MH01 | [SF36V2R24_SF36V2F1] | Item # 9b, | Have you been very nervous? |
| | | | Range 1-5 | |
| 25 | MH02 | [SF36V2R25_SF36V2F1] | Item # 9c, | Have you felt so down in the dumps that |
| | | | Range 1-5 | nothing could cheer you up? |
| 26 | MH03 | [SF36V2R26_SF36V2F1] | Item # 9d, | Have you felt calm and peaceful? |
| | | | Range 1-5 | |
| 27 | VT02 | [SF36V2R27_SF36V2F1] | Item # 9e, | Did you have a lot of energy? |
| | | | Range 1-5 | |
| 28 | MH04 | [SF36V2R28_SF36V2F1] | Item # 9f, | Have you felt downhearted and |
| | | | Range 1-5 | depressed? |

| eCRF | Column label | Annotated SF-36 eCRF | Item Number, | eCRF question / Specification |
|---|---|---|---|---|
| Row | for export to | Variable | Score range | |
| # | comma- or | [Format: | | |
| | tab-separated | SF36V2RXX_SF36V2F1] | | |
| | values file | | | |
| | [*.csv, *.tab] | | | |
| 29 | VT03 | [SF36V2R29_SF36V2F1] | Item # 9g, | Did you feel worn out? |
| | | | Range 1-5 | |
| 30 | MH05 | [SF36V2R30_SF36V2F1] | Item # 9h, | Have you been happy? |
| | | | Range 1-5 | |
| 31 | VT04 | [SF36V2R31_SF36V2F1] | Item # 9i, | Did you feel tired? |
| | | | Range 1-5 | |
| 32 | SF02 | [SF36V2R32_SF36V2F1] | Item # 10, | During the past week, how much of the |
| | | | Range 1-5 | time has your physical health or |
| | | | | emotional problems interfered with your |
| | | | | social activities (like visiting with friends, |
| | | | | relatives, etc.)? |
| 33 | GH02 | [SF36V2R33_SF36V2F1] | Item # 11a, | I seem to get sick a little easier than other |
| | | | Range 1-5 | people |
| 34 | GH03 | [SF36V2R34_SF36V2F1] | Item # 11b, | I am as healthy as anybody I know |
| | | | Range 1-5 | |
| 35 | GH04 | [SF36V2R35_SF36V2F1] | Item # 11c, | I expect my health to get worse |
| | | | Range 1-5 | |
| 36 | GH05 | [SF36V2R36_SF36V2F1] | Item # 11d, | My health is excellent |
| | | | Range 1-5 | |
| | SUBJID | | | Subjects ID |
| | VISID | | | Visid ID |
| | Gender | | | Sex coded as: f/m |
| | DateOfBirth | | | Date of birth formatted as: mm/dd/yyyy |
| | | | | (when scoring software is run in US), or |
| | | | | dd/mm/yyyy (when scoring software is |
| | | | | run in non-US) |
| | RecordID | | | Running number for the exported records |

Abbreviations: eCRF = electronic case report form; SF-36 = Medical Outcomes Study 36-Item Short-Form Health Survey.

The SF-36 Scoring Software will derive raw domain scores and t-scores that can be exported into a comma- or tab-separated values file (\*.csv, \*.tab) with the following columns added:

| Column label added to comma- or tab-<br>separated values file from export | Scoring Software specification |
|---|---|
| [*.csv, *.tab] | |
| PF | Physical Functioning domain score |
| RP | Role Limitations Due To Physical Health domain score |
| BP | Bodily Pain domain score |
| GH | General Health Perceptions domain score |
| VT | Vitality domain score |
| SF | Social Functioning domain score |
| RE | Role Limitations Due To Emotional Problems domain score |
| MH | Mental Health domain score |
| PCS | Physical Component score |
| MCS | Mental health Component score |

For scoring the trial data, the Missing Data Estimator option will not be selected. If an item is missing, there will be no imputation conducted by the Scoring Software. <u>Only</u> complete questionnaire data will be scored.

The Scoring Software also allows for calculating domain and component scores from weights derived from an oblique factor solution for comparative purposes. This option will not be used.

The SF-36 scoring using the Scoring Software will be conducted by a 2 person team overseeing each other in a single scoring session. In case of relevant observations during the scoring, those will be documented in pertinent meeting minutes and filed as part of the study documentation.

# Appendix 7. Anti-infective Medications and Anatomical Therapeutic Chemical (ATC) Code List and Programming Guide

This appendix provides the code list of Anatomical Therapeutic chemical (ATC) of anti-infective medications and the programming guidance.

| ATC | ATC | |
|---|---|---|
| Code | Level | ATC Description (Based on ATC Dictionary 18Jan2016) |
| A01AB | 4 | ANTIINFECTIVES AND ANTISEPTICS FOR LOCAL ORAL TREA |
| A02BD | 4 | COMBINATIONS FOR ERADICATION OF HELICOBACTER PYLOR |
| A07A | 3 | INTESTINAL ANTIINFECTIVES |
| A07AA | 4 | ANTIBIOTICS |
| A07AB | 4 | SULFONAMIDES |
| A07AC | 4 | IMIDAZOLE DERIVATIVES |
| A07AX | 4 | OTHER INTESTINAL ANTIINFECTIVES |
| B05CA | 4 | ANTIINFECTIVES |
| C05AB | 4 | ANTIBIOTICS |
| D01 | 2 | ANTIFUNGALS FOR DERMATOLOGICAL USE |
| D01A | 3 | ANTIFUNGALS FOR TOPICAL USE |
| D01AA | 4 | ANTIBIOTICS |
| D01AC | 4 | IMIDAZOLE AND TRIAZOLE DERIVATIVES |
| D01AE | 4 | OTHER ANTIFUNGALS FOR TOPICAL USE |
| D01B | 3 | ANTIFUNGALS FOR SYSTEMIC USE |
| D01BA | 4 | ANTIFUNGALS FOR SYSTEMIC USE |
| D06 | 2 | ANTIBIOTICS AND CHEMOTHERAPEUTICS FOR DERMATOLOGIC |
| D06A | 3 | ANTIBIOTICS FOR TOPICAL USE |
| D06AA | 4 | TETRACYCLINE AND DERIVATIVES |
| D06AX | 4 | OTHER ANTIBIOTICS FOR TOPICAL USE |
| D06B | 3 | CHEMOTHERAPEUTICS FOR TOPICAL USE |
| D06BA | 4 | SULFONAMIDES |
| D06BB | 4 | ANTIVIRALS |
| D06BX | 4 | OTHER CHEMOTHERAPEUTICS |
| D06C | 3 | ANTIBIOTICS AND CHEMOTHERAPEUTICS, COMBINATIONS |
| D07C | 3 | CORTICOSTEROIDS, COMBINATIONS WITH ANTIBIOTICS |
| D07CA | 4 | CORTICOSTEROIDS, WEAK, COMBINATIONS WITH ANTIBIOTICS |
| D07CB | 4 | CORTICOSTEROIDS, MODERATELY POTENT, COMBINATIONS WITH ANTIBIOTICS |
| D07CC | 4 | CORTICOSTEROIDS, POTENT, COMBINATIONS WITH ANTIBIOTICS |
| D07CD | 4 | CORTICOSTEROIDS, VERY POTENT, COMBINATIONS WITH ANTIBIOTICS |
| D09AA | 4 | MEDICATED DRESSINGS WITH ANTIINFECTIVES |
| D10AF | 4 | ANTIINFECTIVES FOR TREATMENT OF ACNE |
| G01AA | 4 | ANTIBIOTICS |
| G01AC | 4 | QUINOLINE DERIVATIVES |
| G01AE | 4 | SULFONAMIDES |
| G01AF | 4 | IMIDAZOLE DERIVATIVES |

| ATC | ATC | |
|---------|-------|-----------------------------------------------------|
| Code | Level | ATC Description (Based on ATC Dictionary 18Jan2016) |
| G01AG | 4 | TRIAZOLE DERIVATIVES |
| G01AX | 4 | OTHER ANTIINFECTIVES AND ANTISEPTICS |
| G01BA | 4 | ANTIBIOTICS AND CORTICOSTEROIDS |
| G01BC | 4 | QUINOLINE DERIVATIVES AND CORTICOSTEROIDS |
| G01BE | 4 | SULFONAMIDES AND CORTICOSTEROIDS |
| G01BF | 4 | IMIDAZOLE DERIVATIVES AND CORTICOSTEROIDS |
| G04AB | 4 | QUINOLONE DERIVATIVES (EXCL. J01M) |
| G04AC | 4 | NITROFURAN DERIVATIVES |
| G04AG | 4 | OTHER URINARY ANTISEPTICS AND ANTIINFECT |
| G04AH | 4 | SULFONAMIDES IN COMBINATION WITH OTHER DRUGS |
| G04AK | 4 | URINARY ANTISEPT&ANTIINF, COMB EXCL SULFONAMIDES |
| J01 | 2 | ANTIBACTERIALS FOR SYSTEMIC USE |
| J01A | 3 | TETRACYCLINES |
| J01AA | 4 | TETRACYCLINES |
| J01B | 3 | AMPHENICOLS |
| J01BA | 4 | AMPHENICOLS |
| J01C | 3 | BETA-LACTAM ANTIBACTERIALS, PENICILLINS |
| J01CA | 4 | PENICILLINS WITH EXTENDED SPECTRUM |
| J01CE | 4 | BETA-LACTAMASE SENSITIVE PENICILLINS |
| J01CF | 4 | BETA-LACTAMASE RESISTANT PENICILLINS |
| J01CG | 4 | BETA-LACTAMASE INHIBITORS |
| J01CR | 4 | COMBINATIONS OF PENICILLINS, INCL. BETA-LACTAMASE |
| J01D | 3 | OTHER BETA-LACTAM ANTIBACTERIALS |
| J01DA | 4 | CEPHALOSPORINS AND RELATED SUBSTANCES |
| J01DB | 4 | FIRST-GENERATION CEPHALOSPORINS |
| J01DC | 4 | SECOND-GENERATION CEPHALOSPORINS |
| J01DD | 4 | THIRD-GENERATION CEPHALOSPORINS |
| J01DE | 4 | FOURTH-GENERATION CEPHALOSPORINS |
| J01DF | 4 | MONOBACTAMS |
| J01DH | 4 | CARBAPENEMS |
| J01DI | 4 | OTHER CEPHALOSPORINS |
| J01E | 3 | SULFONAMIDES AND TRIMETHOPRIM |
| J01EA | 4 | TRIMETHOPRIM AND DERIVATIVES |
| J01EB | 4 | SHORT-ACTING SULFONAMIDES |
| J01EC | 4 | INTERMEDIATE-ACTING SULFONAMIDES |
| J01ED | 4 | LONG-ACTING SULFONAMIDES |
| J01EE | 4 | COMBINATIONS OF SULFONAMIDES AND TRIMETHOPRIM, INC |
| J01F | 3 | MACROLIDES, LINCOSAMIDES AND STREPTOGRAMINS |
| J01FA | 4 | MACROLIDES MACROLIDES |
| J01FF | 4 | LINCOSAMIDES |
| J01FG | 4 | STREPTOGRAMINS |
| J01G | 3 | AMINOGLYCOSIDE ANTIBACTERIALS |
| J01GA | 4 | STREPTOMYCINS |
| J01GA | 4 | OTHER AMINOGLYCOSIDES |
| J010B | 3 | QUINOLONE ANTIBACTERIALS |
| J01MA | 4 | FLUOROQUINOLONES |
| JULIVIA | 7 | LECONOQUINOLONES |

| ATC | ATC | |
|-------|-------|-----------------------------------------------------|
| Code | Level | ATC Description (Based on ATC Dictionary 18Jan2016) |
| J01MB | 4 | OTHER QUINOLONES |
| J01R | 3 | COMBINATIONS OF ANTIBACTERIALS |
| J01RA | 4 | COMBINATIONS OF ANTIBACTERIALS |
| J01WA | 4 | HERBAL ANTIBACTERIALS FOR SYSTEMIC USE |
| J01WB | 4 | HERBAL URINARY ANTISEPTICS AND ANTIINFECTIVES |
| J01X | 3 | OTHER ANTIBACTERIALS |
| J01XA | 4 | GLYCOPEPTIDE ANTIBACTERIALS |
| J01XB | 4 | POLYMYXINS |
| J01XC | 4 | STEROID ANTIBACTERIALS |
| J01XD | 4 | IMIDAZOLE DERIVATIVES |
| J01XE | 4 | NITROFURAN DERIVATIVES |
| J01XX | 4 | OTHER ANTIBACTERIALS |
| J02 | 2 | ANTIMYCOTICS FOR SYSTEMIC USE |
| J02A | 3 | ANTIMYCOTICS FOR SYSTEMIC USE |
| J02AA | 4 | ANTIBIOTICS |
| J02AB | 4 | IMIDAZOLE DERIVATIVES |
| J02AC | 4 | TRIAZOLE DERIVATIVES |
| J02AX | 4 | OTHER ANTIMYCOTICS FOR SYSTEMIC USE |
| J04AA | 4 | AMINOSALICYLIC ACID AND DERIVATIVES |
| J04AB | 4 | ANTIBIOTICS |
| J04AC | 4 | HYDRAZIDES |
| J04AK | 4 | OTHER DRUGS FOR TREATMENT OF TUBERCULOSIS |
| J04AM | 4 | COMBINATIONS OF DRUGS FOR TREATMENT OF TUBERCULOSI |
| J04B | 3 | DRUGS FOR TREATMENT OF LEPRA |
| J04BA | 4 | DRUGS FOR TREATMENT OF LEPRA |
| J05 | 2 | ANTIVIRALS FOR SYSTEMIC USE |
| J05A | 3 | DIRECT ACTING ANTIVIRALS |
| J05AA | 4 | THIOSEMICARBAZONES |
| J05AB | 4 | NUCLEOSIDES AND NUCLEOTIDES EXCL. REVERSE TRANSCRI |
| J05AC | 4 | CYCLIC AMINES |
| J05AD | 4 | PHOSPHONIC ACID DERIVATIVES |
| J05AE | 4 | PROTEASE INHIBITORS |
| J05AF | 4 | NUCLEOSIDE AND NUCLEOTIDE REVERSE TRANSCRIPTASE IN |
| J05AG | 4 | NON-NUCLEOSIDE REVERSE TRANSCRIPTASE INHIBITORS |
| J05AH | 4 | NEURAMINIDASE INHIBITORS |
| J05AR | 4 | ANTIVIRALS FOR TREATMENT OF HIV INFECTIONS, COMBIN |
| J05AX | 4 | OTHER ANTIVIRALS |
| P01A | 3 | AGENTS AGAINST AMOEBIASIS AND OTHER PROTOZOAL DISE |
| P01AA | 4 | HYDROXYQUINOLINE DERIVATIVES |
| P01AB | 4 | NITROIMIDAZOLE DERIVATIVES |
| P01AC | 4 | DICHLOROACETAMIDE DERIVATIVES |
| P01AR | 4 | ARSENIC COMPOUNDS |
| P01AX | 4 | OTHER AGENTS AGAINST AMOEBIASIS AND OTHER PROTOZOA |
| P01BA | 4 | AMINOQUINOLINES |
| P01BC | 4 | METHANOLQUINOLINES |
| P01BD | 4 | DIAMINOPYRIMIDINES |

| ATC | ATC | |
|-------|-------|----------------------------------------------------------|
| Code | Level | ATC Description (Based on ATC Dictionary 18Jan2016) |
| P01BE | 4 | ARTEMISININ AND DERIVATIVES, PLAIN |
| P01BF | 4 | ARTEMISININ AND DERIVATIVES, COMBINATIONS |
| P01BX | 4 | OTHER ANTIMALARIALS |
| P01C | 3 | AGENTS AGAINST LEISHMANIASIS AND TRYPANOSOMIASIS |
| P01CA | 4 | NITROIMIDAZOLE DERIVATIVES |
| P01CB | 4 | ANTIMONY COMPOUNDS |
| P01CC | 4 | NITROFURAN DERIVATIVES |
| P01CD | 4 | ARSENIC COMPOUNDS |
| P01CX | 4 | OTHER AGENTS AGAINST LEISHMANIASIS AND TRYPANOSOMI |
| P02 | 2 | ANTHELMINTICS |
| P02B | 3 | ANTITREMATODALS |
| P02BA | 4 | QUINOLINE DERIVATIVES AND RELATED SUBSTANCES |
| P02BB | 4 | ORGANOPHOSPHOROUS COMPOUNDS |
| P02BX | 4 | OTHER ANTITREMATODAL AGENTS |
| P02C | 3 | ANTINEMATODAL AGENTS |
| P02CA | 4 | BENZIMIDAZOLE DERIVATIVES |
| P02CB | 4 | PIPERAZINE AND DERIVATIVES |
| P02CC | 4 | TETRAHYDROPYRIMIDINE DERIVATIVES |
| P02CE | 4 | IMIDAZOTHIAZOLE DERIVATIVES |
| P02CF | 4 | AVERMECTINES |
| P02CX | 4 | OTHER ANTINEMATODALS |
| P02D | 3 | ANTICESTODALS |
| P02DA | 4 | SALICYLIC ACID DERIVATIVES |
| P02DW | 4 | HERBAL ANTICESTODALS |
| P02DX | 4 | OTHER ANTICESTODALS |
| P02WA | 4 | HERBAL ANTHELMINTICS |
| P03A | 3 | ECTOPARASITICIDES, INCL. SCABICIDES |
| P03AA | 4 | SULFUR CONTAINING PRODUCTS |
| P03AB | 4 | CHLORINE CONTAINING PRODUCTS |
| P03AC | 4 | PYRETHRINES, INCL. SYNTHETIC COMPOUNDS |
| P03AX | 4 | OTHER ECTOPARASITICIDES, INCL. SCABICIDES |
| P03BA | 4 | PYRETHRINES |
| R02AB | 4 | ANTIBIOTICS |
| S01A | 3 | ANTIINFECTIVES |
| S01AA | 4 | ANTIBIOTICS |
| S01AB | 4 | SULFONAMIDES |
| S01AD | 4 | ANTIVIRALS |
| S01AE | 4 | FLUOROQUINOLONES |
| S01AX | 4 | OTHER ANTIINFECTIVES |
| S01C | 3 | ANTIINFLAMMATORY AGENTS AND ANTIINFECTIVES IN COMB |
| S01CA | 4 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S01CB | 4 | CORTICOSTEROIDS/ANTIINFECTIVES/MYDRIATICS IN COMBI |
| S01CC | 4 | ANTIINFLAMMATORY AGENTS, NON-STEROIDS AND ANTIINFECTIVES |
| S02A | 3 | ANTIINFECTIVES |
| S02AA | 4 | ANTIINFECTIVES |
| S02C | 3 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |

| ATC | ATC | |
|-------|-------|-----------------------------------------------------|
| Code | Level | ATC Description (Based on ATC Dictionary 18Jan2016) |
| S02CA | 4 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S03A | 3 | ANTIINFECTIVES |
| S03AA | 4 | ANTIINFECTIVES |
| S03C | 3 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S03CA | 4 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |

Abbreviation: ATC = World Health Organization Collaborating Centre for Drug Statistics Methodology (WHOCC) Anatomical Therapeutic Chemical (ATC) classification system.

For the above list, the higher level of ATC includes all the lower levels under that level, for example, level 2 term includes all the level 3 terms under it, level 3 term includes all the level 4 terms under it. Therefore, for programming simplicity, the table below provides all the required ATC codes by highest level.

| ATC Level 2 | ATC Level 3 | ATC Level 4 |
|-------------|-------------|-------------|
| | | A01AB |
| | | A02BD |
| | A07A | |
| | | B05CA |
| | | C05AB |
| D01 | | |
| D06 | | |
| | D07C | |
| | | D09AA |
| | | D10AF |
| | | G01AA |
| | | G01AC |
| | | G01AE |
| | | G01AF |
| | | G01AG |
| | | G01AX |
| | | G01BA |
| | | G01BC |
| | | G01BE |
| | | G01BF |
| | | G04AB |
| | | G04AC |
| | | G04AG |
| | | G04AH |
| | | G04AK |
| J01 | | |
| J02 | | |
| | | J04AA |
| | | J04AB |
| | | J04AC |
| | | J04AK |

| ATC Level 2 | ATC Level 3 | ATC Level 4 |
|-------------|-------------|-------------|
| | | J04AM |
| | J04B | |
| J05 | | |
| | P01A | |
| | | P01BA |
| | | P01BC |
| | | P01BD |
| | | P01BE |
| | | P01BF |
| | | P01BX |
| | P01C | |
| P02 | | |
| | P03A | |
| | | P03BA |
| | | R02AB |
| | S01A | |
| | S01C | |
| | S02A | |
| | S02C | |
| | S03A | |
| | S03C | |

Abbreviation: ATC = World Health Organization Collaborating Centre for Drug Statistics Methodology (WHOCC) Anatomical Therapeutic Chemical (ATC) classification system.

# Appendix 8. MedDRA Preferred Terms for Each Category Associated with Criterion 2 for Anaphylactic Allergic Reactions/Hypersensitivity Events

| Preferred Terms (MedDRA Version 21.0) | |
|---|---|
| Category A: Involvement of the Skin/Mucosal Tissue | |
| Administration site hypersensitivity | Localised oedema |
| Administration site rash | Mouth swelling |
| Administration site urticarial | Nasal obstruction |
| Allergic oedema | Nodular rash |
| Allergic otitis externa | Ocular hyperaemia |
| Angioedema | Oedema |
| Circumoral oedema | Oedema mouth |
| Drug eruption | Oedema mucosal |
| Erythema | Orbital oedema |
| Eye allergy | Palatal oedema |
| Eye oedema | Palatal swelling |
| Eye pruritus | Perineal rash |
| Eye swelling | Periorbital oedema |
| Eyelid oedema | Pruritus |
| Face oedema | Pruritus allergic |
| Flushing | Pruritus generalised |
| Generalised erythema | Rash |
| Gingival oedema | Rash erythematous |
| Gingival swelling | Rash generalised |
| Idiopathic urticaria | Rash pruritic |
| Injection site dermatitis | Skin oedema |
| Injection site hypersensitivity | Skin swelling |
| Injection site rash | Swelling |
| Injection site urticaria | Swelling face |
| Injection site vasculitis | Swollen tongue |
| Lip oedema | Tongue oedema |
| Lip swelling | Urticaria |
| | Urticaria papular |
| Category B: Respiratory Compromise | |
| Acute respiratory failure | Laryngotracheal oedema |
| Allergic cough | Oropharyngeal spasm |
| Allergic pharyngitis | Oropharyngeal swelling |
| Asthma | Pharyngeal oedema |
| Asthmatic crisis Respiratory arrest | |
| Bronchial hyperreactivity | Respiratory distress |
| Bronchial oedema | Respiratory failure |
| Bronchospasm | Respiratory tract oedema |
| Cardio-respiratory distress | Reversible airways obstruction |
| Chest discomfort | Sensation of foreign body |
| Choking | Sneezing |

| Preferred Terms (MedDRA Version 21.0) | |
|---|---|
| Choking sensation | Spasmodic dysphonia |
| Cough | Status athmaticus |
| Cyanosis | Stridor |
| Dyspnoea | Tachypnea |
| Epiglottic oedema | Throat tightness |
| Hyperventilation | Tracheal obstruction |
| Hypoxia | Tracheal oedema |
| Laryngeal dyspnoea | Upper airway obstruction |
| Laryngeal obstruction | Wheezing |
| Laryngeal oedema | , |
| Laryngitis allergic | |
| Laryngospasm | |
| Category C: Reduced Blood Pressure or Associated Sy | mptoms |
| Blood pressure decreased | Hypoperfusion |
| Blood pressure diastolic decreased | Hypotension |
| Blood pressure systolic decreased | Hypovolaemic shock |
| Cardiac arrest | Incontinence |
| Cardiopulmonary failure | Mean arterial pressure decreased |
| Cardio-respiratory arrest | Peripheral circulatory failure |
| Cardiovascular insufficiency | Presyncope |
| Circulatory collapse | Shock |
| Diastolic hypotension | Shock symptom |
| Distributive shock | Syncope |
| Dizziness | Urinary Incontinence |
| Category D: Persistent Gastrointestinal Symptoms | <u> </u> |
| Abdominal discomfort | Gastrointestinal pain |
| Abdominal pain | Intestinal angioedema |
| Abdominal pain lower | Nausea |
| Abdominal pain upper | Retching |
| Diarrhoea | Visceral pain |
| Epigastric discomfort | Vomiting |
| Gastrointestinal oedema | |

Abbreviations: MedDRA = Medical Dictionary for Regulatory Activities.

### Appendix 9. Allergic Reactions/Hypersensitivity MedDRA Preferred Terms

Allergic reactions/hypersensitivities will be defined using the following MedDRA Preferred Terms as defined in MedDRA:

- Broad and narrow terms in the Anaphylactic reaction SMQ (20000021)
- Broad and narrow terms in the Angioedema SMQ (20000024)
- Broad and narrow terms in the Severe cutaneous adverse reactions SMQ (20000020)
- Broad and narrow terms in the Hypersensitivity SMQ (20000214) excluding the preferred terms as noted below.

The following Preferred Terms (based on review of MedDRA Version 21.0) from the Hypersensitivity SMQ will be excluded from the analysis:

| Administration site derma | tıtıs |
|---------------------------|-------|
| Administration site eczem | a |

Administration site rash Administration site recall reaction

Allergic otitis externa Allergic otitis media Allergic sinusitis

Allergic transfusion reaction Allergy alert test positive Allergy test positive Allergy to surgical sutures

Allergy to vaccine

Anaphylactic transfusion reaction

Antiallergic therapy Application site dermatitis Application site eczema

Application site hypersensitivity

Application site rash

Application site recall reaction Application site urticaria Application site vasculitis

Arthritis allergic

Aspirin-exacerbated respiratory disease Asthma-chronic obstructive pulmonary disease

overlap syndrome Blepharitis allergic

Blood immunoglobulin E abnormal Blood immunoglobulin E increased

Bromoderma

Catheter site dermatitis Catheter site eczema Injection site rash

Injection site recall reaction Injection site urticaria Injection site vasculitis

Instillation site hypersensitivity

Instillation site rash Instillation site urticaria

Iodine allergy

Mast cell degranulation present Medical device site dermatitis Medical device site eczema

Medical device site hypersensitivity

Medical device site rash

Medical device site recall reaction Medical device site urticaria

Nodular rash Pathergy reaction

Radioallergosorbent test positive

Reaction to azo-dyes Reaction to colouring Rhinitis allergic

Shock

Shock symptom Skin test positive Solvent sensitivity

Stoma site hypersensitivity

Stoma site rash Urticaria contact Urticarial vasculitis Vaccination site dermatitis

Vaccination site exfoliation

Catheter site hypersensitivity

Catheter site rash Catheter site urticaria Catheter site vasculitis

Chronic eosinophilic rhinosinusitis

Chronic hyperplastic eosinophilic sinusitis

Circulatory collapse Conjunctivitis allergic Contact stomatitis

Complement factor decreased Complement factor increased Complement factor C1 decreased Complement factor C1 increased Complement factor C2 decreased Complement factor C2 increased Complement factor C3 decreased Complement factor C3 increased Complement factor C4 decreased Complement factor C4 increased Complement fixation abnormal

Complement fixation test positive Contrast media allergy Contrast media reaction Dennie-Morgan fold Dermatitis acneiform Dermatitis contact Dermatitis herpetiformis

Dermatitis infected

Device allergy

Dialysis membrane reaction

Distributive shock Drug cross-reactivity Drug provocation test Eczema infantile

Eczema vaccinatum First use syndrome Fixed drug eruption

Giant conjuctivitis Hand dermatitis

Heparin-induced thrombocytopenia

Hereditary angioedema Implant site dermatitis

Implant site hypersensitivity

Implant site rash Implant site urticaria

Immune-mediated adverse reaction

Incision site dermatitis Incision site rash Infusion site dermatitis Vaccination site eczema

Vaccination site hypersensitivity

Vaccination site rash

Vaccination site recall reaction

Vaccination site urticaria Vaccination site vasculitis

Vaccination site vesicles Vessel puncture site rash

Vessel puncture site vesicles

Vulvovaginal rash Acute respiratory failure Allergy to chemicals

Allergy to fermented products Anti-insulin antibody increased Anti-insulin antibody positive

Anti-insulin receptor antibody increased Anti-insulin receptor antibody positive Blood immunoglobulin A abnormal Blood immunoglobulin A increased

Blood immunoglobulin D increased Blood immunoglobulin G abnormal Blood immunoglobulin G increased Blood immunoglobulin M abnormal

Blood immunoglobulin M increased Immune complex level increased

Immunoglobulins abnormal Immunoglobulins increased Immunology test abnormal Haemolytic transfusion reaction

Infantile asthma Fixed eruption Rhinitis perennial Seasonal allergy

| Infusion site eczema |
|---------------------------------|
| Infusion site hypersensitivity |
| Infusion site rash |
| Infusion site recall reaction |
| Infusion site urticaria |
| Infusion site vasculitis |
| Injection site dermatitis |
| Injection site eczema |
| Injection site hypersensitivity |

## Appendix 10. Algorithm for Calculating Composite Psoriatic Disease Activity Index (CPDAI)

Composite Psoriatic Disease Activity Index (CPDAI) is a validated instrument to assess composite psoriatic disease activity and response to therapy (Mumtaz et al. 2011). This instrument assesses individual domains:

- peripheral arthritis as assessed by the number of tender and swollen joints and the Health Assessment Questionnaire—Disability Index(HAQ-DI)
- skin as assessed by the Psoriasis Area and Severity Index (PASI) and the Dermatology Life Quality Index (DLQI)
- enthesitis as assessed by the number of sites with enthesitis and the HAQ-DI
- dactylitis as assessed by the number of digits affected and the HAQ-DI
- Spinal disease as assessed by the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and Ankylosing Spondylitis Quality of Life (ASQoL)

The table below shows the instruments for each domain and the range in their total score:

| Domain | Instrument | <b>Total Score Range</b> |
|----------------------|-------------|--------------------------|
| Peripheral arthritis | TJC/SJC | 0-68/0-66 |
| | HAQ-DI | 0-3 |
| Skin disease | PASI | 0-72 |
| | DLQI | 0-30 |
| Enthesitis | LEI | 0-6 |
| | HAQ-DI | 0-3 |
| Dactylitis | Digit Score | 0-20 |
| | HAQ-DI | 0-3 |
| Spinal disease | BASDAI | 0-10 |
| | ASQoL | 0-18 |

Abbreviations: ASQoL = Ankylosing Spondylitis Quality of Life; BASDAI = Bath Ankylosing Spondylitis Disease Activity Index; DLQI = Dermatology Life Quality Index; HAQ-DI = Health Assessment Questionnaire—Disability Index; LEI = Leeds Enthesitis Index; PASI = Psoriasis Area and Severity Index; SJC = swollen joint count; TJC = tender joint count.

Each domain is scored from 0 to 3. Individual domain scores are summed to give an overall composite CPDAI score. The composite scores range from 0 to 15 for the assessment, with a higher score indicating higher disease activity. See the table below for details:

| Domain | Not involved (0) | Mild (1) | Moderate (2) | Severe (3) |
|---|---|---|---|---|
| Peripheral arthritis | TJC and $SJC = 0$ | TJC or SJC $\leq$ 4; and | TJC or SJC $\leq$ 4 and | TJC or SJC $>$ 4 and |
| | | HAQ-DI < 0.5 | $HAQ-DI \ge 0.5$ ; or | HAQ-DI ≥0.5 |
| | | | TJC or SJC $>$ 4 and | |
| | | | HAQ-DI < 0.5 | |
| Skin disease | Absence of plaque | $PASI \le 10$ and | $PASI \le 10$ and | PASI > 10 and |
| | psoriasis as defined | DLQI ≤ 10 | DLQI > 10; or | DLQI > 10 |
| | PASI = 0 | | PASI > 10 and | |
| | | | DLQI ≤ 10 | |
| Enthesitis | Absence of | LEI ≤ 3 sites; | LEI $\leq$ 3 sites and | LEI > 3 and HAQ- |
| | enthesitis as defined | HAQ-DI < 0.5 | $HAQ-DI \ge 0.5$ ; or | DI ≥0.5 |
| | (LEI = 0 | | LEI > 3 sites and | |
| | | | HAQ-DI < 0.5 | |
| Dactylitis | Absence of dactylitis | Digit score ≤ 3 | Digit score $\leq 3$ and | Digit score > 3 and |
| | as defined by the | digits; | $HAQ-DI \ge 0.5$ ; or | HAQ-DI ≥0.5 |
| | Digit score $= 0$ | HAQ-DI < 0.5 | Digit score > 3 and | |
| | | | HAQ-DI < 0.5 | |
| Spinal disease | BASDAI = 0 and | BASDAI < 4; | BASDAI < 4 and | BASDAI > 4 and |
| | ASQoL = 0 | ASQoL < 6 | $ASQoL \ge 6$ ; or | $ASQol \ge 6$ |
| | | | BASDAI $\geq$ 4 and | |
| | | | ASQoL < 6 | |

Abbreviations: BASDAI = Bath Ankylosing Spondylitis Disease Activity Index; DLQI = Dermatology Life Quality Index; HAQ-DI = ; LEI = Leeds Enthesitis Index; PASI = Psoriasis Area and Severity Index; SJC = swollen joint count; TCJ = tender joint count;

The modified CPDAI will sum up each domain with the exception of spinal disease. The composite scores range from 0 to 12 for the assessment, with a higher score indicating higher disease activity.

## Appendix 11. Lilly-defined MedDRA V21.0 Preferred Terms for Inflammatory Bowel Disease (IBD)

| Condition | Preferred Term (MedDRA version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| Inflammatory bowel disease | Inflammatory bowel disease | Narrow |
| Crohn's disease | Crohn's disease | Narrow |
| Ulcerative colitis | Acute haemorrhagic ulcerative colitis | Narrow |
| | Colitis ulcerative | Narrow |
| | Proctitis ulcerative | Narrow |
| Non-specific terms | Abscess intestinal | Broad |
| | Anal abscess | Broad |
| | Anal fistula | Broad |
| | Anal fistula excision | Broad |
| | Anal fistula infection | Broad |
| | Anovulvar fistula | Broad |
| | Aorto-duodenal fistula | Broad |
| | Colitis | Broad |
| | Colon fistula repair | Broad |
| | Colonic fistula | Broad |
| | Diverticular fistula | Broad |
| | Duodenal fistula | Broad |
| | Enterocolitis haemorrhagic | Broad |
| | Enterocolonic fistula | Broad |
| | Enterocutaneous fistula | Broad |
| | Enterovesical fistula | Broad |
| | Gastrointestinal fistula | Broad |
| | Gastrointestinal fistula repair | Broad |
| | Fistula of small intestine | Broad |
| | Intestinal fistula | Broad |
| | Intestinal fistula infection | Broad |
| | Intestinal fistula repair | Broad |
| | Jejunal fistula | Broad |

| Condition | Preferred Term (MedDRA version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Large intestinal ulcer perforation | Broad |
| | Rectal fistula repair | Broad |
| | Faecal calprotectin abnormal | Broad |
| | Faecal calprotectin increased | Broad |
| | Proctitis haemorrhagic | Broad |
| | Pseudopolyposis | Broad |
| | Rectoprostatic fistula | Broad |
| | Rectourethral fistula | Broad |

Abbreviations: MedDRA = Medical Dictionary for Regulatory Activities.

## Appendix 12. Lilly-defined MedDRA V21.0 Preferred Terms for Opportunistic Infections (OI)

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | (NEUDKA VEISION 21.0) | Classification |
| Pneumocystis jirovecii (II) | Pneumocystis jirovecii pneumonia | Narrow |
| 3 3 ( ) | Pneumocystis jirovecii infection | |
| | Pneumocystis test positive | Broad |
| | Blood beta-D-glucan | |
| | Blood beta-D-glucan abnormal | |
| | Blood beta-D-glucan increased | |
| | Gomori methenamine silver stain | |
| | Carbon monoxide diffusing capacity decreased | |
| II | Carbon monoxide diffusing capacity | Name |
| Human polyomavirus infection | Human polyomavirus infection | Narrow |
| including BK virus disease including | Polyomavirus-associated nephropathy BK virus infection | |
| PVAN (V), and | Progressive multifocal | |
| Progressive Multifocal<br>Leukoencephalopathy (IV) | leukoencephalopathy | |
| Leukoencepharopathy (11) | JC virus infection | |
| | JC virus miccuon JC virus granule cell neuronopathy | |
| | Anti-JC virus antibody index | Broad |
| | Polyomavirus test | Dioad |
| | Polyomavirus test positive | |
| | Giant papillary conjuctivitis | |
| | JC virus test | |
| | JC virus test positive | |
| | JC polyomavirus test | |
| Cytomegalovirus disease (V) | Cytomegalovirus chorioretinitis | Narrow |
| - 3 3 | Cytomegalovirus colitis | |
| | Cytomegalovirus duodenitis | |
| | Cytomegalovirus enteritis | |
| | Cytomegalovirus enterocolitis | |
| | Cytomegalovirus gastritis | |
| | Cytomegalovirus gastroenteritis | |
| | Cytomegalovirus gastrointestinal infection | |
| | Cytomegalovirus gastrointestinal ulcer | |
| | Cytomegalovirus hepatitis | |
| | Cytomegalovirus infection | |
| | Cytomegalovirus mononucleosis | |
| | Cytomegalovirus mucocutaneous ulcer | |
| | Cytomegalovirus myelomeningoradiculitis Bartonellosis | |
| | (disseminated disease only) (V) | |
| | Cytomegalovirus nephritis | |
| | Cytomegalovirus oesophagitis | |
| | Cytomegalovirus pancreatitis | |
| | Cytomegalovirus pericarditis | |
| | Cytomegalovirus syndrome | |
| | Cytomegalovirus urinary tract infection | |
| | Cytomegalovirus viraemia | 1 |

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Disseminated cytomegaloviral infection | |
| | Encephalitis cytomegalovirus | |
| | Pneumonia cytomegaloviral | |
| | Cytomegalovirus test | Broad |
| | Cytomegalovirus test positive | |
| Post-transplant lymphoproliferative disorder (EBV) (V) | Epstein-Barr virus associated lymphoma Epstein-Barr virus associated lymphoproliferative disorder | Narrow |
| | Epstein-Barr virus positive mucocutaneous ulcer | |
| | Post transplant lymphoproliferative disorder | |
| | Epstein-Barr viraemia | Broad |
| | Epstein-Barr virus infection | Broad |
| | Lymphoproliferative disorder | |
| | Lymphoproliferative disorder in remission | |
| | Oral hairy leukoplakia | |
| Bartonellosis (disseminated disease | Bacillary angiomatosis | Narrow |
| only) (V) | Peliosis hepatis | |
| 3, \ , | Splenic peliosis | |
| | Systemic bartonellosis | |
| | Trench fever | |
| | Bartonella test | Broad |
| | Bartonella test positive | |
| | Bartonellosis | |
| | Cat scratch disease | |
| Blastomycosis (IV) | Blastomycosis | Narrow |
| | Epididymitis blastomyces | |
| | Osteomyelitis blastomyces | |
| | Pneumonia blastomyces | |
| | N/A | Broad |
| Toxoplasmosis (myocarditis, | Cerebral toxoplasmosis | Narrow |
| pneumonitis, or characteristic | Eye infection toxoplasmal | |
| retinochoroiditis only) (IV) | Hepatitis toxoplasmal | |
| | Meningitis toxoplasmal | |
| | Myocarditis toxoplasmal | |
| | Pneumonia toxoplasmal | Dunad |
| | Toxoplasma serology Toxoplasma serology positive | Broad |
| | Toxoplasmosis Toxoplasmosis | |
| Coccidioidomycosis. (II) | Coccidioides encephalitis | Narrow |
| Coccidioraciny costs. (11) | Coccidioidomycosis | T tuil o w |
| | Cutaneous coccidioidomycosis | |
| | Meningitis coccidioides | |
| | N/A | Broad |
| Histoplasmosis (II) | Acute pulmonary histoplasmosis | Narrow |
| | Chronic pulmonary histoplasmosis | |
| | Endocarditis histoplasma | |
| | Histoplasmosis | |
| | Histoplasmosis cutaneous | |
| | Histoplasmosis disseminated | |
| | Meningitis histoplasma | |
| | Pericarditis histoplasma | |
| | Retinitis histoplasma | |

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Presumed ocular histoplasmosis syndrome | Broad |
| Aspergillosis (invasive disease only) | Aspergillosis oral | Narrow |
| (II) | Cerebral aspergillosis | |
| | Meningitis aspergillus | |
| | Oro-pharyngeal aspergillosis | |
| | Aspergillus infection | Broad |
| | Aspergillus test | |
| | Aspergillus test positive | |
| | Bronchopulmonary aspergillosis | |
| | Sinusitis aspergillus | 2.7 |
| Candidiasis (invasive disease or oral | Candida endophthalmitis | Narrow |
| not limited to the tongue) (II) | Candida osteomyelitis | |
| | Candida pneumonia | |
| | Candida retinitis | |
| | Candida sepsis<br>Cerebral candidiasis | |
| | Endocarditis candida | |
| | Fungal oesophagitis Gastrointestinal candidiasis | |
| | Hepatic candidiasis | |
| | Hepatosplenic candidiasis | |
| | Meningitis candida | |
| | Oesophageal candidiasis | |
| | Oropharyngeal candidiasis | |
| | Peritoneal candidiasis | |
| | Splenic candidiasis | |
| | Systemic candida | |
| | Bladder candidiasis | Broad |
| | Candida infection | Droad |
| | Candida test | |
| | Candida test positive | |
| | Mucocutaneous candidiasis | |
| | Oral candidiasis | |
| | Oral fungal infection | |
| | Respiratory moniliasis | |
| Cryptococcosis (II) | Cryptococcal cutaneous infection | Narrow |
| ()F() | Cryptococcal fungaemia | |
| | Cryptococcosis | |
| | Disseminated cryptococcosis | |
| | Gastroenteritis cryptococcal | |
| | Meningitis cryptococcal | |
| | Neurocryptococcosis | |
| | Osseous cryptococcosis | |
| | Pneumonia cryptococcal | |
| | Cryptococcus test | Broad |
| | Cryptococcus test positive | |
| Other invasive fungi: Mucormycosis | Allescheriosis | Narrow |
| (=zygomycosis) [Rhizopus, Mucor, | Fusarium infection | |
| and Lichtheimia], | Mucormycosis | |
| Scedosporum/Pseudallescheria | Scedosporium infection | |
| boydii, Fusarium (II) | Phaeohyphomycosis | |
| | Phaeohyphomycosis brain abscess | |

| Opportunistic Infection | Preferred Term (MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Pseudallescheria infection | |
| | Pseudallescheria sepsis | |
| | See "Non-specific terms" below | Broad |
| Legionellosis (II) | Legionella infection | Narrow |
| 8() | Pneumonia legionella | 1 - 1 - 1 - 1 |
| | Pontiac fever | |
| | Legionella test | Broad |
| | Legionella test positive | |
| Listeria monocytogenes (invasive | Listeria encephalitis | Narrow |
| disease only) (II) | Listeria sepsis | |
| | Meningitis listeria | |
| | Listeriosis | Broad |
| | Listeria test | |
| | Listeria test positive | |
| | Listeraemia | |
| Tuberculosis (I) | Adrenal gland tuberculosis | Narrow |
| (-) | Bone tuberculosis | 1 - 1 - 1 - 1 |
| | Choroid tubercles | |
| | Conjunctivitis tuberculous | |
| | Cutaneous tuberculosis | |
| | Disseminated Bacillus Calmette-Guerin infection | |
| | Disseminated tuberculosis | |
| | Ear tuberculosis | |
| | Epididymitis tuberculous | |
| | Extrapulmonary tuberculosis | |
| | Immune reconstitution inflammatory syndrome | |
| | associated tuberculosis | |
| | Intestinal tuberculosis | |
| | Joint tuberculosis | |
| | Lymph node tuberculosis | |
| | Male genital tract tuberculosis | |
| | Meningitis tuberculous | |
| | Oesophageal tuberculosis | |
| | Oral tuberculosis | |
| | Pericarditis tuberculous | |
| | Peritoneal tuberculosis | |
| | Prostatitis tuberculous | |
| | Pulmonary tuberculoma | |
| | Pulmonary tuberculosis | |
| | Renal tuberculosis | |
| | Salpingitis tuberculous | |
| | Silico tuberculosis | |
| | Spleen tuberculosis | |
| | Thyroid tuberculosis | |
| | Tuberculid | |
| | Tuberculoma of central nervous system | |
| | Tuberculosis | |
| | Tuberculosis bladder | |
| | Tuberculosis gastrointestinal | |
| | Tuberculosis liver | |
| | Tuberculosis of central nervous system | |
| | Tuberculosis of eye | |

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Tuberculosis of genitourinary system | |
| | Tuberculosis of intrathoracic lymph nodes | |
| | Tuberculosis of peripheral lymph nodes | |
| | Tuberculosis ureter | |
| | Tuberculous abscess central nervous system | |
| | Tuberculous endometritis | |
| | Tuberculous laryngitis | |
| | Tuberculous pleurisy | |
| | Tuberculous tenosynovitis | |
| | Interferon gamma release assay | Broad |
| | Interferon gamma release assay positive | |
| | Mycobacterium tuberculosis complex test | |
| | Mycobacterium tuberculosis complex test positive | |
| | Tuberculin test | |
| | Tuberculin test false negative | |
| | Tuberculin test positive | |
| Nocardiosis (II) | Cutaneous nocardiosis | Narrow |
| , , | Nocardia sepsis | |
| | Nocardiosis | |
| | Pulmonary nocardiosis | |
| | Nocardia test positive | Broad |
| Nontuberculous mycobacterium | Atypical mycobacterial infection | Narrow |
| disease (II) | Atypical mycobacterial lower respiratory tract infection | |
| , , | Atypical mycobacterial lymphadenitis | |
| | Atypical mycobacterial pneumonia | |
| | Atypical mycobacterium pericarditis | |
| | Borderline leprosy | |
| | Bovine tuberculosis | |
| | Indeterminate leprosy | |
| | Leprosy | |
| | Lepromatous leprosy | |
| | Mycobacterial infection | |
| | Mycobacterial peritonitis | |
| | Mycobacterium abscessus infection | |
| | Mycobacterium avium complex immune restoration | |
| | disease | |
| | Mycobacterium avium complex infection | |
| | Mycobacterium chelonae infection | |
| | Mycobacterium fortuitum infection | |
| | Mycobacterium kansasii infection | |
| , | Mycobacterium marinum infection | |
| | Mycobacterium ulcerans infection | |
| | Superinfection mycobacterial | |
| , | Tuberculoid leprosy | |
| | Type 1 lepra reaction | |
| , | Type 2 lepra reaction | Broad |
| , | Atypical mycobacterium test positive | Broad |
| | Mycobacterial disease carrier Mycobacterium leprae | |
| | test positive Myschostorium test | |
| | Mycobacterium test | |
| | Mycobacterium test positive | |

| Opportunistic Infection | Preferred Term | Lilly Defined |
|---|---|---|
| | (MedDRA Version 21.0) | Classification |
| only) (II) | Arthritis salmonella | |
| | Meningitis salmonella | |
| | Osteomyelitis salmonella | |
| | Paratyphoid fever | |
| | Pneumonia salmonella | |
| | Salmonella sepsis | |
| | Salmonella bacteraemia | |
| | Typhoid fever | |
| | Salmonella test positive | Broad |
| | Salmonellosis | |
| HBV reactivation (IV) | Hepatitis B reactivation | Narrow |
| | Asymptomatic viral hepatitis | Broad |
| | Chronic hepatitis B | |
| | HBV-DNA polymerase increased | |
| | Hepatitis B | |
| | Hepatitis B DNA assay | |
| | Hepatitis B DNA assay positive | |
| | Hepatitis B DNA increased | |
| | Hepatitis B antigen | |
| | Hepatitis B antigen positive | |
| | Hepatitis B core antigen | |
| | Hepatitis B core antigen positive | |
| | Hepatitis B e antigen | |
| | Hepatitis B e antigen positive | |
| | Hepatitis B surface antigen | |
| | Hepatitis B surface antigen positive | |
| | Hepatitis B virus test | |
| | Hepatitis B virus test positive | |
| | Hepatitis infectious | |
| | Hepatitis post transfusion | |
| | Hepatitis viral | |
| II | Withdrawal hepatitis | Name |
| Herpes simplex (invasive disease | Colitis herpes | Narrow |
| only) (IV) | Gastritis herpes | |
| | Herpes oesophagitis | |
| | Herpes sepsis | |
| | Herpes simplex colitis | |
| | Herpes simplex encephalitis | |
| | Herpes simplex gastritis Herpes simplex hepatitis | |
| | Herpes simplex meningitis | |
| | Herpes simplex meningues Herpes simplex meningoencephalitis | |
| | Herpes simplex meningoencephantis Herpes simplex meningomyelitis | |
| | Herpes simplex meningomyenus Herpes simplex necrotising retinopathy | |
| | Herpes simplex oesophagitis | |
| | Herpes simplex pneumonia | |
| | Herpes simplex sepsis | |
| | Herpes simplex visceral | |
| | Herpes simplex visceral Herpes simplex viraemia | |
| | Meningitis herpes | |
| | Meningoencephalitis herpetic | |
| | Meningomyelitis herpes | |

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Pneumonia herpes viral | |
| | Eczema herpeticum | Broad |
| | Herpes ophthalmic | |
| | Herpes simplex | |
| | Herpes simplex DNA test positive | |
| | Herpes virus infection | |
| | Herpes virus test abnormal | |
| | Herpes simplex virus test positive | |
| | Ophthalmic herpes simplex | |
| Herpes zoster (any form) (II) | Disseminated varicella zoster vaccine virus infection | Narrow |
| 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | Encephalitis post varicella | |
| | Genital herpes zoster | |
| | Herpes zoster | |
| | Herpes zoster cutaneous disseminated | |
| | Herpes zoster disseminated | |
| | Herpes zoster infection neurological | |
| | Herpes zoster meningitis | |
| | Herpes zoster meningoencephalitis | |
| | Herpes zoster meningomyelitis | |
| | Herpes zoster meningoradiculitis | |
| | Herpes zoster necrotising retinopathy | |
| | Herpes zoster oticus | |
| | Herpes zoster olicus Herpes zoster pharyngitis | |
| | Necrotising herpetic retinopathy | |
| | Ophthalmic herpes zoster | |
| | Varicella zoster virus infection | Broad |
| | Varicella virus test | Dioau |
| | Varicella virus test positive | |
| Stronglyoides (hyperinfection | Strongyloidiasis | Narrow |
| syndrome and disseminated forms | N/A | Broad |
| only) (IV) | IV/A | Dioau |
| Paracoccidioides infections (V) | Paracoccidioides infection | Narrow |
| , | Pulmonary paracoccidioidomycosis | |
| | N/A | Broad |
| Penicillium marneffei (V) | Penicillium infection | Narrow |
| 33 ( ) | Penicillium test positive | Broad |
| Sporothrix schenckii (V) | Cutaneous sporotrichosis | Narrow |
| eporoum un semement (+) | Pulmonary sporotrichosis | 11411011 |
| | Sporotrichosis | |
| | N/A | Broad |
| Cryptosporidium species (chronic | Biliary tract infection cryptosporidial | Narrow |
| disease only) (IV) | Cryptosporidiosis infection | Broad |
| anocaso omy, (11) | Gastroenteritis cryptosporidial | Dioud |
| Microsporidiosis (IV) | Microsporidia infection | Narrow |
| wherespondies (1 v ) | N/A | Broad |
| Laighmaniagia (Viceanal anta) (IV) | | |
| Leishmaniasis (Visceral only) (IV) | Visceral leishmaniasis | Narrow |
| T | Leishmaniasis | Broad |
| Trypanosoma cruzi infection | Chagas' cardiomyopathy | Narrow |
| (Chagas' Disease) (disseminated | Meningitis trypanosomal | 1 |
| disease only) (V) | American trypanosomiasis | Broad |
| | Trypanosomiasis | |

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Trypanosoma serology positive | |
| Campylobacteriosis (invasive disease only) (V) | Campylobacter sepsis | Narrow |
| | Campylobacter infection | Broad |
| 3/ \ / | Campylobacter test positive | |
| Shigellosis (invasive disease only) | Shigella sepsis | Narrow |
| (V) | Shigella infection | Broad |
| | Shigella test positive | |
| Vibriosis (invasive disease due to <i>V</i> . | N/A | Narrow |
| vulfnificus) (V) | Vibrio test positive | Broad |
| | Vibrio vulnificus infection | 31044 |
| HCV progression (V) | N/A | Narrow |
| rie · progression ( · ) | Chronic hepatitis C | Broad |
| | Hepatitis C | Broad |
| | Hepatitis C RNA | |
| | Hepatitis C virus test | |
| | Hepatitis C RNA increased | |
| | Hepatitis C RNA positive | |
| | Hepatitis C RNA fluctuation | |
| | Hepatitis C virus test positive | |
| Non-specific terms | N/A | Narrow |
| Tron-specific terms | Abscess fungal | Broad |
| | Alternaria infection | Broad |
| | Arthritis fungal | |
| | Biliary tract infection fungal | |
| | Central nervous system fungal infection | |
| | Cerebral fungal infection | |
| | Encephalitis fungal | |
| | Erythema induratum | |
| | Eye infection fungal | |
| | Fungaemia | |
| | Fungal abscess central nervous system | |
| | Fungal endocarditis | |
| | Fungal labyrinthitis | |
| | Fungal peritonitis | |
| | Fungal pharyngitis | |
| | Fungal retinitis | |
| | Fungal sepsis | |
| | Hepatic infection fungal | |
| | Meningitis fungal | |
| | Mycotic endophthalmitis | |
| | Myocarditis mycotic | |
| | Oropharyngitis fungal | |
| | Osteomyelitis fungal | |
| | Otitis media fungal | |
| | Pancreatitis fungal | |
| | Parasitic lung infection | |
| | Parasitic pneumonia | |
| | Pericarditis fungal | |
| | Phaehyphomycosis Phaehyphomycosis | |
| | Pneumonia fungal | |
| | Pulmonary mycosis | |
| | Pulmonary trichosporonosis | |

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| | Sinusitis fungal Splenic infection fungal Systemic mycosis | |

Abbreviations: MedDRA = Medical Dictionary for Regulatory Activities.

Leo Document ID = e23de465-31a7-4763-9651-e1da7e0a70e4

Approver: PPD

Approval Date & Time: 25-Oct-2018 18:34:52 GMT Signature meaning: Approved